| | CLINICAL PROTOCOL |
|---|---|
| Title: | A PHASE 1B DOSE-ESCALATION AND PHASE 2A STUDY OF TRC105 IN COMBINATION WITH PAZOPANIB IN PATIENTS WITH ADVANCED SOFT TISSUE SARCOMA |
| Protocol Number: | 105SAR101 |
| Study Sponsor: | TRACON Pharmaceuticals, Inc. 8910 University Center Lane, Suite 700 San Diego, CA 92122 |
| | Phone: (858) 550-0780 Facsimile: (858) 550-0786 |
| Medical Monitor: | Charles Theuer, MD, PhD 8910 University Center Lane, Suite 700 San Diego, CA 92122 Direct Phone: (858) 550-0780 x233 Fax: (858) 550-0786 Cell Phone: (858) 344-9400 Email: ctheuer@traconpharma.com |
| Signature & Date: | Signed: Charles Theren Dated: 23 AUG 7016 |
| Version Date: | Original Protocol: April 18 <sup>th</sup> , 2013 Amendment #1: October 1 <sup>st</sup> , 2013 Amendment #2: July 23 <sup>rd</sup> , 2014 Amendment #3: December 2 <sup>nd</sup> , 2014 Amendment #4: April 6th, 2015 Amendment #5: June 2 <sup>nd</sup> , 2015 Amendment #6: December 15 <sup>th</sup> , 2015 Amendment #7: July 22 <sup>nd</sup> , 2016 |

### Statement of Confidentiality:

The information in this document is confidential and proprietary. Any other distribution, copying or disclosure is strictly prohibited unless required by federal regulations or state law. Persons receiving this information must be notified that it is confidential and may not be further disclosed.

# PROCEDURES IN CASE OF EMERGENCY

**Table 1:** Emergency Contact Information

| Role in Study | Name | Address and Telephone number |
|---|---|---|
| Medical Monitor | Charles Theuer, MD, PhD | 8910 University Center Lane, Suite 700 San Diego, CA 92122 Office: (858) 550-0780 x233 Mobile Phone: (858) 344-9400 Email: <a href="mailto:ctheuer@traconpharma.com">ctheuer@traconpharma.com</a> |
| Secondary Medical Monitor | Ronald Shazer, MD | Mobile Phone: (310) 922-8039<br>Email: <u>rshazer@traconpharma.com</u> |

### 1. SYNOPSIS

Name of Sponsor/Company: TRACON Pharmaceuticals, Inc.

Name of Investigational Product: TRC105

Name of Active Ingredient: TRC105

### Title of Study:

A PHASE 1B DOSE-ESCALATION AND PHASE 2A STUDY OF TRC105 IN COMBINATION WITH PAZOPANIB IN PATIENTS WITH ADVANCED SOFT TISSUE SARCOMA

Study center(s): This study will be performed at approximately 9 US centers (sites to be determined).

**Investigators:** To be determined

### **Studied period (years):**

Date first patient enrolled: Oct 2013

Estimated date maximum tolerated dose (MTD) obtained: July 2014

Estimated date last patient enrolled phase 2: December 2016

Estimated date last patient completed: June 2017

# **Phase of development:** 1b/2a

#### Rationale:

Pazopanib is an oral inhibitor of multiple receptor tyrosine kinases, including vascular endothelial growth factor receptor VEGFR-1. VEGFR-2 and VEGFR-3 at the rapeutic plasma concentrations. These receptors are implicated in pathologic angiogenesis, tumor growth, and cancer progression. Pazopanib is approved for the treatment of advanced soft tissue sarcoma, following progression on one prior systemic therapy, based on improved progression free survival, TRC105 is an antibody to CD105, an important angiogenic target on vascular endothelial cells that is distinct from VEGFR. TRC105 inhibits angiogenesis, tumor growth and metastases in preclinical models and complements the activity of bevacizumab and multi-kinase inhibitors that target the VEGFR. In a phase 1 study of advanced solid tumors, TRC105 therapy caused a global reduction in angiogenic biomarkers and reduced tumor burden at doses that were well-tolerated. In a phase 1b study, the combination of TRC105 and bevacizumab produced radiographic reductions in tumor volume in bevacizumabrefractory patients, and was well tolerated. TRC105 potentiates bevacizumab and VEGFR tyrosine kinases (VEGFR TKI) in preclinical models. By targeting a non-VEGF pathway that is upregulated following VEGF inhibition, TRC105 has the potential to complement VEGFR TKIs and could represent a major advance in cancer therapy. Together, the use of TRC105 with pazopanib may result in more effective angiogenesis inhibition and improved clinical efficacy over that seen with pazopanib alone. In the phase 1b portion of the study, TRC105 at its recommended phase 2 dose of 10 mg/kg given by weekly intravenous infusion was combined safely with pazopanib given at 800 mg p.o. once daily. Interim data from the Phase 1b/2 study presented at ASCO 2015 indicated that two patients with cutaneous angiosarcoma achieved complete responses by RECIST. Additionally, a third patient with cutaneous angiosarcoma treated in the phase 2 portion had a 25% reduction in the size of metastatic disease.

| Ot | ojec | tives |
|----|------|-------|
|----|------|-------|

Phase 1b:

### Primary:

• To evaluate safety and tolerability and determine a recommended phase 2 dose for TRC105 when added to standard dose pazopanib in patients with advanced soft tissue sarcoma

### Secondary:

- To assess preliminary evidence of antitumor activity when TRC105 is added to pazopanib, by assessing response rate and progression-free survival
- To characterize the pharmacokinetic profile of TRC105 when given with pazopanib
- To evaluate the formation of TRC105 anti-product antibodies
- To correlate efficacy with expression of endoglin on sarcoma tissue
- To explore pharmacodynamic effects on circulating angiogenic biomarkers

#### Phase 2:

### Primary:

- To estimate the PFS of patients with advanced soft tissue sarcoma by RECIST 1.1
- To estimate the ORR in a cohort of patients with angiosarcoma by RECIST 1.1

### Secondary:

- To estimate the ORR in patients with advanced soft tissue sarcoma by RECIST 1.1, including duration of response
- To estimate the PFS in a cohort of patients with angiosarcoma by RECIST 1.1
- To determine the frequency and severity of adverse events as assessed by NCI CTCAE (Version 4.0)
- To characterize the pharmacokinetic profile of TRC105 and pazopanib
- To evaluate the formation of TRC105 anti-product antibodies
- To explore the correlation of efficacy variables (e.g., PFS and ORR) with endoglin expression on sarcoma
- To explore the effects of TRC105 on circulating angiogenic protein biomarkers

### Methodology:

### Phase 1b:

This is a multicenter, open-label, nonrandomized, phase 1b, dose-finding study of TRC105 in combination with standard dose pazopanib in patients with advanced soft tissue sarcoma. Escalating doses of i.v. TRC105 will be administered weekly or every two weeks beginning with Dose Level 1 in combination with oral pazopanib given as 800 mg p.o. once daily. Intermediate TRC105 doses (below the MTD established during the trial) may be explored based upon clinical, PK, and/or biomarker data.

| Dose Level | Number of<br>Evaluable<br>Subjects | Pazopanib mg p.o., once daily (with dose reduction allowed based on tolerability) | TRC105<br>mg/kg<br>IV |
|---|---|---|---|
| -1 | 3-6 | 800 | 6 (weekly beginning cycle 2 day 1) a |
| 1 (starting dose) | 3-6 | 800 | 8 (weekly beginning cycle 2 day 1) <sup>a</sup> |
| 2 | 3-6 | 800 | 10 (weekly beginning cycle 2 day 1) <sup>a</sup> |
| Expanded Cohort 1 | 9-12 (up to 15 total at the MTD) | 800 | MTD (weekly beginning cycle 2 day 1) <sup>a</sup> |
| 3 | 3-6 | 800 | <ul> <li>10 mg/kg weekly during cycle 1</li> <li>15 mg/kg every two weeks beginning cycle 2 day 1<sup>b</sup></li> </ul> |
| Expanded Cohort 2 | At least 6 patients will be treated at the MTD | 800 | <ul> <li>10 mg/kg weekly during cycle 1</li> <li>15 every two weeks beginning cycle 2 day 1<sup>b</sup></li> </ul> |

<sup>&</sup>lt;sup>a</sup> In dose levels -1 to Expanded Cohort 1, pazopanib will be dosed alone during cycle 1 and dosing with TRC105 will begin on cycle 2 day 1. The first weekly TRC105 dose will be split into two doses whereby 3 mg/kg is administered on cycle 2 day 1 and the balance is administered on cycle 2 day 4, the full dose is then given weekly thereafter starting with cycle 2 day 8.

In dose levels -1, 1, 2 and Expanded Cohort 1, patients will receive 800 mg of pazopanib daily p.o. in cycle 1 for two to four weeks prior to the initial dose of TRC105 on cycle 2 day 1. Dose reductions of pazopanib are allowed during this two to four week period of dosing based on individual patient tolerability. TRC105 dosing will begin at 8 mg/kg (Dose Level 1) on cycle 2 day 1. A -1 Dose Level has also been included (6 mg/kg) and will be enrolled if 8 mg/kg TRC105 dosed with pazopanib exceeds the weekly MTD. For dose levels -1, 1, 2, and Expanded Cohort 1, the DLT evaluation period, for purposes of dose expansion, will be the first 28 days of dosing pazopanib and TRC105 together (e.g., from cycle 2 day 1 through cycle 2 day 28). Each cycle will be 28 days in duration. For dose levels 3, and Expanded Cohort 2, both pazopanib and TRC105 dosing will begin on C1D1 and the DLT evaluation period will be the first 28 days of dosing pazopanib with TRC105 every 2

<sup>&</sup>lt;sup>b</sup> In dose levels 3 and Expanded Cohort 2, pazopanib and TRC105 dosing will begin on cycle 1 day 1. Pazopanib dosing will begin on cycle 1 day 1 and once daily thereafter, and TRC105 will be administered weekly during cycle 1. The first weekly TRC105 dose will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4. Starting on cycle 2 day 1 and beyond, TRC105 will be administered every two weeks on days 1 and 15 once it is determined that the every two week dosing MTD has not been exceeded.

weeks (i.e., from cycle 2 day 1 through cycle 2 day 28). At least 6 patients will be treated at the every two week dosing MTD (or top dose level if a MTD is not determined).

Three patients will be initially enrolled and treated at each dose level. If none of these 3 patients experiences a dose-limiting toxicity (DLT) during the 28-day DLT evaluation period, dose escalation will proceed following review of safety data with site staff including the principal investigators at all sites.

If 1 of 3 patients experiences DLT, the dose level will be expanded to 6 patients. The maximum tolerated dose (MTD) will have been exceeded if  $\geq$  33% of patients experience DLT at a given dose level. DLT will have occurred when a patient has 1 or more toxicity listed in the table below that is at least possibly related to the combination of pazopanib and TRC105 during the 28 day DLT evaluation period. Patients who exit the study for reasons other than DLT or any TRC105 dose delay >2 days in cycle 2 prior to completion of the 28-day DLT evaluation period will be replaced to ensure an adequate safety assessment in each cohort. Patients who experience DLT who receive less than the prescribed dose of TRC105 or pazopanib due to documented toxicity during the DLT evaluation period will be considered evaluable for dose escalation purposes. A given TRC105 dose level may be reenrolled at  $\geq$  50% of the pazopanib dose intensity upon agreement of study investigators.

| Toxicity Category | Drug-Related Toxicity/Grade |
|---|---|
| Hematologic | Grade 4 neutropenia for ≥ 5 days |
| | Febrile neutropenia: grade 4 neutropenia with fever > 38.5 °C both sustained over a 24 hour period. |
| | Neutropenic infection: grade $\geq 3$ neutropenia with grade $\geq 3$ infection |
| | Anemia ≥ grade 4 |
| | Grade > 4 thrombocytopenia or grade ≥ 3 thrombocytopenia and grade ≥ 3 hemorrhage |
| Nonhematologic | Grade 3 or 4 nonhematologic toxicity with the following exceptions: • Nausea, vomiting or diarrhea for < 48 hours <sup>a</sup> |
| | Asymptomatic electrolyte abnormalities<br>that are corrected to grade 1 or better in<br>< 72 hours <sup>b</sup> |
| | headache lasting less than 48 hours |

<sup>&</sup>lt;sup>a</sup>Patients with related grade 3 or 4 diarrhea, nausea or vomiting for ≥ 48 hours despite optimal medical therapy will require a one-level dose-reduction of TRC105.

#### Phase 2:

This is a multicenter, non-randomized, phase 2 study of TRC105 in combination with standard dose pazopanib in patients who have not received pazopanib previously. Sixty three patients are expected to be treated in the phase 2 portion of the study at 10 mg/kg. Patients will receive pazopanib once

<sup>&</sup>lt;sup>b</sup>Patients with related grade 3 or 4 electrolyte abnormalities that persist for ≥ 72 hours will require a one-level dose reduction of TRC105.

daily and will receive TRC105 at 3 mg/kg on cycle 1 day 1, 7 mg/kg on cycle 1 day 4, and 10 mg/kg on cycle 1 day 8 and weekly thereafter. Each cycle is 28 days in duration.

An additional phase 2 cohort of up to thirteen patients with angiosarcoma (angiosarcoma cohort 1) that have progressed following treatment with prior systemic therapy, will be assessed at a TRC105 dose of 10 mg/kg weekly. Patients will initially receive weekly single-agent TRC105 with transition to treatment with the combination of TRC105 and pazopanib at progression per RECIST 1.1.

An additional phase 2 cohort (angiosarcoma cohort 2) of up to thirteen patients with angiosarcoma that have progressed following treatment with prior systemic therapy, will be assessed at a TRC105 dose of 10 mg/kg weekly in combination with 800 mg pazopanib once daily for the first cycle starting on cycle 1 day 1 followed by TRC105 15 mg/kg administered every two weeks starting from cycle 2 day 1 onward in combination with pazopanib 800 mg once daily.

Active patients that are past cycle 1, may be switched to an every 2 week dosing schedule at a TRC105 dose of 15 mg/kg every two weeks once **SPONSOR SENDS NOTIFICATION TO PROCEED WITH EVERY TWO WEEK DOSING**.

Every two week Administration:

- TRC105 will be administered weekly at 10 mg/kg during cycle 1.
  - The first weekly TRC105 dose (10 mg/kg) will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4.
- Starting on cycle 2 day 1 and beyond, TRC105 may be administered every two weeks on days 1 and 15 at the every two week dosing MTD.

Dose reductions of pazopanib are allowed based on individual patient tolerability.

Each cycle in this cohort is 28 days in duration.

### **Number of patients (planned):**

Up to 30 patients with advanced soft tissue sarcoma will be enrolled in the phase 1b portion and 63 patients will be enrolled in the phase 2 portion, and two additional cohorts of up to 13 patients each with angiosarcoma will be enrolled.

### Diagnosis and main criteria for inclusion:

For the phase 1b dose levels -1, 1, 2, and Expanded Cohort 1, prior to administration of TRC105 on cycle 2 day 1, all study patients must maintain eligibility criteria indicating adequate organ function, medical status and ECOG performance status (i.e., all patients must maintain inclusion criterion #4, 5 and 6 and exclusion criteria #8-21 to continue into cycle 2).

### **Inclusion Criteria:**

- 1. Histologically confirmed unresectable soft tissue sarcoma (i.e., non-GIST, non-adipocytic) that has progressed following treatment with chemotherapy. Prior pazopanib is allowed if the drug was not discontinued for toxicity ( Phase 1b only)
- 2. Histologically confirmed metastatic soft tissue sarcoma (i.e., non-GIST, non-adipocytic) that has progressed by RECIST following treatment with anthracycline chemotherapy. Patients

- may have received up to four lines of systemic therapy for metastatic disease and no more than two lines of combination treatment (Phase 2 only)
- 3. Histologically confirmed locally advanced (e.g. unresectable) or metastatic angiosarcoma that has progressed following treatment with prior systemic therapy. Progression must be documented on or following the most recent systemic therapy. Prior pazopanib is allowed if the drug was not discontinued for toxicity (Phase 2 angiosarcoma cohorts only)
- 4. Measurable disease by RECIST
- 5. Age of 12 years or older (patient must weigh  $\geq$  40 kg)
- 6. ECOG performance status  $\leq 1$
- 7. Resolution of all acute adverse events resulting from prior cancer therapies to NCI CTCAE grade ≤ 1 or baseline (except alopecia or neuropathy)
- 8. Adequate organ function as defined by the following criteria:
  - Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5 x ULN in cases of liver metastases
  - Total serum bilirubin  $\leq 1.5$  times the upper limit of normal
  - Absolute neutrophil count (ANC)  $\geq 1500/\mu L$
  - Platelets  $\geq 100,000/\mu L$  without transfusion support within the past 28 days
  - Hemoglobin ≥ 9.0 g/dL without transfusion support within the past 14 days (erythropoietin or darbepoietin permitted)
  - Serum creatinine ≤ 1.5 times the upper limit of normal or creatinine clearance > 30 mL/min by Cockcroft-Gault formula
  - INR from 0.8 to 1.2
- 9. Willingness and ability to consent for self to participate in study
- 10. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
- 11. Available archival tumor specimen of the soft tissue sarcoma that meets inclusion criterion #1, #2 or #3

### **Exclusion Criteria:**

- 1. Prior treatment with TRC105
- 2. Prior treatment with a VEGFR TKI (including pazopanib) (Phase 2 only)
- 3. Current treatment on another therapeutic clinical trial
- 4. Receipt of systemic anticancer therapy, including investigational agents, within 28 days of starting study treatment. If anticancer therapy was given within 28 days of starting study treatment, patients may be included if 5 times the elimination half-life of the drug has passed.
- 5. No major surgical procedure or significant traumatic injury within 6 weeks prior to study registration, and must have fully recovered from any such procedure; date of surgery (if

- applicable) or the anticipated need for a major surgical procedure within the next six months. Note: the following are not considered to be major procedures and are permitted up to 7 days before therapy initiation: Thoracentesis, paracentesis, port placement, laparoscopy, thorascopy, tube thoracostomy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, incisional biopsies, imaging-guided biopsy for diagnostic purposes, and routine dental procedures
- 6. Patients who have received wide field radiotherapy ≤ 28 days (defined as > 50% of volume of pelvic bones or equivalent) or limited field radiation for palliation < 14 days prior to cycle 1 day 1 or those patients who have not recovered adequately from side effects of such therapy
- 7. Uncontrolled chronic hypertension defined as systolic > 150 or diastolic > 90 despite optimal therapy (initiation or adjustment of BP medication prior to study entry is allowed provided that the average of 3 BP readings at a visit prior to enrollment is < 150/90 mm Hg)
- 8. Significant ascites or pericardial or pleural effusion
- 9. History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease. Patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered for at least 28 days.
- 10. Angina, MI, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, PTCA or CABG within the past 6 months. Deep venous thrombosis within 6 months, unless the patient is anti-coagulated without the use of warfarin for at least 2 weeks. In this situation, low molecular weight heparin is preferred.
- 11. Active bleeding or pathologic condition that carries a high risk of bleeding (e.g. hereditary hemorrhagic telangiectasia). Patients who have been uneventfully anti-coagulated with low molecular weight heparin are eligible.
- 12. Thrombolytic use (except to maintain i.v. catheters) within 10 days prior to first day of study therapy
- 13. Known active viral or nonviral hepatitis or cirrhosis
- 14. History of hemorrhage or hemoptysis (> ½ teaspoon bright red blood) within 3 months of starting study treatment
- 15. History of peptic ulcer within the past 3 months of treatment, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 28 days of starting study treatment
- 16. History of gastrointestinal perforation or fistula in the past 6 months, or while previously on antiangiogenic therapy, unless underlying risk has been resolved (e.g., through surgical resection or repair)
- 17. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
- 18. Receipt of a strong CYP3A4 inducer within 12 days prior to cycle 1 day 1 or a strong CYP3A4 inhibitor within 7 days prior to cycle 1 day 1 (Table 14)
- 19. Pregnancy or breastfeeding. Female patients must be surgically sterile (i.e.: hysterectomy) or be postmenopausal, or must agree to use effective contraception during the study and for 3

months following last dose of TRC105. All female patients of reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to first dose. Male patients must be surgically sterile or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. The definition of effective contraception will be based on the judgment of the Principal Investigator or a designated associate.

20. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study

# TRC105 investigational product dose and mode of administration:

#### Phase 1b

Dosing will begin at 8 mg/kg (Dose Level 1); however a -1 Dose Level has also been included (6 mg/kg) and will be enrolled if 8 mg/kg is found to exceed the MTD.

For Dose Level -1, 1, 2 and Expanded Cohort 1, following the appropriate premedication regimen, the first weekly TRC105 dose (cycle 2 day 1) will be split into two doses whereby 3 mg/kg is administered on cycle 2 day 1 and the balance (e.g., 5 mg/kg for Dose Level 1) is administered on cycle 2 day 4. Beginning with cycle 2 day 8 and thereafter, the full (e.g., 8 mg/kg for Dose Level 1) TRC105 dose will be administered i.v. weekly during each 28-day cycle.

For Dose Levels 3, and Expanded Cohort 2, following the appropriate pre-medication regimen, TRC105 will be administered weekly at a dose of 10 mg/kg during cycle 1. The first weekly TRC105 dose will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4. Beginning with cycle 1 day 8 and for the rest of cycle 1, the full (e.g., 10 mg/kg) TRC105 dose will be administered i.v. weekly. Starting on cycle 2 day 1 and beyond, TRC105 will be administered at a dose of 15 mg/kg (Dose Level 3) every two weeks on days 1 and 15 of each 28-day cycle.

### Phase 2

Patients will receive pazopanib once daily and following appropriate premedication regimen will receive TRC105 at 3 mg/kg on cycle 1 day 1, 7 mg/kg on cycle 1 day 4, and 10 mg/kg on cycle 1 day 8 and weekly thereafter. Each cycle is 28 days in duration.TRC105 dose modification is allowed beginning with cycle 2.

### Angiosarcoma cohort 1

Following the appropriate premedication regimen, TRC105 will be administered weekly with the first weekly dose of TRC105 split, with 3 mg/kg administered on cycle 1 day 1 and 7 mg/kg administered on cycle 1 day 4, and then the full dose of 10 mg/kg given on cycle 1 day 8 and weekly thereafter. TRC105 dose modification is allowed beginning with cycle 2.

### Angiosarcoma cohort 2

Following the appropriate premedication regimen, TRC105 will be administered weekly with the first weekly dose of TRC105 split, with 3 mg/kg administered on cycle 1 day 1 and 7 mg/kg administered on cycle 1 day 4, and then the full dose of 10 mg/kg given on cycle 1 day 8 and weekly during Cycle

1. Starting on cycle 2 day 1 and beyond, TRC105 will be administered at a dose of 15 mg/kg every two weeks on days 1 and 15 of each 28-day cycle.

Active patients that are past cycle 1, may be switched to an every 2 week dosing schedule at a TRC105 dose of 15 mg/kg every two weeks once **SPONSOR SENDS NOTIFICATION TO PROCEED WITH EVERY TWO WEEK DOSING**.

### Pazopanib dose and administration:

In phase 1b and phase 2, patients will receive pazopanib 800 mg once daily beginning on cycle 1 day 1.

Angiosarcoma cohort 1 patients will receive pazopanib 800 mg once daily starting at the time of disease progression on TRC105 single-agent.

Angiosarcoma cohort 2 patients will receive pazopanib 800 mg once daily starting on cycle 1 day 1.

Dose modification is allowed based on patient tolerability.

### **Duration of treatment:**

Patients are eligible for treatment until disease progression, unacceptable toxicity or withdrawal of consent, or other reasons. A patient should be withdrawn from study treatment if, in the opinion of the Investigator, it is medically necessary, or if it is the wish of the patient. In addition, patients will be withdrawn from treatment in the case of:

- 1. RECIST 1.1-defined disease progression. In cases where RECIST cannot be applied, progression should be based on unequivocal evidence of progressive disease sufficient to require a change in therapy. In the angiosarcoma cohort 1, disease progression for withdrawal refers to disease progression while receiving TRC105 plus pazopanib combination therapy.
- 2. A need for surgery, radiation, or for other anticancer therapy not specified in the protocol.
- 3. Unable to tolerate pazopanib during cycle 1 (phase 1b dose levels -1, 1, 2 and Expanded Cohort 1 only).
- 4. Lost to follow-up or noncompliant.
- 5. Any TRC105 dose delay > 2 days between cycle 2 day 1 and cycle 2 day 28 (phase 1b only).
- 6. Pregnancy. Pregnant patients should be followed for the duration of the pregnancy and the outcome of the pregnancy should be documented.
- 7. Arterial thrombosis of any grade (including cerebrovascular ischemia, cardiac ischemia/infarction, or peripheral or visceral arterial ischemia) or grade 3 or 4 venous thrombosis (including pulmonary embolism).
- 8. Missed study drug treatment for > 8 consecutive weeks (i.e., both TRC105 and pazopanib dosing held). However, patients who cannot tolerate pazopanib or TRC105 therapy and who demonstrate a response of complete response (CR), partial response (PR) or stable disease (SD) with the combination and are thought to benefit from continued single agent therapy may continue on study on TRC105 or pazopanib alone.

### Parameters to be assessed:

# Safety:

Safety assessments will include physical exams, performance status, laboratory results (complete blood counts and serum chemistry) and 12-lead ECG's, and additional studies as clinically indicated.

A formally chartered Safety Review Team will review safety data. In addition, recurring teleconferences will be held with Investigators at all clinical sites.

### Pharmacokinetics:

Serum TRC105 concentrations will be measured using validated methods at the time points specified in the Schedule of Events.

### Immunogenicity:

Anti-product antibodies will be measured using validated methods at time points specified in the Schedule of Events.

# **Exploratory Biomarkers:**

Concentrations of a panel of angiogenic protein biomarkers in plasma will be measured at baseline and during treatment to explore TRC105 pharmacodynamics.

### **Efficacy**:

RECIST 1.1 will be applied to measurable disease to assess response and progression. Tumor markers will also be evaluated where available.

### **Archival Tumor Specimens:**

Endoglin expression on archival tumor specimens will be correlated with efficacy endpoints (e.g., PFS and ORR).

#### Statistical methods:

### Evaluable Study Population:

The study population for safety and efficacy includes all patients receiving at least a portion of 1 dose of TRC105.

The number of patients to be enrolled in this study will depend upon the observed safety profile, which will determine the number of patients per dose level and the number of dose escalations. It is anticipated that a total of up to 30 patients will be treated in the phase 1b portion and 89 patients will be treated in the phase 2 portion.

#### Phase 1:

The probability of escalation to the next higher dose for each underlying true DLT rate is shown in the table below. For example, for a toxicity that occurs in 5% of patients, there is a > 95% probability of escalating. Conversely, for a common toxicity that occurs with a rate of 70%, the probability of escalating is < 5%.

### Probability of Escalation to the Next Dose for Each True Underlying DLT Rate at a Dose Level

| True Underlying DLT<br>Rate | 5% | | 20% | 30% | 40% | 50% | 60% | 70% | 80% | 90% |
|---|---|---|---|---|---|---|---|---|---|---|
| Probability of Escalating<br>Dose | 0.97 | 0.91 | 0.71 | 0.49 | 0.31 | 0.17 | 0.08 | 0.03 | 0.01 | 0.001 |

The probability of failing to observe toxicity in a sample size of 3 or 6 patients given various true underlying toxicity rates in shown in the table below. For example, with 6 patients, the probability of failing to observe toxicity occurring at least 40% of the time is < 5%.

# Probability of Failing to Observe True Underlying DLT Rate at a Dose Level

| True Underlying DLT Rate | 5% | 10% | 20% | 30% | 40% | 50% | 60% | 70% | 80% | 90% |
|---|---|---|---|---|---|---|---|---|---|---|
| Probability of<br>Failing to<br>Observe Toxicity,<br>N = 3 | 0.86 | 0.73 | 0.51 | 0.34 | 0.22 | 0.13 | 0.006 | 0.027 | 0.008 | 0.001 |
| Probability of Failing to Observe Toxicity, N = 6 | 0.74 | 0.53 | 0.26 | 0.12 | 0.05 | 0.016 | 0.004 | <0.001 | <0.001 | <0.001 |

#### Phase 2:

### Primary analysis:

The primary analysis will test the null hypothesis that the median PFS is equal to 4.6 months. The time-to-event distribution for PFS will be estimated using the Kaplan-Meier method and the analysis will be based on the two-sided 90% confidence interval for the median (equivalent to the use of a one-sided test at the alpha=0.05 level of significance).

An additional phase 2 cohort of up to 13 patients with angiosarcoma will be enrolled (angiosarcoma cohort 1). Assuming a 15% response rate by RECIST with pazopanib alone, 5 responders with TRC105 alone will provide >90% confidence that the true response rate is >15%.

A second additional phase 2 cohort of up to 13 patients with angiosarcoma will be enrolled (angiosarcoma cohort 2). Assuming a 15% response rate by RECIST with pazopanib alone, 5 responders with TRC105 in combination with pazopanib will provide >90% confidence that the true response rate is >15%.

### Sample size justification:

Assuming a true median PFS of 4.6 months, a 9-month accrual period, a 6-month follow-up period, and based on the use of a one-sided test at the alpha=0.05 level of significance, a sample size of 63 patients will provide 86% power to detect a 50% increase in the median PFS (i.e., a median of 6.9 months). For the angiosarcoma cohorts, the two-sided exact 90% binomial with 5 of 13 responders is 16.57% and 64.52%.

# TABLE OF CONTENTS

| 1. | SYNOPSIS | 3 |
|---|---|---|
| 2. | BACKGROUND | 23 |
| 2.1. | Angiogenesis and Cancer | 23 |
| 2.1.1. | Angiogenesis and Advanced Soft Tissue Sarcoma | 23 |
| 2.1.2. | CD105 and Angiogenesis | 24 |
| 2.2. | TRC105 Background | 26 |
| 2.2.1. | Studies with TRC105 | 26 |
| 2.2.1.1. | 105ST101 Phase 1 Monotherapy | 26 |
| 2.2.1.2. | Phase 1b 105ST102 Study with Bevacizumab | 30 |
| 2.2.1.3. | Phase 1b 105RC101 Study with Axitinib | 32 |
| 2.2.1.4. | Phase 1b 105SAR101 Study with Pazopanib | 32 |
| 2.3. | Study Rationale | 32 |
| 2.4. | Population to be Studied | 33 |
| 2.5. | Potential Risks and Benefits to Human Patients | 33 |
| 2.5.1. | Potential Risks | 33 |
| 2.5.2. | Potential Benefits | 36 |
| 2.6. | Justification of the Dose, Schedule and Route of Administration of TRC105 | 36 |
| 2.6.1. | Phase 1b Justification | 36 |
| 2.6.2. | Phase 2 Justification | 37 |
| 2.7. | Conduct | 38 |
| 3. | TRIAL OBJECTIVES AND PURPOSE | 39 |
| 3.1. | Phase 1b Objectives | 39 |
| 3.1.1. | Purpose | 39 |
| 3.1.2. | Primary objectives | 39 |
| 3.1.3. | Secondary objectives | 39 |
| 3.2. | Phase 2 Objectives | 40 |
| 3.2.1. | Purpose | 40 |
| 3.2.2. | Primary objectives | 40 |
| 3.2.3. | Secondary objectives | 40 |
| 4. | INVESTIGATIONAL PLAN | 41 |
| 4.1. | Overall Study Design and Plan | 41 |

# 105SAR101 Protocol Amendment #7, July 22, 2016

| 4.1.1. | Overview | 41 |
|----------|-----------------------------------------|----|
| 4.1.1.1. | Phase 1b Overview | 41 |
| 4.1.1.2. | Phase 2 Overview | 43 |
| 4.1.2. | Trial Procedures | 44 |
| 4.1.2.1. | Screening | 44 |
| 4.1.2.2. | Trial Period | 45 |
| 4.1.3. | End of Study Assessments | 47 |
| 4.1.4. | Post Treatment Follow-up | 48 |
| 5. | SELECTION AND WITHDRAWAL OF PATIENTS | 63 |
| 5.1. | Patient Inclusion Criteria | 63 |
| 5.2. | Exclusion Criteria | 64 |
| 5.3. | Patient Withdrawal Criteria | 65 |
| 6. | TREATMENT OF PATIENTS | 67 |
| 6.1. | Description of TRC105 Study Drug | 67 |
| 6.1.1. | Composition of TRC105 | 67 |
| 6.1.2. | TRC105 Dose Level | 67 |
| 6.1.2.1. | Phase 1b | 67 |
| 6.1.2.2. | Phase 2 | 67 |
| 6.1.3. | TRC105 Packaging and Labeling | 68 |
| 6.1.4. | TRC105 Storage and Shipping | 68 |
| 6.1.5. | TRC105 Preparation | 68 |
| 6.1.6. | TRC105 Administration | 69 |
| 6.1.7. | TRC105 Dose Modification/Dose Delays | 71 |
| 6.1.8. | Management of TRC105 Infusion Reactions | 74 |
| 6.1.9. | TRC105 Study Drug Accountability | 74 |
| 6.1.10. | TRC105 Study Drug Handling and Disposal | 75 |
| 6.2. | Description of Pazopanib | 75 |
| 6.2.1. | Composition of Pazopanib. | 75 |
| 6.2.2. | Pazopanib Dose Level | 75 |
| 6.2.3. | Pazopanib Packaging and Labeling | 75 |
| 6.2.4. | Pazopanib Storage Handling and Disposal | 75 |
| 6.2.5. | Pazopanib Dosing | 76 |

| 6.2.6. | Pazopanib Dose Modification | 76 |
|----------|----------------------------------------------------------|----|
| 6.2.7. | Pazopanib Drug Accountability | 77 |
| 6.3. | Concomitant Medications | 77 |
| 6.4. | Treatment Compliance | 78 |
| 6.4.1. | TRC105 Treatment Compliance | 78 |
| 6.4.2. | Pazopanib Treatment Compliance | 78 |
| 6.5. | Patient Enrollment | 78 |
| 7. | ASSESSMENT OF EFFICACY | 79 |
| 7.1. | Radiological Tumor Assessment | 79 |
| 7.1.1. | Measurability of Tumor Lesions | 79 |
| 7.1.1.1. | Recording Tumor Measurements | 80 |
| 7.1.2. | Definitions of Tumor Response | 80 |
| 7.1.2.1. | Target Lesions | 80 |
| 7.1.2.2. | Non-Target Lesions | 80 |
| 7.1.2.3. | Determination of Overall Response. | 81 |
| 8. | ASSESSMENT OF SAFETY | 82 |
| 8.1. | Safety Parameters | 82 |
| 8.1.1. | Laboratory Safety Assessments | 82 |
| 8.1.1.1. | Hematology, Serum Chemistry, Coagulation, Pregnancy Test | 82 |
| 8.1.1.2. | Urinalysis | 82 |
| 8.1.1.3. | Physical Examination | 83 |
| 8.1.1.4. | Vital Signs | 83 |
| 8.1.1.5. | Performance Status | 83 |
| 8.1.1.6. | ECG | 83 |
| 8.2. | Adverse Events | 83 |
| 8.2.1. | Definition of Adverse Event | 83 |
| 8.2.2. | Serious Adverse Events | 84 |
| 8.2.2.1. | Hospitalization | 85 |
| 8.3. | Reporting Adverse Events | 86 |
| 8.3.1. | Eliciting Adverse Event Information | 86 |
| 8.3.2. | Adverse Event Reporting Period | 86 |
| 8.3.3. | Reporting Requirements | 86 |

| 8.3.4. | Recording Adverse Events in the Case Report Forms | 87 |
|---|---|---|
| 8.3.5. | Grading of Adverse Event Severity | 88 |
| 8.3.6. | Relationship to TRC105 Study Drug/Pazopanib | 88 |
| 8.3.7. | Expectedness | 88 |
| 8.3.8. | Exposure in Utero. | 89 |
| 8.3.9. | Follow-up of Unresolved Adverse Events | 90 |
| 8.4. | Safety Monitoring | 90 |
| 9. | OTHER ASSESSMENTS | 91 |
| 9.1. | Other Laboratory Assessments | 91 |
| 9.1.1. | Pharmacokinetics | 91 |
| 9.1.1.1. | TRC105 Peak and Trough Concentration (Phase 1b dose levels -1, 1, 2 and expanded cohort 1 and angiosarcoma cohort 2) | 91 |
| 9.1.1.2. | TRC105 and Pazopanib Trough Concentration (Phase 1b dose levels 3, expanded cohort 2 and Phase 2 including angiosarcoma cohort 1) | 91 |
| 9.1.2. | TRC105 Immunogenicity | 91 |
| 9.1.3. | Protein Biomarkers | 91 |
| 9.1.4. | Archival Tumor Specimens | 92 |
| 10. | STATISTICS | 93 |
| 10.1. | Statistical Design/Sample Size | 93 |
| 10.1.1. | Phase 1b Statistical Design/Sample Size | 93 |
| 10.1.1.1. | Definition of Analyzed Study Populations | 93 |
| 10.1.2. | Phase 2 Statistical Design/Sample Size. | 94 |
| 10.1.2.1. | Definition of Analyzed Study Populations | 94 |
| 10.2. | Data Analysis | 95 |
| 10.2.1. | Analysis of Primary Objective | 95 |
| 10.2.1.1. | Phase 1b Analysis of Primary Objective | 95 |
| 10.2.1.2. | Phase 2 Analysis of Primary Objective | 95 |
| 10.2.2. | Analysis of Pharmacokinetics | 95 |
| 10.2.3. | Objective Response | 96 |
| 10.2.4. | Analysis of Protein Biomarkers | 96 |
| 10.2.5. | Analysis of Immunogenicity | 96 |
| 10.2.6. | Analysis of Archival Tumor Tissue | 96 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 97 |

| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 98 |
|---|---|---|
| 13. | ETHICS | 99 |
| 13.1. | Institutional Review Board (IRB)/Independent Ethics Committee (IEC) | 99 |
| 13.2. | Ethical Conduct of the Study | 99 |
| 13.3. | Written Informed Consent | 99 |
| 13.4. | Patient Compensation | 99 |
| 14. | DATA HANDLING AND RECORDKEEPING | 100 |
| 14.1. | Inspection of Records | 100 |
| 14.2. | Retention of Records | 100 |
| 15. | DEFINITION OF END OF TRIAL | 101 |
| 15.1. | End of Trial in all Participating Countries | 101 |
| 15.2. | End of Trial in a Member State | 101 |
| 15.3. | TRACON Discontinuation Criteria | 101 |
| 16. | PUBLICATION OF TRIAL RESULTS | 102 |
| 17. | FINANCING AND INSURANCE | 103 |
| 18. | INVESTIGATOR PROTOCOL AGREEMENT: 105SAR101 | 104 |
| 19. | REFERENCES | 105 |
| 20. | APPENDICES | 110 |
| 20.1. | Appendix 1: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) | 110 |
| 20.2. | Appendix 2: ECOG Performance Status | 111 |
| | LIST OF TABLES | |
| Table 1: | Emergency Contact Information | 2 |
| Table 2: | Abbreviations and Specialist Terms | |
| Table 3: | Dose Limiting Toxicity Definition and Criteria | 43 |
| Table 4: | Schedule of Assessments Phase 1b Dose Levels -1, 1, 2 & Expanded Cohort 1 | |
| Table 5: | Schedule of Assessments Phase 1b Dose Levels 3and Expanded Cohort 2 | |
| Table 6: | Schedule of Assessments Phase 2 Soft Tissue Sarcoma | 56 |
| Table 7: | Schedule of Assessments Phase 2 Angiosarcoma Cohorts 1 &2 | 59 |
| Table 8: | TRC105 10 mg/kg Weekly Ideal Dosing Schema | 70 |

# 105SAR101 Protocol Amendment #7, July 22, 2016

| Table 9: | TRC105 15 mg/kg Every Two Weeks Ideal Dosing Schema (Ph1b Dose Level 3) | 71 |
|---|---|---|
| Table 10: | Allowable TRC105 Dose Modifications | 72 |
| Table 11: | TRC105 dosing after Dose Delay (with no split dosing) | 73 |
| Table 12: | TRC105 Dosing after Dose Delay (with split dosing) | 73 |
| Table 13: | Management of TRC105 Infusion Reactions | 74 |
| Table 14: | Strong CYP3A4 Inducers and Inhibitors <sup>a</sup> | 78 |
| Table 15: | Response Evaluation Criteria in Solid Tumors | 81 |
| Table 16: | Adverse Event Grading. | 88 |
| Table 17: | Probability of Escalation to the Next Dose for Each True Underlying DLT Rate at a Dose Level | 93 |
| Table 18: | Probability of Failing to Observe True Underlying DLT Rate at a Dose Level | 93 |
| | LIST OF FIGURES | |
| Figure 1: S | Single-Dose and Multiple-Dose Pharmacokinetic Data from Study 105ST101 | 27 |

**Table 2:** Abbreviations and Specialist Terms

| Abbreviation or specialist term | Explanation |
|---|---|
| ADCC | Antibody-Dependent Cell-mediated Cytotoxicity |
| AE | Adverse Event |
| AFP | Alpha Fetoprotein |
| AIDS | Acquired Immunodeficiency Syndrome |
| ALKs | Activin receptor-Like Kinases |
| ALT | Alanine Aminotransferase |
| ANC | Absolute Neutrophil Count |
| APA | Anti-Product Antibody |
| AST | Aspartate Aminotransferase |
| AUC | Area Under the Curve |
| AUC <sub>last</sub> | Time of Last Measurable Concentration of Area Under the Curve |
| BALB/c mice | Mouse Strain |
| BMP | Bone Morphogenic Protein |
| BUN | Blood Urea Nitrogen |
| CABG | Coronary Artery Bypass Graft |
| CBC | Complete Blood Count |
| CEA | Carcinoembryonic Antigen |
| СНОР | Cyclophosphamide Hydroxydaunomycin Oncovin® Prednisone |
| CL | Clearance |
| C <sub>max</sub> | Maximum Serum Concentration |
| CPA | Cyclophosphamide |
| CR | Complete Response |
| CRF | Case Report Form |
| CT | Computed Tomography |
| CTC | Common Terminology Criteria |
| dL | Deciliter |
| DLT | Dose Limiting Toxicity |
| DVT | Deep Vein Thrombosis |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| ECM | Extracellular Matrix |
| EGFR | Epidermal Growth Factor Receptor |
| ELISA | Enzyme-Linked ImmunoSorbent Assay |
| EOS | End of Study |
| FDA | Food and Drug Administration |
| FGF | Fibroblast Growth Factor |
| FU | Fluorouracil |
| g | Gram |
| GOG | Gynecologic Oncology Group |
| GCP | Good Clinical Practice |
| GIST | Gastrointestinal Stromal Tumor |
| HACA | Human Anti-Chimeric Antibodies |
| HAMA | Human Anti-Murine Antibodies |
| Her-2 | Human epidermal growth factor receptor 2 |

# 105SAR101 Protocol Amendment #7, July 22, 2016

| HHT-1 | Hereditary Hemorrhagic Telangiectasia Type 1 |
|----------------|-----------------------------------------------------|
| HIF-1-α | Hypoxia-Inducible Factor-1-α |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | Human Immunodeficiency Virus |
| HRA | Health Regulatory Authority |
| HUVECs | Human Umbilical Vein Endothelial Cells |
| ICH | International Conference on Harmonization |
| ID | Identification |
| IEC | Independent Ethics Committee |
| IgG | Immunoglobulin G |
| IgM | Immunoglobulin M |
| IL | Interleukin |
| INR | International Normalized Ratio |
| IP | Intraperitoneal |
| IRB | Institutional Review Board |
| i.v. | Intravenous |
| K <sub>d</sub> | Avidity Binding Constant |
| kg | Kilogram |
| L | Liter |
| LDH | Lactate Dehydrogenase |
| LOQ | Limit of Quantification |
| μL | Microliter |
| Mg | Milligram |
| mL | Milliliter |
| MACA | Monkey Anti-Chimeric Antibody |
| MAMA | Monkey Anti-Murine Antibody |
| MI | Myocardial Infarction |
| mm | Millimeter |
| MRI | Magnetic Resonance Imaging |
| MTD | Maximum Tolerated Dose |
| NCI | National Cancer Institute |
| NCIC | National Cancer Institute of Canada |
| ng | Nanogram |
| NHP | Nonhuman Primate |
| NOAEL | No Adverse Effect Level |
| PBS | Phosphate-Buffered Saline |
| PD | Progressive Disease |
| PDGF | Platelet Derived Growth Factor |
| PDGFR | Platelet Derived Growth Factor Receptor |
| PIGF | Placental Growth Factor |
| pM | Picomolar |
| PR | Partial Response |
| PSA | Prostate Specific Antigen |
| PTCA | Percutaneous Transluminal Coronary Angioplasty |
| PTT | Partial Thromboplastin Time |
| QA | Quality assurance |
| RCC | Renal cell carcinoma |

# 105SAR101 Protocol Amendment #7, July 22, 2016

| RECIST | Response Evaluation Criteria in Solid Tumors |
|---|---|
| SAE | Serious Adverse Event |
| sCD105 | Soluble CD105/endoglin |
| SCID | Severe Combined Immunodeficient |
| SD | Stable Disease |
| SGOT | Serum Glutamic Oxaloacetic Transaminase |
| SGPT | Serum Glutamic Pyruvic Transaminase |
| SN6j | Murine parent antibody of TRC105 |
| sVEGFR2 | Soluble VEGF Receptor 2 |
| TGF-β | Transforming Growth Factor |
| TSH | Thyroid Stimulating Hormone |
| ULN | Upper Limit of Normal |
| US | United States of America |
| VEGF | Vascular Endothelial Growth Factor |
| VEGFR | Vascular Endothelial Growth Factor Receptor |
| VEGFR TKI | Vascular Endothelial Growth Factor Receptor Tyrosine Kinase Inhibitor |

# 2. BACKGROUND

# 2.1. Angiogenesis and Cancer

Angiogenesis is required for the survival and growth of solid cancers [2, 3]. It is generally accepted that solid cancers have two phases, an avascular phase and a vascular phase [3]. During the initial avascular phase, tumors exist as small aggregates of malignant cells supported by simple diffusion of oxygen and nutrients. The progressive growth of solid cancers beyond clinically occult sizes requires the continuous formation of new blood vessels, a process known as tumor angiogenesis. Tumor growth and metastasis require angiogenesis. Therefore, inhibition of tumor angiogenesis and selective inhibition of the tumor vasculature represent potentially effective strategies for the prevention and treatment of solid cancers.

Therapies that are directed against targets implicated in the development of tumor angiogenesis are attractive for many reasons. First, except for female reproduction and wound healing, angiogenesis in adults is generally part of a pathologic process such as tumor growth or choroidal neovascularization. Second, treatments that interrupt tumor angiogenesis should apply broadly to all solid cancers. Third, angiogenic targets are present in the plasma or on endothelial cells themselves. These targets are readily accessible to antibody treatments, in contrast to targets expressed within tumors that are more difficult for antibodies to access. Fourth, angiogenic targets on vascular endothelial cells are less prone to genetic mutation than targets expressed by genetically unstable cancer cells. As a result, development of resistance may be more predictable for agents that target endothelial cell functions than for those targeting cancer cells.

Indeed, agents that target pathways required for tumor angiogenesis have an important role in the therapy of cancer patients. The monoclonal antibody bevacizumab, which binds to the angiogenic cytokine VEGF, significantly prolongs overall survival for patients with advanced colorectal cancer or non-small cell lung cancer when added to standard chemotherapy regimens [4, 5]. Bevacizumab is also effective therapy for renal cell cancer and malignant glioma [6-8]. Orally available small molecule VEGF inhibitors include sunitinib, sorafenib, pazopanib, and axitinib which have been shown to prolong survival in patients with metastatic renal cell cancer, hepatocellular cancer, colorectal cancer, and sarcoma [9-12].

### 2.1.1. Angiogenesis and Advanced Soft Tissue Sarcoma

Sarcomas are rare tumors that originate from mesenchymal tissues (e.g., bone, cartilage, fat and muscle). In the United States, the incidence of bone and soft tissue sarcomas is approximately 13,000 new cases per year, leading to more than 5,000 deaths annually [13]. According to the WHO classification of 2002, over 70 different types of sarcoma have been described [14]. Localized tumors are curable but patients with metastatic disease have a median survival of approximately 12 months. Standard systemic chemotherapy regimens are poorly tolerated and of limited usefulness with response rates in the range of 10-40% [15].

Recently, the VEGFR TKI pazopanib was approved in patients with advanced soft tissue sarcoma who have received prior chemotherapy. Pazopanib improved progression free survival in chemotherapy refractory patients compared to placebo (PFS of 4.6 months with pazopanib versus 1.6 months with placebo) and was generally well tolerated, with the most common

adverse events seen at higher levels than in patients treated with placebo being fatigue, diarrhea, nausea, weight decreased and hypertension.

The short time to progression following pazopanib treatment emphasizes that sarcoma is a disease in need of more effective and well tolerated treatment options. CD105 (endoglin) is a membrane receptor expressed by the proliferating endothelium in sarcoma vasculature as well as sarcomatous cells that may be a suitable target for the treatment of sarcoma.

CD105 is a marker of mesenchymal stem cells, the normal cell type from which sarcomas originate [16, 17]. CD105-expressing sarcomas are relatively frequent and express CD105 at higher density than carcinoma cell lines. In one report, high surface expression of CD105 by whole cell flow cytometry was seen in 7 of 8 sarcoma cell lines and only 4 of 16 carcinoma cell lines [18]. Moreover, the level of CD105 expression correlated with proliferative capacity, and the addition of neutralizing anti-CD105 antibodies reversed the increase in proliferation.

CD105 expression in human sarcoma tumor tissue has been reported by several groups. Gromova et al found CD105 on 26 of 49 human gastrointestinal stromal tumors (GIST), and higher expression correlated with more aggressive tumors and high risk disease [19]. They concluded that CD105 deserves consideration as a target for therapy of GIST. CD105 expression on Ewing's sarcoma has also been reported, and high expression correlates with poor survival. Moreover, CD105 knockdown reversed the increased tumor cell plasticity, invasiveness, and anchorage independent growth associated with CD105 expression [20]. Other CD105-expressing sarcomas identified in the literature include angiosarcoma, osteosarcoma, leiomyosarcoma, malignant fibrous histiocytoma (undifferentiated pleomorphic sarcoma), Kaposi's sarcoma, Wilms tumor, and chondrosarcoma [21-25].

In addition to endothelial cells and sarcoma cells, CD105 is found on the surface of benign stromal cells present in sarcomatous tumors. Morozov et al identified a CD105-positive sarcoma-derived benign mesenchymal stromal cell (SDBMSC) present in primary sarcoma cultures [23]. These cells express pericyte markers and cooperate with endothelial cells in vascular tube formation assays. In coculture experiments, SDBMSCs as well as normal CD105-positive human pericytes markedly stimulated the growth of sarcoma cell lines.

# 2.1.2. CD105 and Angiogenesis

CD105 (endoglin) is a homodimeric cell membrane glycoprotein that was initially identified as a human leukemia-associated antigen [26] and later also found on endothelial cells [27, 28]. CD105 is a TGF-β coreceptor that is essential for angiogenesis [29, 30] and CD105 is strongly expressed on the proliferating vascular endothelium of solid tumors [28, 31]. All of these properties make CD105 an attractive target for the antiangiogenic therapy of cancer [32]. Vascular targeted therapy may more effectively address large established tumors than conventional antiangiogenic therapy such as anti-VEGF therapy [33]. In animal models, CD105 targeted therapy has demonstrated both vascular targeting effects and antiangiogenic effects by inducing regression of established tumors as well as by preventing new tumor formation and inhibiting expansion of existing tumors [28, 34-37]. Therefore, CD105 offers a novel alternative target relative to the VEGF inhibitors currently available for antiangiogenesis therapy.

CD105 acts to modulate signaling of multiple kinase receptor complexes of the TGF-β superfamily, including TGF-β receptors, activin receptor-like kinases (ALKs) and activin

receptors [38]. In the absence of CD105, activation of TGF-β receptors results in phosphorylation of SMAD proteins that inhibit endothelial cell growth. However, activation of CD105 by TGF-β modulates SMAD protein phosphorylation. The end result is release of the growth inhibitory effects of TGF-β receptor activation on endothelium. Not surprisingly, prevention of CD105 activation by anti-CD105 antibody acts synergistically with TGF-β to inhibit endothelial cell growth [39]. Similarly, CD105 acts in concert with the bone morphogenic protein (BMP) receptor to phosphorylate SMAD 1 and 5 in response to binding BMP 9 and 10, to activate endothelium [40].

CD105 expression is required for endothelial cell proliferation, and CD105 is upregulated in the setting of hypoxia through the induction of hypoxia-inducible factor-1-α (HIF-1-α) [41, 42]. CD105 has also been shown to protect hypoxic cells from apoptosis [43]. The expression of CD105 by endothelial cells is essential for the development of new vasculature. Targeted inactivation (knockout) of murine CD105 results in defective vascular development. Mice lacking CD105 die *in utero* from defective vascular development by gestational day 11 [30].

CD105 is critical for normal human blood vessel development [44]. CD105 haplotype insufficiency causes a well-described syndrome known as hereditary hemorrhagic telangiectasia type 1 (HHT-1 or Osler-Weber-Rendu Syndrome). HHT-1 is a rare autosomal dominant genetic disorder characterized by localized angiodysplasia involving the nasal, buccal, gastrointestinal mucosa and skin microvasculature. Angiodysplasia also occurs in vessels from internal organs including the lungs, liver and brain [45]. The genotype is manifested *in utero*, but the phenotype does not become apparent for many years following birth. Affected patients commonly present with epistaxis in the second decade of life. The phenotype of this disorder is limited to vascular effects, indicating the specific role of CD105 in the vasculature [46].

CD105 is highly expressed on the proliferating endothelial cells of tumor vessels including lung, breast, colorectal, gastric, liver, endometrial, renal cell, head and neck, and ovarian cancers. In adults, CD105 expression is limited to vascular endothelial cells and proerythroblasts, a red blood cell precursor [47].

CD105 expression is a prognostic factor in solid tumor patients. High microvessel density of CD105-positive vessels has been correlated with poor prognosis in clinical studies of breast cancer [48, 49], lung cancer [50], prostate cancer [51, 52], colorectal cancer [53, 54], ovarian cancer [55, 56], gastric cancer [57], endometrial cancer [58], astrocytic brain tumors [59], hepatocellular carcinoma [60], esophageal adenocarcinoma [61], and head and neck cancer [62, 63].

Plasma CD105 levels are prognostic in retrospective studies of cancer patients. In one study, the mean plasma CD105 concentration in 76 patients with colorectal cancer was 4-fold higher than the mean value in 40 healthy subjects without cancer [53]. In the study, a positive correlation was observed between plasma CD105 concentration and stage of disease.

Importantly, CD105 expression is upregulated in tumor endothelial cells following inhibition of the VEGF pathway. CD105 expression increased more than 2-fold in human pancreatic cancers grown in mice treated with an antibody that binds VEGF [64]. As well, treatment of human bladder cancers grown in mice with an antibody that blocks activation of the VEGF receptor increased CD105 expression within the core tumor vasculature [65].

TRC105 is a novel IgG1 that binds CD105 with high avidity. Recent studies at Duke University explored the *in vitro* effects of dual angiogenesis inhibition using bevacizumab and TRC105 in human umbilical vein endothelial cells (HUVEC). Combination therapy was found to be more potent in decreasing HUVEC proliferation, migration, and tubular network formation than bevacizumab or TRC105 treatment alone (manuscript in preparation). Furthermore, TRC105 induced apoptosis in HUVEC, and promotes SMAD2/3 phosphorylation while inhibiting SMAD1/5/8 signaling, thereby inhibiting angiogenesis in response to VEGF and basic FGF [40]. Finally, antibody to mouse CD105 potentiates the activity of multitargeted kinase inhibition that targets the VEGFR-2, in mouse bearing cancer grafts (manuscript in preparation). For these reasons, CD105 blockade using TRC105 in combination with VEGF inhibition by pazopanib may provide greater clinical benefit than would be seen with either drug alone.

# 2.2. TRC105 Background

TRC105 is a genetically engineered human/murine chimeric monoclonal antibody directed against human CD105 [66], a growth proliferation receptor found on the surface of normal and proliferating endothelial cells [28, 34, 42].

The antibody is an IgG1 kappa immunoglobulin containing murine variable region sequences and human constant region sequences [66]. TRC105 has an approximate molecular weight of 148 kDa. TRC105 has a binding avidity for human CD105 of approximately 5 pM. TRC105 is formulated as a phosphate-buffered saline (PBS) solution at a concentration of 7 mg/mL.

SN6j, the murine parent antibody of TRC105, binds to human umbilical vein endothelial cells (HUVECs) with nearly identical avidity as TRC105. SN6j has been shown to bind the tumor vasculature of malignant tissues including breast, colon, rectum, kidney and lung cancers and to inhibit the growth of tumor xenografts [35]. Reactivity with tumor tissues is restricted to the tumor endothelium, as CD105 is not generally expressed on epithelial tumor cells [34]. TRC105 induces ADCC on proliferating HUVECs at low conentrations and induces apoptosis and growth inhibition at higher concentrations.

### **2.2.1. Studies with TRC105**

Several studies with TRC105 are underway or have been completed. An open-label, phase 1, multicenter study of TRC105 (Study 105ST101) enrolled fifty patients, who were treated until disease progression with TRC105 at 0.01-15 mg/kg/q2wk or 10-15 mg/kg/wk. Studies of TRC105 in prostate, bladder, and ovarian cancer, phase 1b study of TRC105 in combination with bevacizumab and a phase 1b study of TRC105 in combination with capecitabine in breast cancer have also been completed. Ongoing studies include a phase 1b study of TRC105 in combination with sorafenib in liver cancer, a phase 1b/2 study of TRC105 in combination with axitinib in renal cell carcinoma, and phase 2 studies of TRC105 monotherapy in liver cancer and in combination with bevacizumab in glioblastoma multiforme (2 studies) and renal cell carcinoma.

### **2.2.1.1. 105ST101 Phase 1 Monotherapy**

# 2.2.1.1.1. 105ST101 Phase 1 Monotherapy Pharmacokinetics

In Study 105ST101, TRC105 pharmacokinetics were assessed on patients enrolled at doses up to 15 mg/kg weekly. Circulating TRC105 was not measurable above the lower limit of quantitation

of the assay (78 ng/mL) in patients receiving doses below 0.3 mg/kg. TRC105 was measurable above the target concentration based on preclinical data (200 ng/mL) for 4 hours at 0.3 mg/kg, 1 day at 1 mg/kg, 5 days at 3 mg/kg, 7 days at 10 mg/kg TRC105 dosed every two weeks. Serum concentrations expected to saturate CD105 binding sites (≥ 200 ng/mL) were achieved continuously at 15 mg/kg q2wk and 10 mg/kg weekly, and TRC105 accumulated at 15 mg/kg weekly (Figure 1).

Figure 1: Single-Dose and Multiple-Dose Pharmacokinetic Data from Study 105ST101



### 2.2.1.1.2. 105ST101 Phase 1 Monotherapy Immunogenicity

In Study 105ST101, serum samples for evaluation of TRC105 immunogenicity, including HAMA and HACA, were collected pre-dose on day 1 of each 28 day cycle, at the end of study, and then at 4 and 12 weeks after the end of study visit.

HAMA and HACA data are available from the phase 1 monotherapy TRC105 trial. Neither HAMA nor HACA were detected in patients treated with CHO-produced TRC105, which will be used for all future clinical trials, including this study.

# 2.2.1.1.3. 105ST101 Phase 1 Monotherapy Safety

A total of 50 patients were treated on Study 105ST101 with escalating doses of TRC105 at 0.01, 0.03, 0.1, 0.3, 1, 3, 10 and 15 mg/kg every two weeks and then 10 and 15 mg/kg weekly. Dose escalation proceeded stepwise until the top dose was reached. The maximum tolerated dose was exceeded at 15 mg/kg weekly and the recommended phase 2 dose of TRC105 was therefore determined to be 10 mg/kg weekly or 15 mg/kg every 2 weeks. Three of 4 patients at 15 mg/kg weekly developed grade 3 hypoproliferative anemia (without leucopenia or thrombocytopenia) in cycle 2, and one of the three progressed to grade 4 in cycle 3. Anemia was associated with accumulation of TRC105 and characterized by a low reticulocyte production index. Additional laboratory and clinical evaluations excluded common causes of anemia including blood loss, hemolysis, plasma volume expansion, inadequate erythropoietin, iron deficiency, and vitamin B-12 or folate deficiency. The anemia is believed to result from TRC105-mediated suppression of proerythroblasts, the only cells in the bone marrow known to express substantial levels of CD105 [47]. Anemia was reversible and manageable with dose reduction and standard supportive measures including erythropoietin and blood transfusion.

Infusion reactions, anemia, fatigue, epistaxis and headache were the most frequently observed adverse events considered related to TRC105. The majority of treatment-related adverse events were grade 1 or 2.

Infusion reactions, among the most common adverse events, were usually with the initial TRC105 dose and included one or more of the following signs or symptoms: rigors, bronchospasm, urticaria, hypertension, hypotension, tachycardia or bradycardia. Infusion reactions were initially reported at 1 mg/kg every 2 weeks for patients receiving TRC105 produced in NS0 cells without premedication. TRC105 produced in CHO cells was known to more potently engage ADCC *in vitro* than TRC105 produced in NS0 cells. Because of this, the initial dose level for patients receiving CHO-produced TRC105 was de-escalated to 0.3 mg/kg. Despite dose de-escalation, the first two patients at 0.3 mg/kg treated with CHO-produced TRC105 experienced grade 2 and grade 3 infusion reactions with the first dose in the absence of premedication. The protocol was therefore amended to require a glucocorticoids -based premedication regimen and extend the initial infusion duration from 1 to 4 hours.

The amendment mandating premedication and extended initial infusion duration successfully reduced the frequency and severity of infusion reactions and allowed dose escalation to continue. One additional patient who received CHO-produced TRC105 at 1 mg/kg developed a grade 3 infusion reaction with the third dose given over 2 hours. This patient had experienced a grade 2 infusion reaction when the dose was administered over 4 hours. In all three patients with grade 3 infusion reactions, TRC105 was not detectable in serum at the time of dosing, which allowed *de novo* binding of TRC105 to CD105 expressing endothelium within the vasculature. Grade 3 infusion reactions were not observed in patients dosed at 10 or 15 mg/kg who maintained TRC105 serum levels known to saturate CD105 binding sites for the full dosing interval. At dose levels where continuous TRC105 serum levels were achieved, glucocorticoids were safely discontinued and the infusion duration reduced to 1 hour.

Three patients developed grade 1 cutaneous telangiectasia on the trunk early in the course of therapy, all at dose levels of 10 or 15 mg/kg weekly that resulted in continuous serum levels of TRC105 known to saturate CD105 sites on human endothelium. Grade 1 or 2 hemorrhage was reported, including intermittent postcoital vaginal bleeding (that also occurred prior to TRC105 treatment), epistaxis, and superficial gingival bleeding.

Grade 1 or 2 headaches were observed, mainly in patients treated at doses of TRC105 above 3 mg/kg. Headaches began the day following infusion and were generally manageable with acetaminophen. However, grade 2 headache in one patient at 15 mg/kg weekly prompted discontinuation prior to completion of the dose-limiting toxicity evaluation period. Fatigue was one of the more common adverse events attributable to TRC105 and was more prevalent at doses above 3 mg/kg.

One patient developed dose-limiting toxicity of grade 4 hemorrhage presenting as melena from a gastric ulcer within 5 days of the initial TRC105 infusion at 0.1 mg/kg. He discontinued TRC105 treatment, was transfused 2 units of packed red blood cells and the bleeding resolved with nonsurgical management by the time of upper endoscopy. Serious bleeding was not observed following protocol amendment to exclude patients with a history of peptic ulcer disease (unless healing was documented) and patients on ulcerogenic medications including non-steroidal anti-inflammatory drugs.

Classic toxicities associated with VEGF inhibition, including hypertension, proteinuria and thrombosis were not prominent. One patient with recurrent anal cancer treated at 0.1 mg/kg developed proteinuria considered possibly related to TRC105, but proteinuria was also noted prior to TRC105 dosing. Transient hypertension (156/112) without QT changes occurred in a single patient one day following infusion of 15 mg/kg, and was controlled by a single dose of oral antihypertensive medication. There were no arterial or venous thromboembolic events, nor gastrointestinal or other perforations in these patients.

### 2.2.1.1.4. 105ST101 Phase 1 Monotherapy Efficacy

In study 105ST101 stable disease  $\geq 2$  months was observed in 21 of 45 patients (47%) and stable disease  $\geq 4$  months in 6 of 44 patients (14%). Decreases in CEA, PSA, or CA-125 were noted in 7 of 21 patients (33%) and a global decrease in key angiogenic biomarkers was observed with treatment. One patient with castrate-refractory prostate cancer remains on TRC105 treatment after 6 years at a TRC105 dose of 0.01 mg/kg every 2 weeks. He has an ongoing complete PSA response, with resolution of bone pain and bone scan normalization. One patient with metastatic carcinosarcoma, manifested decreased tumor burden on computerized tomographic scanning and maintained stable disease for 20 months on therapy. The latter is especially notable when one considers that this patient had received three prior treatments -- carboplatin + paclitaxel for 4 months, anastrozole for 8 months, and ifosfamide for 2 months -- and had manifested tumor progression on each. In effect, TRC105 provided the most favorable clinical outcome and did so as a fourth-line therapy.

# 2.2.1.2. Phase 1b 105ST102 Study with Bevacizumab

# **2.2.1.2.1. 105ST102 Summary of Safety**

Administration of TRC105 at a dose of 3 mg/kg weekly in combination with bevacizumab was well tolerated by three patients without the development of dose limiting toxicity (DLT) and dose escalation occurred per the protocol to cohort 2 (6 mg/kg TR105 weekly). However, the concurrent administration of 6 mg/kg TRC105 and bevacizumab on day 1 resulted in the development of moderate or severe headaches (including two grade 3 headaches) in four of five treated patients. The 6 mg/kg dose of TRC105 was tolerated when the initial TRC105 dose was delayed one week following bevacizumab dosing at 10 mg/kg every two weeks. Tolerability was further improved when the initial dose of TRC105 was given over two days during the first week of TRC105 dosing, and dose escalation proceeded to the recommended phase 2 dose of 10 mg/kg TRC105 weekly. At the recommended phase 2 dose of both drugs (10 mg/kg), TRC105 serum concentration were present above target concentration continuously and immunogenicity was rarely observed.

A total of 38 patients were dosed on study across six cohorts and four dose levels. Other than headaches that were mitigated by adjusting the dosing schedule of TRC105, the combination of TRC105 and bevacizumab was well tolerated. Two patients experienced grade 3 serious adverse suspected events as described below. Most adverse events were graded as 1 or 2 and Grade 4 and 5 suspected adverse events were not observed. Grade 3 suspected adverse reactions included anemia (the dose limiting toxicity of TRC105 established as a single agent; 9 patients), headache (4 patients; three of which occurred prior to adjusting the schedule of TRC105), fatigue (2 patients), brain abscess (1 patient), infusion reaction (in a patient dosed at 6 mg/kg), and decreased appetite (1 patient). Headache was the most common suspected adverse event and occurred in 31 patients (86.1%); three patients (7.9%) experienced migraine headaches (two of grade 1 and one of grade 2 severity). Headaches were treated with triptans and NSAIDs.

Two patients experienced serious adverse suspected events as described below. One of the grade 3 headaches (in a patient dosed at 8 mg/kg without splitting the initial TRC105 dose over two days) resulted in hospitalization and patient discontinuation. One patient dosed at 10 mg/kg of TRC105 experienced a serious suspected event of grade 3 brain abscess. Serious adverse events, considered unrelated to TRC105 treatment, included: grade 3 pneumonia and subsequent grade 4 MRSA sepsis that was complicated by a non Q-wave myocardial infarction during a period of hemodynamic instability while hospitalized; grade 3 ileus at the time of symptomatic disease progression; grade 5 disease progression; grade 3 left foot cellulitis; grade 3 recurrent pneumothorax; grade 3 small bowel obstruction; grade 4 urosepsis.

At least one sign of the triad of epistaxis, gingival bleeding and telangiectasia, reflecting vascular ectasia characteristic of the Osler-Weber-Rendu syndrome of endoglin haplotype insufficiency (i.e., an autosomal dominant genetic disorder of heterozygous endoglin expression) was observed frequently. One of these signs or symptoms (of grade 1 or 2 severity) was noted in one of three patients treated at 3 mg/kg, four of eight patients treated at 6 mg/kg, four of eight patients treated at 8 mg/kg and in all nineteen patients treated at 10 mg/kg of TRC105, generally within the first month of dosing. These signs and symptoms are an expected pharmacologic effects of TRC105 binding to the endoglin receptor (i.e., they are characteristic of the Osler-Weber-Rendu syndrome, that is caused by endoglin haploinsufficiency), and were also observed routinely

within the first month of dosing of 10 mg/kg weekly in the single agent TRC105 dose escalation study.

Infusion reactions were, as expected, more notable at lower doses, and were rare at the MTD of TRC105 of 10 mg/kg, when TRC105 serum concentrations were maintained continuously. Two of nineteen patients (10%) dosed with 10 mg/kg of TRC105 each experienced a single infusion reaction of grade 2 severity, both with the initial dose of TRC105, that required a brief interruption of the infusion prior to completion of the scheduled dose.

Clinically significant anemia was not reported in patients dosed with 3 mg/kg or 6 mg/kg of TRC105, was reported in three of seven patients (43%; all grade 3) dosed with 8 mg/kg of TRC105, and was observed in nine of 19 (47%; three of grade 2 and six of grade 3 severity) of patients dosed with 10 mg/kg of TRC105. Anemia prompted transfusion of packed red blood cells in 10 patients and growth factors were used in five patients.

Other, less frequent, suspected adverse reactions included hypothyroidism, periorbital edema (which was generally noted prior to splitting the initial dose of TRC105), gingival pain, nausea, oral pain, vomiting, edema, decreased appetite, dyspnea, nasal congestion, rash and flushing.

Other adverse events characteristic of each individual drug were not increased in frequency or severity when the two drugs were administered together. Of note, the concurrent administration of bevacizumab and TRC105 did not potentiate the known toxicities of bevacizumab of hypertension, hemorrhage (including tumor-associated hemorrhage, and pulmonary hemorrhage or hemoptysis), or proteinuria. Reversible posterior leukoencephalopathy syndrome (RPLS), congestive heart failure, fistulae, gastrointestinal perforation impaired wound healing, and arterial thromboembolic events, were not observed.

Notably, hypertension and proteinuira, known adverse events of bevacizumab, were rarely observed when bevacizumab was given with TRC105. Mild and transient clinically significant hypertension or blood pressure increases were observed in five patients (13%; grade 3 in one case (prior to dosing with study drugs) and grade 2 in four cases) and mild transient proteinuria was observed in two patients (5%; both grade 2).

### **2.2.1.2.2. 105ST102 Summary of Efficacy**

The combination of TRC105 and bevacizumab was active in patients with advanced refractory cancer who had progressed on prior bevacizumab or other VEGF inhibitor treatment. Thirty-three patients had measurable disease (31 patients) or evaluable disease (2 patients) at baseline and received at least one follow up scan and were evaluable for the primary efficacy outcome of ORR by RECIST 1.1. Eighteen patients with measureable disease (58%) had a best response of stable disease or partial response. Two patients (6%), both of whom had been treated with bevacizumab and chemotherapy prior to study entry and were then treated at the top dose level of TRC105 and bevacizumab, had RECIST 1.1- defined partial responses, including one patient with colorectal cancer who continues on treatment for more than 24 months. A total of 14 patients (45%) had decreases in overall tumor burden, of whom 10 received prior VEGF inhibitor treatment (usually bevacizumab with chemotherapy). Notably, the duration of treatment with TRC105 and bevacizumab of six patients (19% of those with measureable disease) exceeded the duration of treatment of the most recent treatment regimen containing a VEGF inhibitor (i.e., VEGFR TKI or bevacizumab), received prior to study entry. These six

patients had decreases in tumor burden and several were responders by Choi criteria or RECIST. Time to progression ranged from 0 to 437+ days. Reductions in tumor markers ranging from 5% to 85% were observed in 15 of 28 (54%) patients with relevant tumor markers. Three patients demonstrated clinical benefit throughout the study (patient 10038102 at cycle 12 day 22, patient 10018106 at cycle 7 day 22 and patient 10028101 at cycle 17 day 1); two of them continue to receive treatment under a continuation protocol (105CON101).

# 2.2.1.3. Phase 1b 105RC101 Study with Axitinib

All eighteen planned patients have been treated in the phase 1 portion of a renal cell cancer study of TRC105 plus axitinib as of the time of this protocol amendment (3 at 8 mg/kg and 15 at 10 mg/kg). Patients have experienced expected TRC105 related adverse events of grade 2 infusion reaction and grade 1 epistaxis, gingival bleeding, headache, rash, and fatigue; and expected axitinib adverse events of grade 1-3 hypertension, grade 1 hand-foot syndrome and grade 1 proteinuria. Two patients dosed with TRC105 at 8 mg/kg plus axitinib developed grade 2 creatinine elevations that reversed with hydration. Adverse events characteristic of each drug were not increased in frequency or severity when both drugs were administered concurrently. Eight of 14 evaluable VEGFR TKI refractory patients demonstrated decreases in tumor burden ranging from 1.2% to 36% (including two partial responses per RECIST in the fourth line treatment setting in ongoing patients).

# 2.2.1.4. Phase 1b 105SAR101 Study with Pazopanib

A total of 18 patients have been treated in the phase 1b portion of this study of TRC105 in combination with pazopanib. Three patients received 8 mg/kg TRC105 weekly, and 15 patients received 10 mg/kg TRC105 weekly in combination with standard dose pazopanib (starting at 800 mg/daily for 28 days of repeating 28 day cycles) without the development of dose limiting toxicity. AEs have been predominantly grade 1 or 2 and have been consistent with the known adverse event profiles of TRC105 and pazopanib.

# 2.3. Study Rationale

Given the novel mechanism of action and safety profile in early phase clinical studies, including a completed study with bevacizumab and an ongoing study with axitinib, TRC105 is a logical therapy for use with pazopanib. Pazopanib inhibits angiogenesis through the inhibition of VEGFR tyrosine kinases. TRC105 is an antibody to CD105, an important angiogenic target on proliferating endothelial cells that is distinct from the VEGFR and upregulated following VGEF inhibition. TRC105 inhibits angiogenesis, tumor growth and metastases in preclinical models and complements the activity of bevacizumab and multi-kinase inhibitors that target the VEGFR. In a phase 1b study, the combination of TRC105 and bevacizumab produced radiographic reductions in tumor volume in bevacizumab refractory patients. Together, the use of TRC105 with pazopanib may result in more effective angiogenesis inhibition and improved clinical outcome beyond that seen with pazopanib alone in patients with advanced soft tissue sarcoma who have progressed following treatment with first line chemotherapy. Angiosarcoma has been shown to express CD105 directly on tumor tissue, in addition to the proliferating tumor vascular endothelial cells. Thus, this soft tissue sarcoma histologic subtype may have increased responsiveness to TRC105 administered as a single-agent.

This trial is a phase 1b/2a dose escalation study of pazopanib in combination with TRC105 in order to assess the safety and efficacy of CD105 blockade combined with the VEGFR TKI pazopanib. A standard "3+3" dose- escalation design of patients with advanced soft tissue sarcoma will be employed in the phase 1b portion, followed by a phase 2 portion to assess progression free survival (PFS) and overall response rate (ORR), safety, and correlative studies of expression of endoglin on tumor tissue and plasma angiogenic biomarkers. The purpose of the dose escalation portion is to determine the maximum tolerated dose (MTD) of TRC105 when given in combination with pazopanib and to determine the dose limiting toxicities. Patients included in the study will have advanced soft tissue sarcoma that has progressed following first line chemotherapy. The phase 2 angiosarcoma cohorts will evaluate TRC105 administered as a single-agent and in combination with pazopanib.

# 2.4. Population to be Studied

Patients with histologically confirmed advanced soft tissue sarcoma will be enrolled in this trial.

# 2.5. Potential Risks and Benefits to Human Patients

### 2.5.1. Potential Risks

### TRC105

Grade 3 anemia has occurred with TRC105 therapy at the recommended phase 2 dose. All patients treated with TRC105 should be monitored closely for anemia and treated appropriately, including the possibility of TRC105 dose reductions. Anemia may be caused by correctable mineral or vitamin deficiency. The anemia related to TRC105 is hypoproductive in nature and is reversible with interruption of treatment, transfusion, erythropoietin, and other interventions as appropriate.

Gastrointestinal hemorrhage has occurred with TRC105 therapy. Patients with active ulcer disease or risk factors for ulcer disease are excluded from this study.

Grade 1 and 2 cutaneous telangiectasia related to TRC105 occur early in the course of therapy and have been the source of gingival bleeding and epistaxis. Telangiectasia are also seen in patients with hereditary hemorrhagic telangiectasia (HHT), a disease of CD105 haplotype insufficiency. Patients with HHT are at risk of hemorrhage from abnormal blood vessels and this could be exacerbated by treatment with TRC105. Other contraindications to TRC105 therapy include a history of significant hemorrhage or tumors located in the central chest or another location where bleeding is associated with high morbidity. All patients treated with TRC105 should be monitored for signs of hemorrhage and the risks and benefits of drug treatment reevaluated in any patient with hemorrhage.

Premedication including the use of glucocorticoids is required prior to infusion of TRC105 to reduce the frequency and severity of infusion reactions. Infusion reactions following TRC105 dosing generally occur with the first TRC105 dose and include a grade 4 vasovagal reaction that resolved without sequellae. Signs and symptoms of TRC105 infusion reactions include hypertension, hypotension, dyspnea, bronchospasm, chills/rigors, chills, sweats, fever, nausea, tachycardia, bradycardia, EKG changes, flushing, urticaria, pruritus, and headache, generally of grade 1 and 2 severity. Potential infusion reactions seen with other therapeutic antibodies include

angioedema, asthenia, throat irritation, rhinitis, vomiting, joint pain, fatigue and neurologic disorders including inflammation of the spine and/or brain.

Hypersensitivity reactions with infusions are a potential risk for sensitized patients, and TRC105 should be used with caution in patients with known hypersensitivity to any component of the drug product. Host anti-TRC105 antibodies to the murine or human portions of CHO-produced TRC105 are rare. In general, the risk of immunogenicity to therapeutic chimeric antibodies is small (<10%) and the clinical significance of immunogenicity is not well defined. The current trial will collect serial blood samples for anti-product antibody concentrations to further characterize the immunogenicity of TRC105 and potential clinical implications.

Grade 3 cerebrovascular hemorrhage resulting in hemiparesis occurred in one patient with hepatocellular cancer who was thrombocytopenic (who entered the study with a platelet count of 60,000/uL) in a study of TRC105 with sorafenib. Patients must have a platelet count of > 100,000/uL to enter this study (see inclusion criteria). A grade 2 transient ischemic attack was reported in a study of TRC105 and pazopanib. Transient Grade 3 hepatic encephalopathy occurred in one patient with cirrhosis and hepatocellular carcinoma who received TRC105 in combination with sorafenib. Grade 3 pancreatitis was also observed in this study. Grade 5 intracranial hemorrhage occurred in one glioblastoma patient with markedly abnormal blood clotting parameters in a study of TRC105 with bevacizumab. A patient with glioblastoma developed temporary confusion and slurred speech following treatment with TRC105 and bevacizumab that required hospitalization for observation. Another patient with glioblastoma, who underwent resection and had a history of an abnormal collection of cerebral spinal fluid, developed a grade 2 cerebral spinal fluid leak. A third patient with glioblastoma with a history of recurrent meningitis developed recurrent grade 3 bacterial meningitis while treated with bevacizumab and TRC105.

Grade 3 myocardial infarction (non-Q wave infarct associated with hypertension following an infusion reaction) was observed in a patient with hepatocellular cancer following treatment with TRC105 that resolved without sequellae. In addition, a Grade 5 myocardial infarction occurred in a patient with coronary artery disease who received TRC105 in combination with sorafenib. Patients with evidence of active coronary artery disease are excluded from participation in this trial (see exclusion criteria).

Adult respiratory distress syndrome that required temporary intubation occurred in one patient who received TRC105 with pazopanib, from which the patient recovered. Of note, interstitial lung disease has been added as an adverse drug reaction and warning/precaution to the core safety information for pazopanib. Pneumothorax (collapsed lung) has been observed in trials of TRC105 administered with VEGF inhibitors in patients with lung metastases. In addition, pnemothorax was observed in one patient, also with lung metastases, receiving single-agent TRC105.

Infections have been observed rarely. Grade 3 infected lipoma/cyst was observed in a Phase 2 study of TRC105 as a single agent in patients with metastatic bladder cancer. Grade 3 orbital cellulitis and grade 3 brain abscess were observed in patients treated with TRC105 and bevacizumab and considered possibly related to TRC105. Grade 1 and 2 gingivitis including infection and ulceration has also been observed. Overall, infections have been observed in fewer

than 5% of patients and have largely been considered unrelated to treatment with TRC105. Reversible grade 3 colitis was reported in a patient treated with TRC105 and pazopanib.

Grade 1-3 headaches have been observed following TRC105 treatment, generally within hours following completion of the initial infusion. Headaches are throbbing in nature, are not associated with radiographic abnormalities, and have responded to treatment with non-steroidal anti-inflammatory agents and to triptans. Headaches were particularly common when TRC105 and bevacizumab were initially dosed on the same day and were ameliorated when TRC105 was dosed one week following bevacizumab dosing and given over two days during the initial week of dosing.

Nasal congestion and periorbital edema have been observed with TRC105 dosing, particularly when dosed in combination with bevacizumab. The edema has been transient in nature and treated with corticosteroids

Fatigue of grade 1- 3 severity has been reported following dosing with TRC105. Maculopapular rash and skin flushing of grade 1 and grade 2 severity have also been reported. A patient receiving treatment with TRC105 and sorafenib developed self-limited pancreatitis of grade 2 severity.

# **Pazopanib**

The most common adverse reactions in patients with advanced soft tissue sarcoma (≥20%) are fatigue, diarrhea, nausea, decreased weight, hypertension, decreased appetite, vomiting, tumor pain, hair color changes, musculoskeletal pain, headache, dysgeusia, dyspnea and skin hypopigmentation.

Further details are available in the package insert [67].

### Computed Tomography (CT) Scans

Patients will be exposed to a small amount of radiation as a result of the CT scans required in this study. This degree of exposure has not been associated with harmful health effects. In addition, the frequency of CT scans performed in this study is similar to the standard of care frequency. Patients with a medical contraindication to CT scans or known Iodinated contrast allergies may undergo MRI. There is minimal risk of MRI imaging in patients able to undergo this type of exam including very rare reports of gadolinium-induce nephrogenic systemic fibrosis in patients with poor renal function.

# Magnetic Resonance Imaging (MRI):

MRI is a noninvasive imaging test used to diagnose and evaluate medical conditions. MRI does not use radiation and there are no known harmful side-effects. However, MRI may cause anxiety for people due to the loud banging made by the machine and the confined space of the testing area. People with pacemakers, aneurysm clips, artificial heart valves, ear implants, or metal implants or foreign objects in their body are not permitted to have an MRI.

### Bone Scans:

A bone scan is a test that can find cancer that has spread to the bones. A bone scan can often find a problem days to months earlier than a regular X-ray test. During a bone scan, a radioactive substance called a tracer is injected into a vein in your arm. The tracer travels through your bloodstream and into your bones. Then a special camera takes pictures of the tracer in your bones. A bone scan poses no greater risk than do conventional X-ray procedures. The tracers used in a bone scan produce very little radiation exposure — less than half that of a CT scan.

# Venipuncture

Patients could also experience side effects from venipuncture for tests that will be done as part of this study including pain, tenderness or bruising at the site of collection, and rarely infection may occur at the spot where the needle is inserted.

### Other Risks

This study treatment may involve risks to unborn children therefore patients should not become pregnant or father a baby while participating in this study. Patients should not nurse while on this study. Women of childbearing potential must have a negative pregnancy test before taking part in this study. Patients will be asked to practice an effective method of birth control during participation in this study and for three months after the last treatment. The long term risk of infertility is unknown. Ovarian failure has been observed with other antiangiogenic agents.

### 2.5.2. Potential Benefits

TRC105 is an investigational product, and its efficacy has not been established. It is possible that the administration of TRC105 may result in clinical benefit (i.e., tumor response or prolonged stable disease).

# 2.6. Justification of the Dose, Schedule and Route of Administration of TRC105

### 2.6.1. Phase 1b Justification

The dose and schedule of TRC105 (8 mg/kg weekly up to 10 mg/kg weekly, 15 mg/kg every 2 weeks) for phase 1b were selected based on safety, pharmacokinetics and early evidence of activity in the phase 1 study of TRC105 for patients with solid tumors (Study 105ST101) and in the phase 1b study of TRC105 with bevacizumab. In phase 1, a weekly dose of 10 mg/kg and a dose of 15 mg/kg every two weeks were well tolerated and associated with clinical activity. Dose reduction was possible for treatment of anemia. Doses of 8 and 10 mg/kg TRC105 weekly were tolerated in combination with bevacizumab, pazopanib (dose levels 1 and 2 of this study) and axitinib and doses of TRC105 of 15 mg/kg every 2 weeks were tolerated in combination with sorafenib. Notably, while the initial schedule of TRC105 was adjusted to decrease the frequency of headaches observed with the combination of TRC105 and bevacizumab, there was no potentiation of life threatening toxicities associated with bevacizumab, nor potentiation of common VEGF inhibitor toxicities (e.g., hypertension and proteinuria).
Given the limited experience dosing TRC105 with VEGF inhibitors, it is possible that TRC105 toxicities will potentiate pazopanib toxicities, and vice versa. Therefore a TRC105 starting dose of 8 mg/kg weekly, which is 20% lower than the single-agent TRC105 MTD identified in the phase 1 single agent study and phase 1b study with bevacizumab, was selected. In addition a 6 mg/kg (-1) dose level has also been included and will be enrolled should 8 mg/kg of TRC105 in combination with pazopanib exceed the MTD. As an added precaution, the first dose of TRC105 will be delayed by 2 to 4 weeks following pazopanib dosing and administered over 2 days. In addition, pazopanib will be introduced at 800 mg and dose reduced based on patient tolerability over a two to four week period prior to the introduction of TRC105. This administration schedule will limit immediate  $C_{max}$  effects of the combination of two drugs that could result in toxicity.

In the phase 1b portion of the study, dose levels 1 and 2, TRC105 at its recommended phase 2 dose of 10 mg/kg given by weekly intravenous infusion was combined safely with pazopanib given at 800 mg p.o. once daily.

The phase 1b portion of the study will also evaluate TRC105 administered every two weeks at 15 mg/kg starting at cycle 2, following initial dosing with 10 mg/kg weekly for the initial 28 day cycle. TRC105 will be given in combination with pazopanib 800 mg daily. In the phase 1 study of single-agent TRC105 (105ST101), TRC105 15 mg/kg administered every 2 weeks was well tolerated and resulted in continuous serum concentrations known to saturate CD105 binding sites on proliferating endothelium. An alternative dosing schedule of every 2 weeks TRC105 treatment in combination with pazopanib, if tolerable, may offer patients more convenience without sacrificing safety and efficacy.

#### 2.6.2. Phase 2 Justification

The Phase 2 portion of the trial is designed to assess the activity of TRC105 in combination with the approved dose of pazopanib, as compared to the single agent activity established for pazopanib in a prior study. Activity of the combination will be assessed as PFS (primary endpoint) and also ORR. Efficacy endpoints will be retrospectively correlated with expression of endoglin on tumor tissue to determine if direct endoglin expression on sarcoma (in addition to the tumor vasculature) may be used as a marker to enrich for responsive sarcoma subtypes in future studies.

Given that the two drugs were well tolerated together at their single agent doses, the phase 2 portion of the study will dose both drugs starting in cycle 1. Dose reductions of pazopanib, based on individual patient tolerability, are permitted starting in cycle 1.

Five patients with cutaneous angiosarcoma were enrolled in the phase 1b/Phase 2 portion of this study and all five patients had tumor reductions, including two patients who progressed on pazopanib prior to trial enrollment. Notabaly, two patients have ongoing complete responses (at 15 and 22 months of treatment) including one patient who progressed previously after pazopanib and docetaxel. These data were presented at ASCO 2016. Given these signs of activity, two additional phase 2 cohorts of up to 13 patients, each with histologically confirmed angiosarcoma that have progressed following prior systemic treatment, will be enrolled to assess the overall response rate in this subtype of soft tissue sarcoma.

### IND 131053 5.3.5.2 Clinical Protocol

Patients in angiosarcoma cohort 1 will initially receive weekly single-agent TRC105 with transition to treatment with the combination of TRC105 and pazopanib at progression per RECIST 1.1.

Patients in angiosarcoma cohort 2 will receive TRC105 in combination with pazopanib starting on cycle 1 day 1.

# 2.7. Conduct

The 105SAR101 clinical trial will be conducted in compliance with the protocol, GCP, and the applicable regulatory requirements.

### 3. TRIAL OBJECTIVES AND PURPOSE

# 3.1. Phase 1b Objectives

#### **3.1.1. Purpose**

The purpose of this study is to evaluate the safety and effectiveness of TRC105 in combination with pazopanib.

## 3.1.2. Primary objectives

• To evaluate safety and tolerability and determine a recommended phase 2 dose for TRC105 when added to standard dose pazopanib in patients with advanced soft tissue sarcoma.

# 3.1.3. Secondary objectives

- To assess preliminary evidence of improved antitumor activity when TRC105 is added to pazopanib, by assessing response rate and progression-free survival
- To characterize the pharmacokinetic profile of TRC105 when given with pazopanib
- To evaluate the formation of TRC105 anti-product antibodies
- To correlate efficacy with expression of endoglin on sarcoma tissue
- To explore pharmacodynamic effects on circulating angiogenic biomarkers

# 3.2. Phase 2 Objectives

#### **3.2.1. Purpose**

The purpose of this study is to evaluate the safety and effectiveness of TRC105 in combination with pazopanib.

#### 3.2.2. Primary objectives

- To estimate the PFS of patients with advanced soft tissue sarcoma by RECIST 1.1
- To estimate the ORR in a cohort of patients with angiosarcoma by RECIST 1.1

### 3.2.3. Secondary objectives

- To estimate the ORR in patients with advanced soft tissue sarcoma by RECIST 1.1, including duration of response
- To estimate the PFS in a cohort of patients with angiosarcoma by RECIST 1.1
- To determine the frequency and severity of adverse events as assessed by NCI CTCAE (Version 4.0)
- To characterize the pharmacokinetic profile of TRC105 and pazopanib
- To evaluate the formation of TRC105 anti-product antibodies
- To explore the correlation of efficacy variables (e.g., PFS and ORR) with endoglin expression on sarcoma
- To explore the effects of TRC105 on circulating angiogenic protein biomarkers

#### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

#### 4.1.1. Overview

All patients must sign a consent form prior to undertaking any study-related procedures. Prospective patients will be screened to determine if they qualify for the study within 28 days of enrollment. Toxicities will be graded according to the NCI CTCAE Version 4.0.

#### **4.1.1.1. Phase 1b Overview**

This is a multicenter, open-label, nonrandomized, phase 1b, dose-finding study of TRC105 in combination with standard dose pazopanib in patients with advanced soft tissue sarcoma. Escalating doses of i.v. TRC105 will be administered weekly or every two weeks beginning with Dose Level 1 in combination with oral pazopanib given as 800 mg p.o. once daily (see TRC105 Administration section 6.1.6 and Pazopanib Dosing section 6.2.5). Intermediate TRC105 doses (below the MTD established during the trial) may be explored based upon clinical, PK, and/or biomarker data.

| Dose Level | Number of<br>Evaluable<br>Subjects | Pazopanib mg p.o.,<br>once daily (with<br>dose reduction<br>allowed based on<br>tolerability) | TRC105<br>mg/kg<br>IV |
|---|---|---|---|
| -1 | 3-6 | 800 | 6 (weekly beginning cycle 2 day 1) <sup>a</sup> |
| 1 (Starting Dose) | 3-6 | 8 (weekly beginning cycle 2 day 1) <sup>a</sup> | |
| 2 | 3-6 | 800 | 10 (weekly beginning cycle 2 day 1) <sup>a</sup> |
| Expanded Cohort 1 | 9-12 (up to 15 total at the MTD) | 800 | MTD (weekly beginning cycle 2 day 1) <sup>a</sup> |
| 3 | 3-6 | 800 | <ul> <li>10 mg/kg weekly during cycle 1</li> <li>15 mg/kg every two weeks beginning cycle 2 day 1<sup>b</sup></li> </ul> |
| Expanded Cohort 2 | At least 6 patients will be treated at the MTD | 800 | <ul> <li>10 mg/kg weekly during cycle 1</li> <li>15 mg/kg every two weeks beginning cycle 2 day 1<sup>b</sup></li> </ul> |

<sup>&</sup>lt;sup>a</sup> In dose levels -1 to Expanded Cohort 1, pazopanib will be dosed alone during cycle 1 and dosing with TRC105 will begin on cycle 2 day 1. The first weekly TRC105 dose (cycle 2 day 1) will be split into two doses whereby 3

mg/kg is administered on cycle 2 day 1 and the balance (e.g., 5 mg/kg for Dose Level 1) is administered on cycle 2 day 4, the full dose is then given weekly thereafter starting with cycle 2 day 8.

<sup>b</sup> In dose levels 3 and expanded cohort 2, pazopanib and TRC105 dosing will begin on cycle 1 day 1. Pazopanib dosing will begin on cycle 1 day 1 and once daily thereafter, and TRC105 will be administered weekly during cycle 1. The first weekly TRC105 dose will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4. Starting on cycle 2 day 1 and beyond, TRC105 will be administered every two weeks on days 1 and 15 once it is determined that the every two week dosing MTD has not been exceeded..

In dose levels -1, 1, 2 and expanded cohort 1, patients will receive 800 mg of pazopanib daily p.o. in cycle 1, which will be two to four weeks in duration prior to the initial dose of TRC105 given on cycle 2 day 1. Cycle 1 will therefore be as short as 14 days or as long as 28 days, based on the time needed to determine a tolerable dose of pazopanib in each patient. Dose reductions of pazopanib are allowed during cycle 1 based on individual patient tolerability (as well as following cycle 1). TRC105 dosing will begin at 8 mg/kg (Dose Level 1) on cycle 2 day 1. Prior to administration of TRC105 on cycle 2 day 1, all study patients must maintain eligibility criteria indicating adequate organ function, medical status and ECOG performance status (i.e., patients must maintain inclusion criterion #6, 8, 9 and 10 and exclusion criteria #8-21 to continue into cycle 2) and must be able to tolerate pazopanib. A -1 Dose Level has also been included (6 mg/kg) and will be enrolled if 8 mg/kg TRC105 dosed with pazopanib exceeds weekly the MTD. For dose levels -1, 1 and 2, the DLT evaluation period, for purposes of dose expansion, will be the initial 28 days of dosing with TRC105 and pazopanib (from cycle 2 day 1 through cycle 2 day 28). Each cycle will be 28 days in duration.

For dose levels 3, and Expanded Cohort 2, both pazopanib and TRC105 dosing will begin on C1D1 and the DLT evaluation will be the first 28 days of dosing pazopanib with TRC105 every 2 weeks (i.e., from cycle 2 day 1 through cycle 2 day 28). At least 6 patients will be treated at the every two week dosing MTD (or top dose level if a MTD is not determined).

Three patients will be initially enrolled and treated at each dose level. If none of these 3 patients experiences a dose-limiting toxicity (DLT) during the 28-day evaluation period (extending from cycle 2 day 1 until cycle 2 day 28), dose escalation will proceed following review of safety data with site staff including the principal investigators at all sites.

If 1 of 3 patients experiences DLT, the dose level will be expanded to 6 patients. The maximum tolerated dose (MTD) will have been exceeded if  $\geq$  33% of patients experience DLT at a given dose level. DLT will have occurred when a patient has 1 or more toxicity listed in the table below that is at least possibly related to the combination of pazopanib and TRC105 during the 28 day DLT evaluation period (cycle 2). Patients who exit the study for reasons other than DLT prior to completion of the 28-day DLT evaluation period (cycle 2) will be replaced to ensure an adequate safety assessment in each cohort. Patients who experience DLT who receive less than the prescribed dose of TRC105 or pazopanib due to documented toxicity during the DLT evaluation period will be considered evaluable for dose escalation purposes. A given TRC105 dose level may be reenrolled at  $\geq$ 50% of the pazopanib dose intensity upon agreement of study investigators.

**Table 3:** Dose Limiting Toxicity Definition and Criteria

| <b>Toxicity Category</b> | Drug-Related Toxicity/Grade |
|---|---|
| Hematologic | Grade 4 neutropenia for ≥ 5 days |
| | Febrile neutropenia: grade 4 neutropenia with fever > 38.5 °C both sustained over a 24 hour period. |
| | Neutropenic infection: grade $\geq 3$ neutropenia with grade $\geq 3$ infection |
| | Anemia ≥ grade 4 |
| | Grade $>$ 4 thrombocytopenia or grade $\ge$ 3 thrombocytopenia and grade $\ge$ 3 hemorrhage |
| Nonhematologic | <ul> <li>Grade 3 or 4 nonhematologic toxicity with the following exceptions:</li> <li>Nausea, vomiting or diarrhea for &lt; 48 hours<sup>a</sup></li> <li>Asymptomatic electrolyte abnormalities that are corrected to grade 1 or better in &lt; 72 hours<sup>b</sup></li> </ul> |
| | <ul> <li>headache lasting less than 48 hours</li> </ul> |

<sup>&</sup>lt;sup>a</sup>Patients with related grade 3 or 4 diarrhea, nausea or vomiting for  $\geq$  48 hours despite optimal medical therapy will require a one-level dose-reduction of TRC105.

#### 4.1.1.2. Phase 2 Overview

This is a multicenter, non-randomized, phase 2 study of TRC105 in combination with standard dose pazopanib. Sixty three patients will be treated in the phase 2 portion of the study at 10 mg/kg weekly; the MTD (top dose level studied as a MTD was not determined) of the phase 1b portion of the study (dose levels -1, 1, 2 and expanded cohort 1). Patients will receive pazopanib once daily and will receive TRC105 at 3 mg/kg on cycle 1 day 1, 7 mg/kg on cycle 1 day 4, and 10 mg/kg on cycle 1 day 8 and weekly thereafter. Each cycle is 28 days in duration.

Two additional phase 2 cohorts of up to thirteen patients each with angiosarcoma that have had disease progression following treatment with prior systemic therapy will be assessed.

Angiosarcoma cohort 1 patients will initially receive weekly single-agent TRC105 at a dose of 10 mg/kg weekly with transition to treatment with the combination of TRC105 and pazopanib at progression per RECIST 1.1.

Angiosarcoma cohort 2 patients will be assessed at a TRC105 dose of 10 mg/kg weekly in combination with 800 mg pazopanib once daily for the first cycle starting on cycle 1 day 1 followed by TRC105 15 mg/kg administered every two weeks starting from cycle 2 day 1 onward in combination with pazopanib 800 mg once daily.

Active patients that are past cycle 1, may be switched to an every 2 week dosing schedule at a TRC105 dose of 15 mg/kg every two weeks once **SPONSOR SENDS NOTIFICATION TO PROCEED WITH EVERY TWO WEEK DOSING**.

• TRC105 will be administered at 10 mg/kg weekly during cycle 1.

<sup>&</sup>lt;sup>b</sup>Patients with related grade 3 or 4 electrolyte abnormalities that persist for ≥ 72 hours will require a one level dose-reduction of TRC105.

- The first weekly TRC105 dose (10 mg/kg) will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4.
- Starting on cycle 2 day 1 and beyond, TRC105 may be administered every two weeks on days 1 and 15 at the every two week dosing MTD.

Pazopanib dosing will start at 800 mg once daily. Dose reductions of pazopanib are allowed based on individual patient tolerability. Each cycle in this cohort is 28 days in duration.

#### 4.1.2. Trial Procedures

All on-study procedures are permitted within the time window indicated in the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7).

### **4.1.2.1.** Screening

The following screening procedures must be performed within 28 days prior to the first day of study therapy. Qualifying hematology (including Fe studies), serum chemistry (including TSH testing), coagulation, physical examination, ECG, pregnancy and urinalysis collected within 7 days of cycle 1 day 1 do not need to be repeated. The following will be performed according to the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7).

- Patient signature on current Institutional Review Board (IRB) approved informed consent form. Prior to undergoing any study-specific procedure, patients must read and sign the current Institutional Review Board (IRB) approved informed consent form. Patients may sign consent prior to the 28 day screening period.
- Medical history, baseline signs and symptoms, prior cancer therapy, prior cancer surgery, prior radiation therapy, drug allergies, primary diagnosis and demographics.
- Physical examination including examination of all major body systems, ECOG performance status, and vital signs.
- Hematology (including serum iron, ferritin and total iron binding capacity), coagulation (INR) and serum chemistry (including thyroid stimulating hormone (TSH)) to be performed locally.
- Serum or urine pregnancy test for all females of childbearing potential to be performed locally.
- Urinalysis to be performed locally. Microscopic analysis and/or urine protein-creatinine ratio (UPCR) should be performed as clinically indicated.
- CT or MRI scans of chest, abdomen and pelvis in addition to any other applicable sites of disease. Brain and bone scans to be performed if metastasis is suspected prior to starting the study. Color photography with caliper or ruler measurements should be used to assess cutaneous tumors (target lesions).
- Single tracing 12-Lead ECG (QT, PR and QRS intervals and heart rate will be captured).
- Assessment of concomitant medications and treatments from 28 days prior to the start of study treatment.

• Archival Tumor Tissue Specimens: Archival specimens (formalin-fixed, paraffin-embedded) of the primary cancer specimen and/or metastatic cancer specimen for each study participant. It is preferable that the entire paraffin block be submitted, but if this is not feasible, then at least 20 unstained slides are requested for immunohistochemical analysis (sections of ~ 5 microns are preferred). See separate laboratory guide for further collection and shipment information.

#### 4.1.2.2. Trial Period

Qualifying hematology (including Fe studies), blood chemistry (including TSH testing), coagulation, urinalysis, physical examination, ECG, and pregnancy test do not need to be repeated on cycle 1 day 1 if acceptable screening assessments are performed within 7 days prior to the start of study therapy. For dose levels -1, 1, 2 and expanded cohort 1 of the phase 1b portion of the study, prior to administration of TRC105 on cycle 2 day 1, all study patients must maintain eligibility criteria indicating adequate organ function, medical status and ECOG performance status (i.e., all patients must maintain inclusion criterion #4, 5 and 6 and exclusion criteria #8-21 to continue into cycle 2). On days of dosing, all assessments should be performed prior to dosing with TRC105 unless otherwise indicated in the Schedule of Assessments. Patients will receive 2 cycles (approximately 6-8 weeks) of treatment. Patients who demonstrate a response of CR, PR or SD, will be eligible for additional treatment until progression. For patients in the angiosarcoma cohort 1, disease progression for withdrawal from study therapy refers to disease progression while receiving TRC105 plus pazopanib combination therapy. Patients who cannot tolerate pazopanib or TRC105 therapy and who demonstrate a response of complete response (CR), partial response (PR) or stable disease (SD) with the combination and are thought to benefit from continued single agent therapy may continue on study on TRC105 or pazopanib alone. Each cycle is 28 days in duration, with the exception of cycle 1 for phase 1b dose levels -1, 1, 2 and expanded cohort 1 which will be 2 to 4 weeks in duration. The following will be performed according to the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7).

- Physical examination including examination of all major body systems, ECOG performance status, weight and vital signs (heart rate, temperature, blood pressure, respiratory rate).
  - O Assessment of vital signs during TRC105 infusion: Vital signs are to be assessed pre-infusion (i.e., within 30 minutes of starting the infusion), every 30 minutes during the infusion (+/- 15 minutes), and at the end of the infusion (i.e., within 30 minutes after completing the infusion). Vital signs should be monitored more frequently and/or beyond the completion of the infusion if medically indicated (e.g. if the patient experiences an infusion reaction that has not yet resolved).
- Hematology, coagulation (INR) and serum chemistry (including TSH) to be performed locally.
- Serum or urine pregnancy test for all females of childbearing potential to be performed locally.
- Single tracing 12-Lead ECG (QT, PR and QRS intervals and heart rate will be captured).

- Urinalysis to be performed locally. Microscopic analysis and/or urine protein-creatinine ratio (UPCR) should be performed as clinically indicated.
- Phase 1b dose levels -1, 1, 2 and expanded cohort 1 and angiosarcoma cohort 2: Blood sampling for TRC105 pharmacokinetics will include a pre-infusion trough sample and an end-of-infusion peak sample to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection times, procedures, processing, storage and shipment).
- Phase 1b dose levels 3, 4 and expanded cohort 2: Blood sampling for **TRC105** and **pazopanib** pharmacokinetics will include trough sample collections to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection times, procedures, processing, storage and shipment).
- Phase 2 including angiosarcoma cohorts: Blood sampling for TRC105 and pazopanib pharmacokinetics will include trough sample collections to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection times, procedures, processing, storage and shipment).
- Blood sampling for immunogenicity to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection, processing, storage and shipment).
- Blood sampling for protein biomarker analysis by a third party laboratory (see laboratory manual for specific instructions regarding collection processing, storage and shipment)
- CT or MRI scans of chest, abdomen and/or pelvis in addition to any other applicable sites of disease. Scan of the chest, abdomen, and pelvis to be performed on-study as outlined in the assessment table. Known areas of disease should be consistently followed throughout the study. Assessments should be performed whenever disease progression is suspected. Allowable window for tumor imaging studies is +/- 7 days. Brain and bone scans to be performed if metastasis is suspected prior to starting the study and during study conduct. Color photography with caliper or ruler measurements should be used to assess cutaneous tumors (target lesions).
  - Patients in angiosarcoma cohort 1 who progress on single agent TRC105 by RECIST, tumor assessments will occur every 6 weeks from the new baseline (ie scans that showed progression on single agent).
- Administration of TRC105. TRC105 diluted in normal saline will be administered as a 1 to 4 hour infusion (+/- 15 minutes) following premedication (see Section 6.1.6) according to the pertinent schedule of assessments.
  - **Phase 1b Dose Levels -1, 1, 2 and Expanded Cohort 1**: TRC105 will not be given in cycle 1. The first TRC105 dose will be split into two doses whereby 3 mg/kg is administered on cycle 2 day 1, and the balance is administered on cycle 2 day 4. The entire weekly dose of TRC105 (6, 8 or 10 mg/kg) is then given on cycle 2 day 8 and weekly thereafter (e.g., if TRC105 is given at 3 mg/kg on cycle 2 day 1 and at 5 mg/kg on cycle 2 day 4, then 8 mg/kg is given on cycle 2 day 8).

- Upon completion of enrollment of phase 1b dose level 3 and notification by the sponsor, active patients that are past cycle 2, may be switched to an every 2 week dosing schedule at the every 2 week dosing MTD.
- **Phase 1b Dose Levels 3and Expanded Cohort 2**: TRC105 dosing will start on cycle 1 day 1 and the first dose will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1, and the balance is administered on cycle 1 day 4. The entire weekly dose of TRC105 (10 mg/kg) is then given on cycle 1 day 8, cycle 1 day 15 and on cycle 1 day 22. Beginning with cycle 2 day 1, TRC105 will be dosed at 15mg/kg and every two weeks thereafter (days 1 and 15).
- Phase 2 Soft Tissue Sarcoma and Phase 2 Angiosarcoma Cohorts: TRC105 dosing will start on cycle 1 day 1 and the first dose will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1, and the balance is administered on cycle 1 day 4. The entire weekly dose of TRC105 (10 mg/kg) is then given on cycle 1 day 8 and weekly thereafter.
  - Upon completion of enrollment of phase 1b dose level 3 and notification by the sponsor, active patients that are past cycle 1, may be switched to an every 2 week dosing schedule at the every 2 week dosing MTD.

TRC105 will be administered intravenously utilizing an infusion pump. TRC105 has been demonstrated to be compatible with polyethylene lined, non-DEHP infusion sets and polyvinyl chloride, non-DEHP infusion sets. TRC105 is required to be administered with a 0.2 micron downstream filter. Duration of infusion administration may be increased as medically necessary.

- Pazopanib dosing. The oral dose of pazopanib is 200 to 800 mg once daily without food (at least 1 hour before or 2 hours after a meal) beginning on cycle 1 day 1 in the absence of toxicity, except in the phase 2 angiosarcoma cohort 1 where pazopanib will be dosed starting at the time of disease progression on TRC105 single-agent and once daily thereafter in the absence of toxicity. The dose of pazopanib will not exceed 800 mg and may be reduced based on individual patient tolerability. Do not crush tablets due to the potential for increased rate of absorption which may affect systemic exposure. If a dose is missed, it should not be taken if it is less than 12 hours until the next dose.
- Assessment of adverse events.
- Assessment of concomitant medications and concomitant treatments.

#### 4.1.3. End of Study Assessments

Assessments other than TRC105 pharmacokinetics, immunogenicity and protein biomarkers only need to be completed if they were not completed during the previous 2 weeks on study (during the last 8 weeks on study for radiologic tumor assessments). The following will be performed according to the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7).

- Physical examination including examination of all major body systems, ECOG performance status, and vital signs.
- Single tracing 12-Lead ECG (QT, PR and QRS intervals and heart rate will be captured).
- Hematology, and serum chemistry (including TSH) to be performed locally.
- Urinalysis to be performed locally. Microscopic analysis and/or urine protein-creatinine ratio (UPCR) should be performed as clinically indicated.
- Phase 1b dose levels -1, 1, 2 and expanded cohort 1: Blood sampling for TRC105 pharmacokinetics to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection times, procedures, processing, storage and shipment).
- Phase 1b dose levels 3, 4 and expanded cohort 2: Blood sampling for **TRC105** and **pazopanib** pharmacokinetics will include trough sample collections to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection times, procedures, processing, storage and shipment).
- Phase 2 including angiosarcoma cohorts: Blood sampling for TRC105 and pazopanib pharmacokinetics be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection times, procedures, processing, storage and shipment).
- Blood sampling for immunogenicity to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection, processing, storage and shipment).
- Blood sampling for protein biomarker analysis by a third party laboratory (see laboratory manual for specific instructions regarding collection processing, storage and shipment)
- CT or MRI scans of chest, abdomen and pelvis in addition to any other applicable sites of disease. Color photography with caliper or ruler measurements should be used to assess cutaneous tumors (target lesions).
- Assessment of adverse events.
- Assessment of concomitant medications and concomitant treatments.

#### 4.1.4. Post Treatment Follow-up

The following will be performed according to the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7). Samples should be collected and assessments performed even if new anti-cancer therapy commences during the follow-up period.

• Assessment of adverse events. The Investigator should continue to report any related or possibly related adverse events that occur beyond the adverse event reporting period.

- Phase 1b dose levels -1, 1, 2 and expanded cohort 1: Blood sampling for TRC105 pharmacokinetics to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection, processing, storage and shipment).
- Phase 1b dose levels 3, 4 and expanded cohort 2: Blood sampling for **TRC105** and **pazopanib** pharmacokinetics will include trough sample collections to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection times, procedures, processing, storage and shipment).
- Phase 2 including angiosarcoma cohorts: Blood sampling for TRC105 and pazopanib pharmacokinetics to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection times, procedures, processing, storage and shipment).
- Blood sampling for immunogenicity to be analyzed by a third party laboratory (see laboratory manual for specific instructions regarding collection, processing, storage and shipment).
- Serum or urine pregnancy test for all females of childbearing potential to be performed locally.
- Assessment of concomitant medications and concomitant treatments.

Table 4: Schedule of Assessments Phase 1b Dose Levels -1, 1, 2 & Expanded Cohort 1

| | Screening | Cycle | e 1 [23] | | Су | cle 2 [23] | | | | Cycle 3+ | [21] [23] | | End | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activities Baseline Documentation | Day -28 | Day 1 | Day 8<br>(Day 15)<br>(Day 22)<br>[1] | Day 1<br>[1] | Day 4 | Day<br>8<br>[1] | Day 15<br>[1] | Day<br>22<br>[1] | Day 1 | Day 8 | Day<br>15<br>[1] | Day<br>22<br>[1] | of<br>Stud<br>y<br>[3] | 28 Day<br>Follow-up<br>[22] |
| Informed Consent [4] | Х | | | | | | | | | | | | | |
| Medical/Oncology History [5] | Х | | | | | | | | | | | | | |
| Baseline Signs and Symptoms [5] | Х | | | | | | | | | | | | | |
| Physical Examination [6] | Х | Х | | Х | | | | | Х | | | | Х | |
| Vital Signs [7] | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Laboratory Studies | | | | | | | | | | | | | | |
| Hematology [8] | X+Fe | X+Fe | | X+Fe<br>Day -7 | | | Х | | Х | | Х | | Х | |
| Coagulation [8] | X | Х | | X Day -7 | | | | | | | | | | |
| Blood Chemistry [8] | X+TSH | X+TSH | | X+TSH<br>Day -7 | | | Х | | X +<br>TSH | | | | X+<br>TSH | |
| Pregnancy Test [9] | Day -7 | | | | | | | | | | | | | Х |
| Urinalysis [10] | Х | Х | | X Day -7 | | | | | Х | | | | X | |
| Treatment w/ Study Drug | | | | | | | | | | | | | | |
| TRC105 Dosing [11] | | | | X Split | X Split | Х | Х | Х | Х | Х | Х | Х | | |
| Pazopanib [12] | | Daily | | | | | | | | | | | | |
| Tumor Assessments | | | | | | | | | | | | | | |
| CT or MRI Scans [13] Other Clinical Assessments | X | | | | | | | Х | | | | Even<br>Cycles | Х | |
| 12-Lead ECG [14] | X | | X Day 8 | | | | | | | | | | X | |
| Concomitant | ^ | | A Day o | | | | Х | | | | | | ^ | |
| Medications/Treatments [15] | Х | X | X | Х | Х | Х | Х | X | Х | Х | х | Х | Х | Х |
| Adverse Events [16] | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Special Laboratory Assessments | | | | | | | | | | | | | | |
| TRC105 PK Pre-Dose [17] | | | | | | | Х | | Even<br>Cycles | | | | | |
| TRC105 PK Post-Dose [17] | | | | | | | Х | | Even<br>Cycles | | | | Х | X |
| Anti-product antibodies [18] | | Х | | | | _ | | | | | | | Х | Х |
| Protein Biomarkers [19] | | Х | | Х | | | Х | | Even<br>Cycles | | | | Х | |
| Archival Tumor Tissue [20] | X | | | | | | | | | | | | | |

#### Schedule of Assessments Footnotes Phase 1b Dose Levels -1, 1, 2 & Expanded Cohort 1

- 1. **Days of Treatment with TRC105:** All assessments should be performed prior to the TRC105 infusion unless otherwise indicated. Each cycle is 28 days in duration, with the exception of cycle 1 which is 2-4 weeks in duration.
- 2. **Cycle 1 day 1:** Hematology (including iron studies), blood chemistry (including TSH testing), urinalysis, physical examination, ECG and pregnancy test not required if acceptable screening assessment is performed within 7 days prior to the start of treatment on cycle 1 day 1.
- 3. **End of Study:** The end of study visit should generally occur within 7 days (+/- 1 day) of the last dose of TRC105. Assessments other than TRC105 pharmacokinetics, immunogenicity and protein biomarkers do not need to be repeated if performed within the previous 2 weeks (previous 8 weeks for radiologic tumor assessments). Follow-up visits should occur 28 days following the last dose of TRC105 study drug as outlined in the Schedule of Assessments.
- 4. **Informed Consent:** Must be obtained prior to undergoing any study specific procedure and may occur prior to the 28-day screening period.
- 5. **Medical and Oncologic History, Demographics and Baseline Signs and Symptoms:** All information related to prior anticancer treatment should be recorded. Significant medical history and baseline signs and symptoms should be captured from the date of informed consent.
- 6. Physical Examination: Examination of major body systems and ECOG performance status.
- 7. **Vital Signs:** Heart rate, temperature, blood pressure, respiratory rate, weight. Assessment of vital signs during TRC105 Infusions: Vital signs are to be assessed pre-infusion (i.e., within 30 minutes of starting the infusion) every 30 minutes during the infusion (+/- 15 minutes) and at the end of the infusion (i.e. within 30 minutes after completing the infusion). Vital signs should be monitored more frequently and/or beyond the completion of the infusion if medically indicated (e.g. if the patient experiences an infusion reaction that has not yet resolved).
- 8. **Hematology, Chemistry & Coagulation:** Testing to be performed locally. Thyroid stimulating hormone to be tested at screening, day 1 of each cycle and at the end of study visit. Cycle 1 day 1 assessments only need to be performed if screening assessments were performed more than 7 days prior to cycle 1 day 1. Cycle 2 day 1 labs should be performed within 7 days of cycle 2 day 1, results should be reviewed prior to dosing with TRC105 on cycle 2 day 1. Iron studies (FE) to be performed according to the schedule of assessments and as clinically indicated during the study. Thyroid stimulating hormone (TSH) to be performed according to the schedule of assessments and as clinically indicated during the study. Lab assessments may be performed within 3 days prior to TRC105 dosing. In addition to the assessments scheduled for the clinical trial, patients should undergo assessment as appropriate to ensure safe treatment. See Section 8.1.1.1 for specific panel collection requirements.
- 9. **Pregnancy Test:** Testing to be performed locally. All female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days of cycle 1 day 1 and 28 days following the last dose of TRC105.
- 10. **Urinalysis:** To be performed locally. Cycle 1 day 1 urinalysis only needs to be performed if screening urinalysis was performed more than 7 days prior to cycle 1 day 1. Cycle 2 day 1 urinalysis should be performed within 7 days of cycle 2 day 1, results should be reviewed prior to dosing with TRC105 on cycle 2 day 1. Microscopic analysis and/or urine protein creatinine ratio or 24-hour urine protein collection should be performed as clinically indicated.
- 11. **TRC105** Administration: Intravenous TRC105 diluted in normal saline will be administered every 7 days. The first weekly TRC105 dose will be given on cycle 2 day 1 and split into two doses whereby 3 mg/kg is administered on cycle 2 day 1 and the balance is administered on cycle 2 day 4. The entire weekly dose of TRC105 (6, 8 or 10 mg/kg) is then given on cycle 2 day 8 and weekly thereafter. See Section 6.1.6 for specific TRC105 administration guidelines.
  - Upon completion of enrollment of phase 1b dose levels 3 and notification by the sponsor, active patients that are past cycle 2, may be switched to an every 2 week dosing schedule at the every 2 week dosing MTD.
- 12. **Pazopanib Dosing:** Oral pazopanib will be dosed once daily at 800 mg starting on cycle 1 day 1 in the absence of toxicity on days 1-28 of each 28 day cycle according to the pazopanib package insert. During cycle 1 pazopanib will be given for a total of 2 to 4 weeks, in the absence of TRC105 to determine a tolerable dose in each patient. Dose reductions are allowed based on individual patient tolerability, including during the initial 2 to 4 week period when pazopanib is dosed in the absence of TRC105. See Section 6.2 for specific dosing guidelines.
- 13. **CT or MRI Tumor Imaging:** Images of the chest, abdomen, and pelvis to be performed at screening, and on-study as outlined in the assessment table. Known areas of disease should be consistently followed throughout the study. Assessments should be performed whenever disease progression is suspected. Allowable

- window for tumor imaging studies is +/- 7 days. Brain and bone scans are to be performed if metastases are suspected at screening or during study therapy. Beyond cycle 6 scans will be performed every 3 cycles (cycle 9 day 22, cycle 12 day 22 etc.). Color photography with caliper measurements should be used to assess cutaneous tumors (target lesions).
- 14. **12-Lead ECG:** Single tracing 12-lead ECG will be performed at screening and at the time-points indicated in the Schedule of Assessments (pre-dose). If the patient develops an arrhythmia, the ECG should be repeated on day 1 of each subsequent cycle. For a QTc >500 ms, a repeat ECG for confirmation and evaluation of the ECG by a cardiologist is recommended. Additional ECGs may be performed on study as clinically indicated.
- 15. **Concomitant Medications and Treatments:** Concomitant medications and treatments will be recorded from 28 days prior to the start of study treatment and up to 28 days following the last dose of study treatment. Required TRC105 premedications should be recorded on TRC105 premedications CRF.
- 16. **Adverse Events:** Patients must be followed for adverse events from the first day of treatment with pazopanib or TRC105 study drug until at least 28 days after the last dose of TRC105 or pazopanib study drug treatment, or until all serious or TRC105 related toxicities have resolved or are determined to be "chronic" or "stable", whichever is later. "Baseline-signs and symptoms" will be recorded from the date of informed consent on corresponding case report forms. Any serious AE that is possibly related to TRC105 occurring from the time of first TRC105 dose or at any point after the reporting period must be promptly reported to TRACON.
- 17. **TRC105 Pharmacokinetics Trough Concentration:** A 5 mL blood sample to be collected at the time-points indicated in the Schedule of Assessments, prior to starting the TRC105 infusion. Samples will be stored at approximately -70°C. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional PK samples may also be collected at the time of unexpected clinical events.
  - **TRC105 Pharmacokinetics Peak Concentrations:** A 5 mL blood sample to be collected within 10 minutes of the completion of the TRC105 infusion at the time-points indicated in the Schedule of Assessments. Samples will be stored at approximately -70°C. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional PK samples may also be collected at the time of unexpected clinical events.
- 18. **Anti-product antibodies:** 5 mL blood sample will be collected to assess anti-product antibodies at the time-points indicated in the schedule of assessments and stored at approximately -70°C to be analysed by a central laboratory. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional anti-product antibody samples may also be collected at the time of unexpected clinical events.
- 19. **Protein Biomarkers:** One 10 mL purple top (K<sub>3</sub>EDTA) tube will be collected at the time-points indicated in the schedule of assessments and stored at approximately -70°C to be analysed by a central laboratory. See separate laboratory guide for further collection and shipment information.
- 20. **Archival Tumor Tissue:** Archival specimens (formalin-fixed, paraffin-embedded) are required of the primary cancer and/or metastatic cancer specimen for each study participant. It is preferable that the entire paraffin block be submitted, but if this is not feasible, then at least 20 unstained slides are requested for immunohistochemical analysis (sections of 5 microns are preferred). See separate laboratory guide for further collection and shipment information.
- 21. Cycle 3+ Treatment: Patients who demonstrate a response of CR, PR or SD will be eligible for additional treatment until progression.
- 22. **Follow-up:** The follow-up visit should occur 28 days following the last dose of TRC105. The allowable visit window is +/- 7 days.
- 23. Allowable window for each visit within the cycle is +/- 2 days unless otherwise stated.

Table 5: Schedule of Assessments Phase 1b Dose Levels 3 and Expanded Cohort 2

| | Screening | | (10 mg | Cycle 1<br>g/kg Week | i <b>ly)</b> [23] | | (15 mg/ | cle 2<br>kg every<br>eks) [23] | (15 mg/kg | e 3+<br><b>every two</b><br>[21] [23] | Fad | 28 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activities Baseline Documentation | Day -28 | Day 1<br>[1] [2] | Day 4<br>[1] | Day 8<br>[1] | Day 15<br>[1] | Day 22<br>[1] | Day 1<br>[1] | Day 15<br>[1] | Day 1<br>[1] | Day 15<br>[1] | End<br>of<br>Study<br>[3] | Day<br>Follow<br>-up<br>[22] |
| Informed Consent [4] | Х | | | | | | | | | | | |
| Medical/Oncology History [5] | X | | | | | | | | | | | |
| Baseline Signs and Symptoms [5] | X | | | | | | | | | | | |
| Physical Examination [6] | X | Х | | | | | Х | | Х | | Х | |
| Vital Signs [7] | X | X | Х | Х | Х | Х | X | Х | X | Х | X | |
| Laboratory Studies | Α | | | | ^ | ^ | | | ^ | | | |
| Hematology [8] | X+Fe | Х | | | Х | | Х | Х | Х | Х | Х | |
| Coagulation [8] | Х | Х | | | | | Х | | | | Х | |
| Blood Chemistry [8] | X+TSH | X+TSH | | | | | X+TSH | | X + TSH | | X + TSH | |
| Pregnancy Test [9] | Day -7 | | | | | | Х | | Х | | | Х |
| Urinalysis [10] | X | Х | | | | | Х | | Х | | Х | |
| Treatment w/ Study Drug | | | | | | | | | | | | |
| TRC105 Dosing [11] | | X Split | X Split | Х | Х | Х | Х | Х | Х | Х | | |
| Pazopanib [12] | | | | Daily | | | Daily | | Daily | | | |
| Tumor Assessments | | | | | | | | | | | | |
| CT or MRI Scans [13] | Х | | | | | | | X<br>Day 22 | | Day 22<br>Even<br>Cycles | х | |
| Other Clinical Assessments | | | | | | | | | | | | |
| 12-Lead ECG [14] | X | | | | Х | | | | | | Х | |
| Concomitant Medications/Treatments [15] | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х |
| Adverse Events [16] | | Х | X | X | Х | Х | Х | Х | Х | Х | Х | Х |
| Special Laboratory Assessments | | | | Х | | | | | )/ O | | Х | |
| Trough PK [17] | | Х | | | | | Х | Х | X &<br>Even<br>Cycles | X (Cycle<br>3 only) | Х | Х |
| Anti-product antibodies [18] | | Х | | | | | Х | | Even<br>Cycles | | Х | Х |
| Protein Biomarkers [19] | | Х | | | | | Х | | Even<br>Cycles | | Х | |
| Archival Tumor Tissue [20] | Χ | | | | | | | | | | | |

#### Schedule of Assessments Footnotes for Phase 1b Dose Levels 3, 4 and Expanded Cohort 2

- 1. **Days of Treatment with TRC105:** All assessments should be performed prior to the TRC105 infusion unless otherwise indicated. Each cycle is 28 days in duration.
- 2. **Cycle 1 day 1:** Hematology (including iron studies), blood chemistry (including TSH testing), urinalysis, physical examination, ECG and pregnancy test not required if acceptable screening assessment is performed within 7 days prior to the start of treatment on cycle 1 day 1.
- 3. **End of Study:** The end of study visit should generally occur within 14 days (+/- 1 day) of the last dose of TRC105. Assessments other than pharmacokinetics, immunogenicity and protein biomarkers do not need to be repeated if performed within the previous 2 weeks (previous 8 weeks for radiologic tumor assessments). Follow-up visits should occur 28 days following the last dose of TRC105 study drug as outlined in the Schedule of Assessments.
- 4. **Informed Consent:** Must be obtained prior to undergoing any study specific procedure and may occur prior to the 28-day screening period.
- 5. **Medical and Oncologic History, Demographics and Baseline Signs and Symptoms:** All information related to prior anticancer treatment should be recorded. Significant medical history and baseline signs and symptoms should be captured from the date of informed consent.
- 6. **Physical Examination:** Examination of major body systems and ECOG performance status.
- 7. **Vital Signs:** Heart rate, temperature, blood pressure, respiratory rate, weight. Assessment of vital signs during TRC105 Infusions: Vital signs are to be assessed pre-infusion (i.e., within 30 minutes of starting the infusion) every 30 minutes during the infusion (+/- 15 minutes) and at the end of the infusion (i.e. within 30 minutes after completing the infusion). Vital signs should be monitored more frequently and/or beyond the completion of the infusion if medically indicated (e.g. if the patient experiences an infusion reaction that has not yet resolved).
- 8. **Hematology, Chemistry & Coagulation:** Testing to be performed locally. Thyroid stimulating hormone to be tested at screening, day 1 of each cycle and at the end of study visit. Cycle 1 day 1 assessments only need to be performed if screening assessments were performed more than 7 days prior to cycle 1 day 1. Iron studies (FE) to be performed according to the schedule of assessments and as clinically indicated during the study. Thyroid stimulating hormone (TSH) to be performed according to the schedule of assessments and as clinically indicated during the study. Lab assessments may be performed within 3 days prior to TRC105 dosing. In addition to the assessments scheduled for the clinical trial, patients should undergo assessment as appropriate to ensure safe treatment. See Section 8.1.1.1 for specific panel collection requirements.
- 9. **Pregnancy Test:** Testing to be performed locally. All female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days of cycle 1 day 1, day 1 of every cycle starting with cycle 2, and 28 days following the last dose of TRC105.
- 10. **Urinalysis:** To be performed locally. Cycle 1 day 1 urinalysis only needs to be performed if screening urinalysis was performed more than 7 days prior to cycle 1 day 1. Microscopic analysis and/or urine protein creatinine ratio or 24-hour urine protein collection should be performed as clinically indicated.
- 11. **TRC105 Administration:** Intravenous TRC105 diluted in normal saline will be administered every 7 days during Cycle 1. The first weekly TRC105 dose will be given on cycle 1 day 1 and split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4. The entire dose of TRC105 (10 mg/kg) is then given on cycle 1 day 8, cycle 1 day 15 and cycle 1 day 22. Starting on cycle 2 day 1 and beyond, TRC105 will be administered every two weeks on days 1 and 15. See Section 6.1.6 for specific TRC105 administration guidelines.
- 12. **Pazopanib Dosing:** Oral pazopanib will be dosed once daily at 800 mg starting on cycle 1 day 1 in the absence of toxicity on days 1-28 of each 28 day cycle according to the pazopanib package insert. Dose reductions are allowed based on individual patient tolerability. See Section 6.2 for specific dosing guidelines.
- 13. **CT or MRI Tumor Imaging:** Images of the chest, abdomen, and pelvis to be performed at screening, and on-study as outlined in the assessment table. Known areas of disease should be consistently followed throughout the study. Assessments should be performed whenever disease progression is suspected. Allowable window for tumor imaging studies is +/- 7 days. Brain and bone scans are to be performed if metastases are suspected at screening or during study therapy. Color photography with caliper or ruler measurements should be used to assess cutaneous tumors (target lesions).

- 14. **12-Lead ECG:** Single tracing 12-lead ECG will be performed at screening and at the time-points indicated in the Schedule of Assessments (pre-dose). If the patient develops an arrhythmia, the ECG should be repeated on day 1 of each subsequent cycle. For a QTc >500 ms, a repeat ECG for confirmation and evaluation of the ECG by a cardiologist is recommended. Additional ECGs may be performed on study as clinically indicated.
- 15. **Concomitant Medications and Treatments:** Concomitant medications and treatments will be recorded from 28 days prior to the start of study treatment and up to 28 days following the last dose of study treatment. Required TRC105 premedications should be recorded on TRC105 premedications CRF.
- 16. Adverse Events: Patients must be followed for adverse events from the first day of treatment with pazopanib or TRC105 study drug until at least 28 days after the last dose of TRC105 or pazopanib study drug treatment, or until all serious or TRC105 related toxicities have resolved or are determined to be "chronic" or "stable", whichever is later. "Baseline-signs and symptoms" will be recorded from the date of informed consent on corresponding case report forms. Any serious AE that is possibly related to TRC105 occurring from the time of first TRC105 dose or at any point after the reporting period must be promptly reported to TRACON.
- 17. **TRC105** and Pazopanib Pharmacokinetics Trough Concentration: A 5 mL blood sample each for TRC105 and pazopanib pharmacokinetics to be collected at the time-points indicated in the Schedule of Assessments, prior to starting the TRC105 infusion and prior to pazopanib dosing. Samples will be stored at approximately -70°C. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional PK samples may also be collected at the time of unexpected clinical events.
- 18. **Anti-product antibodies:** 5 mL blood sample will be collected to assess anti-product antibodies at the time-points indicated in the schedule of assessments and stored at approximately -70°C to be analysed by a central laboratory. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional anti-product antibody samples may also be collected at the time of unexpected clinical events.
- 19. **Protein Biomarkers:** One 10 mL purple top (K<sub>3</sub>EDTA) tube will be collected at the time-points indicated in the schedule of assessments and stored at approximately -70°C to be analysed by a central laboratory. See separate laboratory guide for further collection and shipment information.
- 20. **Archival Tumor Tissue:** Archival specimens (formalin-fixed, paraffin-embedded) are required of the primary cancer and/or metastatic cancer specimen for each study participant. It is preferable that the entire paraffin block be submitted, but if this is not feasible, then at least 20 unstained slides are requested for immunohistochemical analysis (sections of 5 microns are preferred). See separate laboratory guide for further collection and shipment information.
- 21. Cycle 3+ Treatment: Patients who demonstrate a response of CR, PR or SD will be eligible for additional treatment until progression.
- 22. **Follow-up:** The follow-up visit should occur 28 days following the last dose of TRC105. The allowable visit window is +/- 7 days.
- 23. Allowable window for each visit within the cycle is +/- 2 days unless otherwise stated.

**Table 6:** Schedule of Assessments Phase 2 Soft Tissue Sarcoma

| | Screening | | Су | cle 1 [23] | | | | Cycle 2+ | [21] [23] | | End | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol Activities Baseline Documentation | Day -28 | Day 1<br>[1] | Day 4<br>[1] | Day<br>8<br>[1] | Day 15<br>[1] | Day<br>22<br>[1] | Day 1<br>[1] | Day 8<br>[1] | Day<br>15<br>[1] | Day<br>22<br>[1] | of<br>Stud<br>y<br>[3] | 28 Day<br>Follow-up<br>[22] |
| Informed Consent [4] | Х | | | | | | | | | | | |
| Medical/Oncology History [5] | X | | | | | | | | | | | |
| Baseline Signs and Symptoms [5] | X | | | | | | | | | | | |
| Physical Examination [6] | X | Χ | | | | | X | | | | Х | |
| Vital Signs [7] | X | Χ | Х | Х | Х | Х | X | Х | Х | Х | Х | |
| Laboratory Studies | | | | | | | | | | | | |
| Hematology [8] | X+Fe | X+Fe | | | Χ | | Х | | Х | | Х | |
| Coagulation [8] | X | Х | | | | | | | | | | |
| Blood Chemistry [8] | X+TSH | X+TSH | | | Х | | X +<br>TSH | | | | X +<br>TSH | |
| Pregnancy Test [9] | X | Х | | | | | | | | | | Χ |
| Urinalysis [10] | X | Х | | | | | Х | | | | Х | |
| Treatment w/ Study Drug | | | | | | | | | | | | |
| TRC105 Dosing [11] | | X Split | X Split | Χ | Χ | X | Х | Х | X | Χ | | |
| Pazopanib [12] | | Daily | | | | | | | | | | |
| Tumor Assessments | | | | | | | | | | | | |
| CT or MRI Scans [13] | Х | | | | | | | | | Even<br>Cycles | Х | |
| Other Clinical Assessments | | | | | | | | | | | | |
| 12-Lead ECG [14] | X | Х | | | Χ | | | | | | X | |
| Concomitant Medications/Treatments [15] | X | X | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х |
| Adverse Events [16] | | Χ | Х | X | Χ | Х | Х | Х | Х | X | X | X |
| Special Laboratory Assessments | | | | | | | | | | | | |
| Anti-Product Antibody [17] | | Х | | | | | Even<br>Cycles | | | | Х | Х |
| Trough PK [18] | | Х | | | | | Even<br>Cycles | | | | Х | Х |
| Protein Biomarkers [19] | | X | | | | | Even<br>Cycles | | | | Х | |
| Archival Tumor Tissue [20] | X | | | | | | | | | | | |

#### Schedule of Assessments Footnotes Phase 2 Soft Tissue Sarcoma

- 1. **Days of Treatment with TRC105:** All assessments should be performed prior to the TRC105 infusion unless otherwise indicated. Each cycle is 28 days in duration.
- 2. **Cycle 1 day 1:** Hematology (including iron studies), blood chemistry (including TSH testing), urinalysis, physical examination, ECG and pregnancy test not required if acceptable screening assessment is performed within 7 days prior to the start of treatment on cycle 1 day 1.
- 3. **End of Study:** The end of study visit should generally occur within 7 days (+/- 1 day) of the last dose of TRC105. Assessments other than pharmacokinetics, immunogenicity and protein biomarkers do not need to be repeated if performed within the previous 2 weeks (previous 8 weeks for radiologic tumor assessments). Follow-up visits should occur 28 days following the last dose of TRC105 study drug as outlined in the Schedule of Assessments.
- 4. **Informed Consent:** Must be obtained prior to undergoing any study specific procedure and may occur prior to the 28-day screening period.
- 5. **Medical and Oncologic History, Demographics and Baseline Signs and Symptoms:** All information related to prior anticancer treatment should be recorded. Significant medical history and baseline signs and symptoms should be captured from the date of informed consent.
- 6. Physical Examination: Examination of major body systems and ECOG performance status.
- 7. **Vital Signs:** Heart rate, temperature, blood pressure, respiratory rate, weight. Assessment during TRC105 Infusions: Vital signs are to be assessed pre-infusion (i.e., within 30 minutes of starting the infusion) every 30 minutes during the infusion (+/- 15 minutes) and at the end of the infusion (i.e. within 30 minutes after completing the infusion). Vital signs should be monitored more frequently and/or beyond the completion of the infusion if medically indicated (e.g. if the patient experiences an infusion reaction that has not yet resolved).
- 8. **Hematology, Chemistry & Coagulation:** Testing to be performed locally. Thyroid stimulating hormone to be tested at screening, day 1 of each cycle and at the end of study visit. Cycle 1 day 1 assessments only need to be performed if screening assessments were performed more than 7 days prior to cycle 1 day 1. Iron studies (FE) to be performed according to the schedule of assessments and as clinically indicated during the study. Lab assessments may be performed within 3 days prior to TRC105 dosing. In addition to the assessments scheduled for the clinical trial, patients should undergo assessment as appropriate to ensure safe treatment. See Section 8.1.1.1 for specific panel collection requirements.
- 9. **Pregnancy Test:** Testing to be performed locally. All female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days of cycle 1 day 1 and 28 days following the last dose of TRC105.
- 10. **Urinalysis:** To be performed locally. Cycle 1 day 1 urinalysis only needs to be performed if screening urinalysis was performed more than 7 days prior to cycle 1 day 1. Microscopic analysis and/or urine protein creatinine ratio or 24-hour urine protein collection should be performed as clinically indicated.
- 11. **TRC105 Administration:** Intravenous TRC105 diluted in normal saline will be administered every 7 days. The first weekly TRC105 dose will be given on cycle 1 day 1 and split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4. The entire weekly dose of TRC105 (10 mg/kg) is then given on cycle 1 day 8 and weekly thereafter. See Section 6.1.6 for specific TRC105 administration guidelines.
  - Upon completion of enrollment of phase 1b dose levels 3 and notification by the sponsor, active patients that are past cycle 2, may be switched to an every 2 week dosing schedule at the every 2 week dosing MTD.
- 12. **Pazopanib Dosing:** Oral pazopanib will be dosed once daily at 800 mg starting on cycle 1 day 1 in the absence of toxicity on days 1-28 of each 28 day cycle according to the pazopanib package insert. Dose reductions are allowed based on individual patient tolerability beginning with cycle 1. See Section 6.2 for specific dosing guidelines. Pazopanib should be dosed following PK collection on cycle 1 day 1 and day 1 of even cycles.
- 13. **CT or MRI Tumor Imaging:** Images of the chest, abdomen, and pelvis to be performed at screening, and on-study as outlined in the assessment table. Known areas of disease should be consistently followed throughout the study. Assessments should be performed whenever disease progression is suspected. Allowable window for tumor imaging studies is +/- 7 days. Brain and bone scans are to be performed if metastases are suspected at screening or during study therapy. Color photography with caliper or ruler measurements, when possible, should be used to assess cutaneous tumors (target lesions).

- 14. **12-Lead ECG:** Single tracing 12-lead ECG will be performed at screening and at the time-points indicated in the Schedule of Assessments (pre-dose). If the patient develops an arrhythmia, the ECG should be repeated on day 1 of each subsequent cycle. For a QTc >500 ms, a repeat ECG for confirmation and evaluation of the ECG by a cardiologist is recommended. Additional ECGs may be performed on study as clinically indicated.
- 15. **Concomitant Medications and Treatments:** Concomitant medications and treatments will be recorded from 28 days prior to the start of study treatment and up to 28 days following the last dose of study treatment. Required TRC105 premedications should be recorded on TRC105 premedications CRF.
- 16. **Adverse Events:** Patients must be followed for adverse events from the first day of treatment with pazopanib or TRC105 study drug until at least 28 days after the last dose of TRC105 or pazopanib study drug treatment, or until all serious or TRC105 related toxicities have resolved or are determined to be "chronic" or "stable", whichever is later. "Baseline-signs and symptoms" will be recorded from the date of informed consent on corresponding case report forms. Any serious AE that is possibly related to TRC105 occurring from the time of first TRC105 dose or at any point after the reporting period must be promptly reported to TRACON.
- 17. **Anti-Product Antibodies:** 5 mL blood sample will be collected to assess Anti-Product Antibodies at the time-points indicated in the schedule of assessments and stored at approximately -70°C to be analysed by a central laboratory. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional Anti-Product Antibody samples may also be collected at the time of unexpected clinical events.
- **18. TRC105** and **Pazopanib Pharmacokinetics Trough Concentration:** A 5 mL blood sample each for TRC105 and pazopanib pharmacokinetics to be collected at the time-points indicated in the Schedule of Assessments, prior to starting the TRC105 infusion and prior to pazopanib dosing. Samples will be stored at approximately -70°C. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional PK samples may also be collected at the time of unexpected clinical events.
- 19. **Protein Biomarkers:** One 10 mL purple top (K<sub>3</sub>EDTA) tube will be collected at the time-points indicated in the schedule of assessments and stored at approximately -70°C to be analysed by a central laboratory. See separate laboratory guide for further collection and shipment information.
- 20. **Archival Tumor Tissue:** Archival specimens (formalin-fixed, paraffin-embedded) are required of the primary cancer and/or metastatic cancer specimen for each study participant. It is preferable that the entire paraffin block be submitted, but if this is not feasible, then at least 20 unstained slides are requested for immunohistochemical analysis (sections of 5 microns are preferred). See separate laboratory guide for further collection and shipment information.
- 21. Cycle 2+ Treatment: Patients who demonstrate a response of CR, PR or SD will be eligible for additional treatment until progression.
- 22. **Follow-up:** The follow-up visit should occur 28 days following the last dose of TRC105. The allowable visit window is +/- 7 days.
- 23. Allowable window for each visit within the cycle is +/- 2 days unless otherwise stated.

Table 7: Schedule of Assessments Phase 2 Angiosarcoma Cohorts 1 &2

| | Screening | | C | ycle 1 [23 | R1 | | | Cycle 2 | 2 [23] | | | Cycle 3+ | [21] [23 | 31 | | 28 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Corcerning | Day 1 | Day4 | Day<br>8 | Day<br>15 | Day<br>22 | Day<br>1 | Day<br>8 | Day<br>15 | Day<br>22 | Day 1 | Day<br>8 | Day<br>15 | Day<br>22 | End<br>of<br>Study | Day<br>Follow<br>-up |
| Protocol Activities | Day -28 | [1] [2] | [1] | [1] | [1] | [1] | [1] | [1] | [1] | [1] | [1] | [1] | [1] | [1] | [3] | [22] |
| Baseline Documentation | , | | | | | | | | | | | | | Ì | | |
| Informed Consent [4] | X | | | | | | | | | | | | | | | |
| Medical/Oncology History [5] | X | | | | | | | | | | | | | | | |
| Baseline Signs and Symptoms [5] | X | | | | | | | | | | | | | | | |
| Physical Examination [6] | Х | Х | | | | | Х | | | | Х | | | | Х | |
| Vital Signs [7] | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | |
| Laboratory Studies | | | | | | | | | | | | | | | | |
| Hematology [8] | X+Fe | Х | | | Х | | Х | | X | | Х | | Х | | Х | |
| Coagulation [8] | Х | Х | | | | | | | | | | | | | | |
| Blood Chemistry [8] | X+TSH | X +<br>TSH | | | Х | | X +<br>TSH | | | | X +<br>TSH | | | | X+<br>TSH | |
| Pregnancy Test [9] | Day -7 | | | | | | X | | | | Χ | | | | | X |
| Urinalysis [10] | X | Х | | | | | Х | | | | Х | | | | X | |
| Treatment w/ Study Drug | | | | | | | | | | | | | | | | |
| TRC105 WEEKLY Dosing [11] | | X Split | X Split | Χ | Х | X | Х | Χ | Χ | Х | Χ | Х | Χ | Χ | | |
| *TRC105 EVERY 2 WEEK | | | | | | | | | | | | | | | | |
| Dosing [11] | | X Split | X Split | X | X | X | Х | | Χ | | Х | | X | | | |
| Pazopanib for <b>Angiosarcoma</b><br><b>cohort 1</b> [12] | | | | | | | | | | | | ssion o | ne of dis<br>on singl<br>2105 | sease<br>e-agent | | |
| Pazopanib for <b>Angiosarcoma cohort 2</b> [12] | | | | | | Daily s | starting | on Cycl | e 1 Day | 1 | | | | | | |
| Tumor Assessments | | | | | | | | | | | | | | | | |
| CT or MRI Scans [13] | X | | | | | Every 6 | 3 weeks 1 | rom cyc | le 1 day | y 1 | | | | | X | |
| Other Clinical Assessments | | | | | | | | | | | | | | | | |
| 12-Lead ECG [14] | X | X | | | X | | | | | | | | | | Х | |
| Concomitant | | | | | | | | | | | | | | | | |
| Medications/Treatments [15] | Х | X | X | X | X | Х | X | X | X | X | X | X | X | X | X | X |
| Adverse Events [16] | | Х | Х | Х | Х | Х | Х | Χ | Χ | X | Х | Х | Х | Х | Х | X |
| Special Laboratory Assessments | | | | | | | | | | | | | | | | |
| | | | | | | | | | | | X &<br>Even | | | | | |
| Trough PK [17] | | | Х | X | Х | | Х | | Х | | Cycles | | | | Х | Х |
| TRC105 Peak PK [17] | | Х | Х | Х | | ] | ] | | | | | | | | | ] |
| Anti-product antibodies [18] | | Х | | | | | Х | | | | Even<br>Cycles | | | | Х | Х |
| Protein Biomarkers [19] | | Х | | | | | Х | | | | Even<br>Cycles | | | | Х | |
| Archival Tumor Tissue [20] | Х | | | | | | | | | | | | | | | |

\* TRC105 may be administered every two weeks starting with cycle 2 day 1 once it is determined that the every two week dosing MTD has not been exceeded. **SPONSOR WILL SEND NOTIFICATION TO PROCEED WITH EVERY TWO WEEK DOSING.** TRC105 will be administered weekly during cycle 1. The first weekly TRC105 dose will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4. Starting on cycle 2 day 1 and beyond, TRC105 may be administered every two weeks on days 1 and 15 at the every two-week dosing MTD. See Section 6.1.6

#### Schedule of Assessments Footnotes Phase 2 Angiosarcoma Cohort

- 1. **Days of Treatment with TRC105:** All assessments should be performed prior to the TRC105 infusion unless otherwise indicated. Each cycle is 28 days in duration.
- 2. **Cycle 1 day 1:** Hematology (including iron studies), blood chemistry (including TSH testing), urinalysis, physical examination, ECG and pregnancy test not required if acceptable screening assessment is performed within 7 days prior to the start of treatment on cycle 1 day 1.
- 3. **End of Study:** The end of study visit should generally occur within 7 days (+/- 1 day) of the last dose of TRC105. Assessments other than pharmacokinetics, immunogenicity and protein biomarkers do not need to be repeated if performed within the previous 2 weeks (previous 8 weeks for radiologic tumor assessments). If the patient permanently discontinues all study therapy due to AE, patient decision, investigator decision or any other reason the end of study assessments should be completed. **Note that in this cohort, disease progression refers to disease progression while receiving TRC105 plus pazopanib combination therapy**. Follow-up visits should occur 28 days following the last dose of TRC105 study drug as outlined in the Schedule of Assessments.
- 4. Informed Consent: Must be obtained prior to undergoing any study specific procedure and may occur prior to the 28-day screening period.
- 5. **Medical and Oncologic History, Demographics and Baseline Signs and Symptoms:** All information related to prior anticancer treatment should be recorded. Significant medical history and baseline signs and symptoms should be captured from the date of informed consent.
- 6. **Physical Examination:** Examination of major body systems and ECOG performance status.
- 7. **Vital Signs:** Heart rate, temperature, blood pressure, respiratory rate, weight. Assessment during TRC105 Infusions: Vital signs are to be assessed preinfusion (i.e., within 30 minutes of starting the infusion) every 30 minutes during the infusion (+/- 15 minutes) and at the end of the infusion (i.e. within 30 minutes after completing the infusion). Vital signs should be monitored more frequently and/or beyond the completion of the infusion if medically indicated (e.g. if the patient experiences an infusion reaction that has not yet resolved). If TRC105 administration is switched to every two week dosing, clinic visits are required only on days of TRC105 infusion (i.e., days 1 and 15 of each every two week administration cycle).
- 8. **Hematology, Chemistry & Coagulation:** Testing to be performed locally. Thyroid stimulating hormone to be tested at screening, day 1 of each cycle and at the end of study visit. Cycle 1 day 1 assessments only need to be performed if screening assessments were performed more than 7 days prior to cycle 1 day 1. Iron studies (FE) to be performed according to the schedule of assessments and as clinically indicated during the study. Lab assessments may be performed within 3 days prior to TRC105 dosing. In addition to the assessments scheduled for the clinical trial, patients should undergo assessment as appropriate to ensure safe treatment. See Section 8.1.1.1 for specific panel collection requirements.
- 9. **Pregnancy Test:** Testing to be performed locally. All female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days of cycle 1 day 1, day 1 of every cycle starting with cycle 2, and 28 days following the last dose of TRC105.
- 10. **Urinalysis:** To be performed locally. Cycle 1 day 1 urinalysis only needs to be performed if screening urinalysis was performed more than 7 days prior to cycle 1 day 1. Microscopic analysis and/or urine protein creatinine ratio or 24-hour urine protein collection should be performed as clinically indicated.
- 11. **TRC105 Administration:** Intravenous TRC105 diluted in normal saline will be administered as outlined in the assessments table. See Section 6.1.6 for specific TRC105 administration guidelines.
  - Angiosarcoma cohort 1: The first weekly TRC105 dose will be given on cycle 1 day 1 and split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4. The entire weekly dose of TRC105 (10 mg/kg) is then given on cycle 1 day 8 and weekly thereafter.

- Active patients that are past cycle 1, may be switched to an every 2 week dosing schedule at a TRC105 dose of 15 mg/kg every 2 weeks (day 1 and day 15 of each 28 day cycle) once sponsor sends notification to proceed with every two week dosing.
- Angiosarcoma cohort 2: TRC105 will be administered at a dose of 10 mg/kg weekly during cycle 1. The first weekly TRC105 dose (10 mg/kg) will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4. Starting on cycle 2 day 1 and beyond, TRC105 will be administered every two weeks on days 1 and 15 at a dose of 15 mg/kg.
- 12. **Pazopanib Dosing: Angiosarcoma cohort 1--**Oral pazopanib will be dosed orally at 800 mg starting at the time of disease progression on TRC105 single-agent and once daily thereafter in the absence of toxicity. Dose reductions are allowed based on individual patient tolerability beginning with cycle 1. **Angiosarcoma cohort 2--**Oral pazopanib will be given orally at 800 mg starting cycle 1 day 1 and once daily thereafter in the absence of toxicity. See Section 6.2 for specific dosing guidelines. Pazopanib should be dosed following PK collection on days when PK sampling is required as noted in the scheduled of assessments.
- 13. **CT or MRI Tumor Imaging:** Images of the chest, abdomen, and pelvis to be performed at screening, and on-study as outlined in the assessment table. Known areas of disease should be consistently followed throughout the study. Assessments should be performed whenever disease progression is suspected. Allowable window for tumor imaging studies is +/- 7 days. Brain and bone scans are to be performed if metastases are suspected at screening or during study therapy. Color photography with caliper or ruler measurements, when possible, should be used to assess cutaneous tumors (target lesions).
- 14. **12-Lead ECG:** Single tracing 12-lead ECG will be performed at screening and at the time-points indicated in the Schedule of Assessments (pre-dose). If the patient develops an arrhythmia, the ECG should be repeated on day 1 of each subsequent cycle. For a QTc >500 ms, a repeat ECG for confirmation and evaluation of the ECG by a cardiologist is recommended. Additional ECGs may be performed on study as clinically indicated.
- 15. **Concomitant Medications and Treatments:** Concomitant medications and treatments will be recorded from 28 days prior to the start of study treatment and up to 28 days following the last dose of study treatment. Required TRC105 premedications should be recorded on TRC105 premedications CRF.
- 16. Adverse Events: Patients must be followed for adverse events from the first day of treatment with pazopanib or TRC105 study drug until at least 28 days after the last dose of TRC105 or pazopanib study drug treatment, or until all serious or TRC105 related toxicities have resolved or are determined to be "chronic" or "stable", whichever is later. "Baseline-signs and symptoms" will be recorded from the date of informed consent on corresponding case report forms. Any serious AE that is possibly related to TRC105 occurring from the time of first TRC105 dose or at any point after the reporting period must be promptly reported to TRACON.
- 17. **TRC105** and Pazopanib Pharmacokinetics Trough and TRC105 Peak Concentration: A 5 mL blood sample each for TRC105 and pazopanib pharmacokinetics to be collected at the time-points indicated in the Schedule of Assessments. Trough samples should be collected prior to starting the TRC105 infusion and prior to pazopanib dosing (once pazopanib dosing begins for angiosarcoma cohort 1). TRC105 peak samples to be collected within 10 minutes of the completion of the TRC105 infusion on the days specified in the schedule of assessments. Samples will be stored at approximately -70°C. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional PK samples may also be collected at the time of unexpected clinical events.
- 18. **Anti-Product Antibodies:** 5 mL blood sample will be collected to assess Anti-Product Antibodies at the time-points indicated in the schedule of assessments and stored at approximately -70°C to be analysed by a central laboratory. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional Anti-Product Antibody samples may also be collected at the time of unexpected clinical events.
- 19. **Protein Biomarkers:** One 10 mL purple top (K<sub>3</sub>EDTA) tube will be collected at the time-points indicated in the schedule of assessments and stored at approximately -70°C to be analysed by a central laboratory. See separate laboratory guide for further collection and shipment information.
- 20. **Archival Tumor Tissue:** Archival specimens (formalin-fixed, paraffin-embedded) are required of the primary cancer and/or metastatic cancer specimen for each study participant. It is preferable that the entire paraffin block be submitted, but if this is not feasible, then at least 20 unstained slides are requested for immunohistochemical analysis (sections of 5 microns are preferred). See separate laboratory guide for further collection and shipment information.

### IND 131053

#### 5.3.5.2 Clinical Protocol

- 21. Cycle 2+ Treatment: Angiosarcoma cohort 1 patients will be eligible for single-agent TRC105 until progression. At the time of progression by RECIST 1.1 on single-agent TRC105, patients will transition to treatment with the combination of TRC105 and pazopanib. Angiosarcoma cohort 2 patients will be eligible for treatment with the combination until progression.
- 22. **Follow-up:** The follow-up visit should occur 28 days following the last dose of TRC105. The allowable visit window is +/- 7 days.
- 23. Allowable window for each visit within the cycle is +/- 2 days unless otherwise stated.

### 5. SELECTION AND WITHDRAWAL OF PATIENTS

For the Phase 1b dose levels -1, 1, 2 and expansion cohort 1, prior to administration of TRC105 on cycle 2 day 1, all study patients must maintain eligibility criteria indicating adequate organ function, medical status and ECOG performance status (i.e., all patients must maintain inclusion criterion #6, 8, 9 and 10 and exclusion criteria #8-21 to continue into cycle 2).

### **5.1.** Patient Inclusion Criteria

- 1. Histologically confirmed unresectable soft tissue sarcoma (i.e., non-GIST, non-adipocytic) that has progressed following treatment with chemotherapy. Prior pazopanib is allowed if the drug was not discontinued for toxicity (Phase 1b only)
- 2. Histologically confirmed metastatic soft tissue sarcoma (i.e., non-GIST, non-adipocytic) that has progressed by RECIST following treatment with anthracycline chemotherapy. Patients may have received up to four lines of systemic therapy for metastatic disease and no more than two lines of combination treatment (Phase 2 only)
- 3. Histologically confirmed locally advanced (e.g. unresectable) or metastatic angiosarcoma that has progressed following treatment with prior systemic therapy. Progression must be documented on or following the most recent systemic therapy. Prior pazopanib is allowed if the drug was not discontinued for toxicity (Phase 2 angiosarcoma cohort only)
- 4. Measurable disease by RECIST
- 5. Age of 12 years or older (patient must weigh  $\geq$  40 kg)
- 6. ECOG performance status  $\leq 1$
- 7. Resolution of all acute adverse events resulting from prior cancer therapies to NCI CTCAE grade ≤ 1 or baseline (except alopecia or neuropathy)
- 8. Adequate organ function as defined by the following criteria:
  - Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5 x ULN in cases of liver metastases
  - Total serum bilirubin  $\leq 1.5$  times the upper limit of normal
  - Absolute neutrophil count (ANC)  $\geq 1500/\mu L$
  - Platelets  $\geq 100,000/\mu L$  without transfusion support within the past 28 days
  - Hemoglobin  $\geq$  9.0 g/dL without transfusion support within the past 14 days (erythropoietin or darbepoietin permitted)
  - Serum creatinine ≤ 1.5 times the upper limit of normal or creatinine clearance > 30 mL/min by Cockcroft-Gault formula
  - INR from 0.8 to 1.2

# IND 131053

### 5.3.5.2 Clinical Protocol

- 9. Willingness and ability to consent for self to participate in study
- 10. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
- 11. Available archival tumor specimen of the soft tissue sarcoma that meets inclusion criterion #1, #2 or #3

### 5.2. Exclusion Criteria

- 1. Prior treatment with TRC105
- 2. Prior treatment with a VEGFR TKI (including pazopanib) (Part 2 only)
- 3. Current treatment on another therapeutic clinical trial
- 4. Receipt of systemic anticancer therapy, including investigational agents, within 28 days of starting study treatment. If anticancer therapy was given within 28 days of starting study treatment, patients may be included if 5 times the elimination half-life of the drug has passed.
- 5. No major surgical procedure or significant traumatic injury within 6 weeks prior to study registration, and must have fully recovered from any such procedure; date of surgery (if applicable) or the anticipated need for a major surgical procedure within the next six months. Note: the following are not considered to be major procedures and are permitted up to 7 days before therapy initiation: Thoracentesis, paracentesis, port placement, laparoscopy, thorascopy, tube thoracostomy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, incisional biopsies, imaging-guided biopsy for diagnostic purposes, and routine dental procedures
- 6. Patients who have received wide field radiotherapy ≤ 28 days (defined as > 50% of volume of pelvic bones or equivalent) or limited field radiation for palliation < 14 days prior to study registration or those patients who have not recovered adequately from side effects of such therapy
- 7. Uncontrolled chronic hypertension defined as systolic > 150 or diastolic > 90 despite optimal therapy (initiation or adjustment of BP medication prior to study entry is allowed provided that the average of 3 BP readings at a visit prior to enrollment is < 150/90 mm Hg)
- 8. Significant ascites, pericardial or pleural effusion
- 9. History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease. Patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered for at least 28 days.
- 10. Angina, MI, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, PTCA or CABG within the past 6 months. Deep venous thrombosis within 6 months, unless the patient is anti-coagulated without the use of warfarin for at least 2 weeks. In this situation, low molecular weight heparin is preferred.

- 11. Active bleeding or pathologic condition that carries a high risk of bleeding (e.g. hereditary hemorrhagic telangiectasia). Patients who have been uneventfully anti-coagulated with low molecular weight heparin are eligible.
- 12. Thrombolytic use (except to maintain i.v. catheters) within 10 days prior to first day of study therapy
- 13. Known active viral or nonviral hepatitis or cirrhosis
- 14. History of hemorrhage or hemoptysis (> ½ teaspoon bright red blood) within 3 months of starting study treatment
- 15. History of peptic ulcer within 3 months of treatment, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 28 days of starting study treatment
- 16. History of gastrointestinal perforation or fistula in the past 6 months, or while previously on antiangiogenic therapy, unless underlying risk has been resolved (e.g., through surgical resection or repair)
- 17. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
- 18. Receipt of a strong CYP3A4 inducer within 12 days prior to cycle 1 day 1 or a strong CYP3A4 inhibitor within 7 days prior to cycle 1 day 1 (Table 14)
- 19. Pregnancy or breastfeeding. Female patients must be surgically sterile (i.e.: hysterectomy) or be postmenopausal, or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. All female patients of reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to first dose. Male patients must be surgically sterile or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. The definition of effective contraception will be based on the judgment of the Principal Investigator or a designated associate.
- 20. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study

#### 5.3. Patient Withdrawal Criteria

A patient should be withdrawn from study treatment if, in the opinion of the Investigator, it is medically necessary, or if it is the wish of the patient. If a patient does not return for a scheduled visit, every effort should be made to contact the patient. In any circumstance, every effort should be made to document patient outcome. Data to be collected at the end of study visit are described in the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7). Patients will be followed for at least 28 days after the last dose of TRC105 study drug for adverse events. If the patient withdraws consent, no further evaluations should be performed, and no attempts should be made to collect additional data. In addition, patients will be withdrawn from treatment in the case of:

- 1. RECIST 1.1-defined disease progression. In cases where RECIST cannot be applied, progression should be based on unequivocal evidence of progressive disease sufficient to require a change in therapy. In the angiosarcoma cohort 1, disease progression for withdrawal refers to disease progression while receiving TRC105 plus pazopanib combination therapy.
- 2. A need for surgery, radiation, or for other anticancer therapy not specified in the protocol.
- 3. Unable to tolerate pazopanib during cycle 1 (phase 1b, dose levels -1, 1, 2 and expanded cohort 1 only).
- 4. Lost to follow-up or noncompliant.
- 5. Any TRC105 dose delay > 2 days between cycle 2 day 1 and cycle 2 day 28 (phase 1b only).
- 6. Pregnancy. Pregnant patients should be followed for the duration of the pregnancy and the outcome of the pregnancy should be documented.
- 7. Arterial thrombosis of any grade (including cerebrovascular ischemia, cardiac ischemia/infarction, or peripheral or visceral arterial ischemia) or grade 3 or 4 venous thrombosis (including pulmonary embolism).
- 8. Missed study drug treatment for > 8 consecutive weeks (i.e., both TRC105 and pazopanib dosing held). However, patients who cannot tolerate pazopanib or TRC105 therapy and who demonstrate a response of complete response (CR), partial response (PR) or stable disease (SD) with the combination and are thought to benefit from continued single agent therapy may continue on study on TRC105 or pazopanib alone.

#### 6. TREATMENT OF PATIENTS

### 6.1. Description of TRC105 Study Drug

TRC105 is a genetically engineered human/murine chimeric monoclonal antibody directed against human CD105 found on the surface of proliferating endothelial cells.

#### 6.1.1. Composition of TRC105

TRC105 is an IgG1, kappa immunoglobulin containing murine light- and heavy-chain variable region sequences and human constant region sequences. TRC105 has an approximate molecular weight of 148 kDa.

### 6.1.2. TRC105 Dose Level

#### 6.1.2.1. Phase 1b

Each patient will be dosed with 6 (Dose Level -1), 8 (Dose Level 1) or 10 mg/kg (Dose Level 2), or 15 mg/kg (Dose Level 3) The maximum weight that should be used for purpose of dose calculation is 85 kg for women and 100 kg for men. Thus, the maximum dose that should be given to a woman at the 10 mg/kg dose is 850 mg and at the 15 mg/kg dose is 1275 mg, and the maximum dose that should be given to a man at the 10 mg/kg dose is 1000 mg and at the 15 mg/kg dose is 1,500 mg. TRC105 is distributed according to lean body mass rather than overall body weight. Patients who are overweight would be at risk for high serum levels of TRC105 if the doses were not capped. Eighty-five kg for women and 100 kg for men represent accepted maximum lean body masses for the two genders.

For dose levels -1, 1, 2, and expanded cohort 1the first weekly TRC105 dose will be given on cycle 2 day 1 following two, three, or four weeks of treatment with pazopanib alone. The first weekly dose will be split into two doses whereby 3 mg/kg will be administered on cycle 2 day 1 and the balance will be administered on cycle 2 day 4). The entire weekly dose of TRC105 (6, 8 or 10 mg/kg) is then given on cycle 2 day 8 and weekly thereafter in combination with oral pazopanib.

For dose levels 3and expanded cohort 2, TRC105 dosing will begin on cycle 1 day 1 with the first weekly dose split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and 7 mg/kg is administered on cycle 1 day 4. The entire weekly dose of TRC105 at 10 mg/kg is then given on cycle 1 day 8 and weekly until cycle 2 day 1 when TRC105 is administered at 15 mg/kg every two weeks. The DLT evaluation period, for purposes of dose escalation, will be cycle 2. Each cycle will be 28 days in duration.

#### 6.1.2.2. Phase 2

Each patient, including patients in the angiosarcoma cohort, will be dosed with 10 mg/kg up to a maximum dose of 850 mg of TRC105 for women and 1,000 mg of TRC105 for men (i.e., 85 kg for women and 100 kg for men is the maximum weight that should be used for purposes of dose calculation on this study). TRC105 is distributed according to lean body mass rather than overall body weight. Patients who are overweight would be at risk for high serum levels of TRC105 if the doses were not capped. 85 kg for women and 100 kg for men represent accepted

maximum lean body masses for the two genders. The first weekly TRC105 dose will be given on cycle 1 day 1. The first weekly dose will be split into two doses whereby 3 mg/kg will be administered on cycle 1 day 1 and the balance will be administered on cycle 1 day 4. The entire weekly dose of TRC105 (10 mg/kg) is then given on cycle 1 day 8 and weekly thereafter. Each cycle following will be 28 days in duration.

TRC105 may be administered every two weeks starting with cycle 2 day 1, once it is determined that the every two week dosing MTD has not been exceeded. SPONSOR <u>WILL</u> SEND NOTIFICATION TO PROCEED WITH EVERY TWO WEEK DOSING.

- TRC105 will be administered at 10 mg/kg weekly during cycle 1.
  - The first weekly TRC105 dose (10 mg/kg) will be split into two doses whereby 3 mg/kg is administered on cycle 1 day 1 and the balance is administered on cycle 1 day 4.
- Starting on cycle 2 day 1 and beyond, TRC105 may be administered every two weeks on days 1 and 15 at 15 mg/kg.

### 6.1.3. TRC105 Packaging and Labeling

TRC105 may be provided in one or more of the following presentations.

Phosphate Buffered Saline Formulation (7 mg TRC105/mL)

210 mg TRC105/30 mL single-use vial

20 mM L-Histidine/L-Histidine Monohydrochloride, 240 mM Trehalose, 0.01% Polysorbate 20 Formulation (25 mg TRC105/mL)

100 mg TRC105/4 mL single-use vial

200 mg TRC105/8 mL single-use vial

400 mg TRC105/16 mL single-use vial

#### 6.1.4. TRC105 Storage and Shipping

TRC105 must be stored upright between 2 °C and 8 °C (36 °F to 46 °F) and protected from light.

#### 6.1.5. TRC105 Preparation

TRC105 will be prepared in the pharmacy and diluted into normal saline using appropriate aseptic technique. TRC105 will be administered using an in-line 0.2 micron filter. No incompatibilities between TRC105 and polyvinyl chloride or polyolefin bags have been observed. Multiple vials will be required for a single dose. The following formulae should be used to calculate the volume of TRC105 to be added to normal saline:

• Patient weight (kg) × dose level (mg/kg) divided by TRC105 concentration (mg/mL) = volume of TRC105 (mL) to be administered.

The volume of TRC105 that is to be administered can be rounded up or down to the nearest 1.0 mL; in the case of an increment of 0.5 mL the volume should be rounded up. **The maximum** 

weight that should be used for dose calculation in this study is 85 kg for women and 100 kg for men (note: there is not a weight restriction for enrollment purposes). If the patient's weight changes by > 10% during the study, the dose of TRC105 will be recalculated. At that time a new baseline weight will be established such that subsequent weight changes by >10% from the new baseline weight would require further recalculation of the TRC105 dose. The calculated volume of TRC105 will be diluted with normal saline. Appropriate judgment should be exercised in withdrawing an adequate amount of saline necessary to permit injection of the appropriate volume of antibody into a normal saline bag in accordance with the dose needed. The final TRC105 concentration must be between 0.6 mg/mL and 10 mg/mL. The prepared TRC105 must be gently inverted several times in order to ensure a homogeneous solution. The diluted infusion solution of TRC105 should be used within 8 hours of preparation if stored at room temperature, or within 24 hours of dilution if stored at 2° to 8°C (36° to 46°F). The expiration time should be labeled on the bag. If the diluted infusion solution of TRC105 cannot be infused within 8 hours of preparation (i.e.: the prepared infusion is at room temperature for more than 8 hours), a second bag will be prepared that contains the balance of the planned dose that was not already delivered. The prepared solution should not be frozen.

#### 6.1.6. TRC105 Administration

Patients should be encouraged to drink abundant fluid (e.g., two eight ounce glasses of water or juice) prior to the first treatment. Intravenous hydration prior to and during therapy is left to the discretion of the Investigator, but should be considered for patients that may be volume depleted.

The following TRC105 premedications should be administered 2 hours to 30 minutes prior to the start of each infusion:

- Acetaminophen 650 mg p.o. x 1
- Methylprednisolone 100 mg i.v. will be given prior to the cycle 1 day 1 and cycle 1 day 4 infusions. In addition, methylprednisolone will be given in the case of a delay of ≥ 10 days between any two scheduled weekly doses or in the case of a delay of ≥ 17 days between any two scheduled every other week doses, or if the patient develops an infusion reaction ≥ grade 2 during the immediate prior infusion.
- Famotidine 20 mg i.v. or p.o. (or similar H2 blocker) x 1. Famotidine (or similar H2 blocker) may be discontinued starting with Cycle 2 for weekly dosing, Cycle 3 for every two week dosing, in the absence of infusion reactions with the prior dose.
- Cetirizine 10 mg i.v. or p.o. x 1 (or similar oral or intravenous antihistamine). Cetirizine (or similar oral or intravenous antihistimine) may be discontinued starting with Cycle 2 for weekly dsoing, Cycle 3 for every two week dosing, in the absence of infusion reactions with the prior dose.

TRC105 infusions will begin 2 hours to 30 minutes following the completion of the TRC105 premedication, including the methylprednisolone infusion.

TRC105 will be administered intravenously utilizing an infusion pump. TRC105 has been demonstrated to be compatible with polyethylene lined, non-DEHP infusion sets and polyvinyl chloride, non-DEHP infusion sets. TRC105 is required to be administered with a 0.2 micron downstream filter. The attachment of the infusion pump administration set to the i.v. bag and

transport of the TRC105 study drug to the patient will be performed as per standard study site procedures.

Following the appropriate premedication regimen, the first weekly TRC105 dose will be split into two doses whereby 3 mg/kg is administered (on cycle 2 day 1 for the phase 1b portion dose levels -1, 1, 2, and expansion cohort 1 and cycle 1 day 1 for the phase 1b dose levels 3, expansion cohort 2 and phase 2 portion) over 4 hours (+/- 15 minutes) and the balance (e.g., 5 mg/kg for Dose Level 1) is administered on day 4 over 2 hours (+/- 15 minutes). Do not increase the infusion rate above 25 mg/min. Thereafter, the full (e.g., 8 mg/kg for Dose Level 1) TRC105 dose will be administered i.v. weekly over 1 hour (+/- 15 minutes) (e.g., the first full dose is given on cycle 2 day 8 for the phase 1b portion and cycle 1 day 8 for the phase 2 portion).

Every two week infusions will begin on cycle 2 day 1 for phase 1b dose levels 3and expanded cohort 2. Patients must complete at least one 4 hour infusion without the development of any infusion reactions, in order to reduce the subsequent TRC105 infusion to 2 hours (+/- 15 minutes) and complete a 2 hour infusion without the development of any infusion reactions in order to reduce subsequent TRC105 infusions to 1 hour (+/- 15 minutes). See Table 8 Table 9 for ideal dosing schemas. Patients with infusion reactions of any kind should be managed appropriately (see Section 6.1.8) and are not permitted to reduce the duration of the next planned infusion.

The rate of TRC105 infusion must not exceed 25 mg/min. When the i.v. bag containing TRC105 is empty, flush the i.v. line with a 20 mL normal saline. The dose level, time of transfer to i.v. bag, and the infusion start and stop times must be recorded in the source documents.

Table 8: TRC105 10 mg/kg Weekly Ideal Dosing Schema

| | C1D1 | C1D4 | C1D8 | C1D15 | C1D22 | C2D1+ |
|---|---|---|---|---|---|---|
| TRC105 Dose (mg/kg) | 3 | 7 | 10 | 10 | 10 | 10 |
| Infusion Duration (hours) | 4 | 2 | 1 | 1 | 1 | 1 |
| Premedication | | | | | | |
| Methylprednisolone (mg) | 100 | 100 | 0 | 0 | 0 | 0 |
| Famotidine (mg) | 20 | 20 | 20 | 20 | 20 | 0 |
| Cetirizine (mg) | 10 | 10 | 10 | 10 | 10 | 0 |
| Acetaminophen (mg) | 650 | 650 | 650 | 650 | 650 | 650 |

Table 9: TRC105 15 mg/kg Every Two Weeks Ideal Dosing Schema (Ph1b Dose Level 3)

| | C1D1 | C1D4 | C1D8 | C1D15 | C1D22 | C2D1 | C2D15 | C3D1+ |
|---|---|---|---|---|---|---|---|---|
| TRC105 Dose (mg/kg) | 3 | 7 | 10 | 10 | 10 | 15 | 15 | 15 |
| Infusion Duration (hours) | 4 | 2 | 1 | 1 | 1 | 1 | 1 | 1 |
| Premedication | | | | | | | | |
| Methylprednisolone (mg) | 100 | 100 | 0 | 0 | 0 | 0 | 0 | 0 |
| Famotidine (mg) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 0 |
| Cetirizine (mg) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 0 |
| Acetaminophen (mg) | 650 | 650 | 650 | 650 | 650 | 650 | 650 | 650 |

### 6.1.7. TRC105 Dose Modification/Dose Delays

In cycle 3 and beyond (and beginning in cycle 2 of the phase 2 portion), TRC105 dose reductions are allowed for grade 3 or 4 related adverse events that resolve to grade 1 or baseline (including anemia). Treatment dose delays cannot exceed 8 consecutive weeks (i.e., both TRC105 and pazopanib dosing held). However, patients who cannot tolerate pazopanib or TRC105 therapy and who demonstrate a response of complete response (CR), partial response (PR) or stable disease (SD) with the combination and are thought to benefit from continued single agent therapy may continue on study on TRC105 or pazopanib alone per Section 5.3 of the protocol.

Table 10: Allowable TRC105 Dose Modifications

| Toxicity Attributed to TRC105 | Dose Adjustment for Next Dose of TRC105 | |
|---|---|---|
| Dose Schedule/Level | 10 mg/kg weekly | 15 mg/kg every 2 weeks |
| Grade 1 or 2 | Maintain Dose Level | Maintain Dose Level |
| Grade 3 or 4 | | |
| • 1 <sup>st</sup> appearance | 8 mg/kg weekly | 12 mg/kg every 2 weeks |
| • 2 <sup>nd</sup> appearance | 6 mg/kg weekly | 10 mg/kg every 2 weeks |
| • 3 <sup>rd</sup> appearance | 4 mg/kg weekly | 8 mg/kg every 2 weeks |
| • 4 <sup>th</sup> appearance | Discontinue TRC105 treatment permanently | Discontinue TRC105 treatment permanently* |

<sup>\*</sup>After discussion with and agreement of the Sponsor, patients receiving TRC105 every two weeks have the option to return to weekly dosing at the lowest level (i.e., 4 mg/kg weekly), if 8 mg/kg every 2 weeks is not tolerable (i.e., 4<sup>th</sup> appearance of a Grade 3 or 4 toxicity attributable to TRC105 occurs) and the investigator believes that the patient is receiving benefit from the treatment.

Patients with arterial thrombosis or grade 3 or 4 venous thrombosis should be removed from study. Patients with grade 1 or 2 venous thrombosis who require anticoagulation will have their TRC105 therapy interrupted. TRC105 therapy may resume once the following criteria are met:

- The patient is on a stable dose of heparin or low molecular weight heparin.
- The patient has a platelet count > 100,000.
- The patient has not had a hemorrhagic event of grade 2 or higher while on study.
- The patient does not have a pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels).
- The patient is benefiting from TRC105 therapy (no evidence of disease progression).

TRC105 and pazopanib should be held for two weeks prior and for two weeks following surgical procedures. However, resumption of study treatment can be shorter (but no less than 7 days) or longer than two weeks based on clinical judgement of adequate wound healing and recovery from the procedure. For **minor procedures** (e.g., port placement), TRC105 (and pazopanib) should be held for at least 1 week prior and for at least 1 week after (or until adequate healing).

TRC105 DOSING DELAY: If a patient misses a scheduled weekly TRC105 dose and dosing is resumed  $\geq 10$  days after the last dose or if a patient misses a scheduled every 2 week dose and dosing is resumed  $\geq 17$  days after the last dose, premedication (including methylprednisolone) and TRC105 are to be administered as described in Table 11. Split dosing is not required. However, it is recommended that if the patient experienced a severe headache with a previous
infusion, the first TRC105 dose upon resumption should be administered over two days as was done for the initial dose, see Table 12.

Table 11: TRC105 dosing after Dose Delay (with no split dosing)

| | CxDy | CxDy | CxDy | CxDy | CxDy+ |
|---|---|---|---|---|---|
| TRC105 Dose (mg/kg) | 10 or 15 | 10 or 15 | 10 or 15 | 10 or 15 | 10 or 15 |
| Infusion Duration (hours) | 4 | 2 | 1 | 1 | 1 |
| Premedication | | | | | |
| Methylprednisolone (mg) | 100 | 0 | 0 | 0 | 0 |
| Famotidine (mg) | 20 | 20 | 20 | 20 | 0 |
| Cetirizine (mg) | 10 | 10 | 10 | 10 | 0 |
| Acetaminophen (mg) | 650 | 650 | 650 | 650 | 650 |

Note that acetaminophen should NOT be discontinued.

Table 12: TRC105 Dosing after Dose Delay (with split dosing)

| | Day 1<br>resuming<br>TRC105 | 3 days<br>later | Weekly or<br>every 2 weeks<br>from Day 1 | Weekly or<br>every 2<br>weeks | CxDy+ |
|---|---|---|---|---|---|
| TRC105 Dose (mg/kg) | 3 | 7 or 12 | 10 or 15 | 10 or 15 | 10 or 15 |
| Infusion Duration (hours) | 4 | 2 | 1 | 1 | 1 |
| Premedication | | | | | |
| Methylprednisolone (mg) | 100 | 100 | 0 | 0 | 0 |
| Famotidine (mg) | 20 | 20 | 20 | 20 | 0 |
| Cetirizine (mg) | 10 | 10 | 10 | 10 | 0 |
| Acetaminophen (mg) | 650 | 650 | 650 | 650 | 650 |

Note that acetaminophen should NOT be discontinued.

The schedule of assessment should be followed with regards to visits, labs, and any other required assessments even if TRC105 dosing is held.

#### 6.1.8. Management of TRC105 Infusion Reactions

If a patient experiences a grade 2 or higher adverse reaction during infusion, the infusion should be interrupted and the patient treated accordingly. Antipyretic, antihistamine, antiemetic, anti-inflammatory, or other symptomatic medications including epinephrine may be administered as indicated. For grade 2 and certain grade 3 infusion reactions, the infusion may be restarted at half of the previous rate if and when the infusion reaction has resolved, and then increased per patient tolerance to a maximum of 25 mg/min. For grade 4 infusion reactions, the infusion should not be restarted and the patient should discontinue TRC105 treatment. Infusion reactions will be recorded as AEs in the case report form. Interventions should be documented as concomitant medications or concomitant treatments as appropriate.

**Table 13:** Management of TRC105 Infusion Reactions

| Infusion Reaction<br>Severity | Recommended Management |
|---|---|
| C 1- 1 (:14) | 1. No intervention |
| Grade 1 (mild) | 2. Continue infusion unless symptoms worsen |
| | 1. Interrupt infusion |
| Grade 2 (moderate) | 2. Treat with symptomatic medications <sup>a</sup> |
| Grade 2 (moderate) | <b>3.</b> Resume infusion at half the previous rate when infusion-related symptoms improve to grade 1 or less. |
| | 1. Interrupt infusion |
| | 2. Treat with symptomatic medications <sup>a</sup> |
| Grade 3 (severe) | <b>3.</b> Monitor patient until infusion-related symptoms resolve, including hospitalization if necessary |
| | <b>4.</b> Discontinue TRC105 treatment unless other factors that contributed to the infusion reaction are identified and corrected |
| | 1. Discontinue infusion |
| Grade 4 (life- | 2. Treat with symptomatic medications <sup>a</sup> |
| threatening) | 3. Hospitalize patient |
| | <b>4.</b> Discontinue TRC105 treatment |

<sup>&</sup>lt;sup>a</sup>Symptomatic medications may include but are not limited to diphenhydramine 50 mg i.v. and/or hydrocortisone 100 mg i.v. (for fever, rash, hypoxia, or other hypersensitivity reactions), meperidine 50-100 mg i.v. (for shaking chills/rigors), oxygen by mask or nasal cannula (for hypoxia), epinephrine 0.5 mg i.m. (for hypotension or bronchospasm), albuterol inhaler or nebulizer (for bronchospasm), i.v. fluids (for hypotension), and ondansetron 0.15 mg/kg i.v. (for nausea).

# 6.1.9. TRC105 Study Drug Accountability

The Investigator must maintain an accurate accounting of TRC105 supplied by TRACON. During the study, the following information must be recorded:

- Date of receipt, quantity and lot number of the TRC105 study drug received from TRACON
- ID number of the patient to whom the product is dispensed
- The date(s) and quantity of the product dispensed
- Dates and quantity of product returned, lost or accidentally or deliberately destroyed

Investigational Drug Accountability Logs should be maintained by the site and must be readily available for inspection.

# 6.1.10. TRC105 Study Drug Handling and Disposal

TRC105 must be stored upright between 2 °C and 8 °C (36 °F to 46 °F) and protected from light. The Investigator should not return clinical study materials to TRACON unless specifically instructed to do so by TRACON. Used vials do not need to be maintained. All expired vials of TRC105 should be retained until destruction is authorized by a TRACON representative. The Site Pharmacist will be responsible for documenting the destruction (according to institutional requirements) of used or expired vials.

# 6.2. Description of Pazopanib

See pazopanib package insert [67].

#### **6.2.1.** Composition of Pazopanib

See pazopanib package insert [67].

#### 6.2.2. Pazopanib Dose Level

Each patient, except for patients in the angiosarcoma cohort, will be dosed with 800 mg of pazopanib on cycle 1 day 1 and daily thereafter, in the absence of toxicity, once daily without food (at least 1 hour before or 2 hours after a meal) for each day of a 28 day cycle [67]. Note that in phase 1b dose levels 1, 2 and expanded cohort 1 only, cycle 1 will be 14 to 28 days in duration during which pazopanib will be dosed alone. Pazopanib dose reductions are allowed based on individual patient tolerability, including during the initial 2 to 4 week period of the phase 1b when pazopanib is dosed in the absence of TRC105.

Patients in the angiosarcoma cohort 1 will start pazopanib dosing at the time of disease progression on TRC105 single-agent. The starting pazopanib dose will be 800 mg daily in accordance with the package insert. Pazopanib dose reductions are allowed based on individual patient tolerability.

#### 6.2.3. Pazopanib Packaging and Labeling

See pazopanib package insert [67].

# 6.2.4. Pazopanib Storage Handling and Disposal

See pazopanib package insert [67].

# 6.2.5. Pazopanib Dosing

The recommended starting dose of pazopanib is 800 mg orally once daily without food (at least 1 hour before or 2 hours after a meal). The dose of pazopanib will not exceed 800 mg.

Do not crush tablets due to the potential for increased rate of absorption which may affect systemic exposure.

If a dose is missed, it should not be taken if it is less than 12 hours until the next dose [67].

#### 6.2.6. Pazopanib Dose Modification

Dose increase or reduction is recommended based on individual safety and tolerability. Decrease or increase should be in 200 mg steps based on individual tolerability. The dose of pazopanib will not exceed 800 mg. If a dose is missed, it should not be taken if it is less than 12 hours until the next dose. Patients who cannot tolerate pazopanib or TRC105 therapy and who demonstrate a response of complete response (CR), partial response (PR) or stable disease (SD) with the combination and are thought to benefit from continued single agent therapy may continue on study on TRC105 or pazopanib alone per Section 5.3 of the protocol.

Hepatic Impairment: No dose adjustment is required in patients with mild hepatic impairment. In patients with moderate hepatic impairment, alternatives to pazopanib should be considered. If pazopanib is used in patients with moderate hepatic impairment, the dose should be reduced to 200 mg per day. Pazopanib is not recommended in patients with severe hepatic impairment.

- Patients with isolated ALT elevations between 3 X ULN and 8 X ULN may be continued on pazopanib with weekly monitoring of liver function until ALT return to Grade 1 or baseline.
- Patients with isolated ALT elevations of >8 X ULN should have pazopanib interrupted until they return to Grade 1 or baseline. If the potential benefit for reinitiating treatment with pazopanib is considered to outweigh the risk for hepatotoxicity, then reintroduce pazopanib at a reduced dose of no more than 400 mg once daily and measure serum liver tests weekly for 8 weeks. Following reintroduction of pazopanib, if ALT elevations >3 X ULN recur, then pazopanib should be permanently discontinued.
- If ALT elevations >3 X ULN occur concurrently with bilirubin elevations >2 X ULN, pazopanib should be permanently discontinued. Patients should be monitored until resolution. pazopanib is a UGT1A1 inhibitor. Mild, indirect (unconjugated) hyperbilirubinemia may occur in patients with Gilbert's syndrome. Patients with only a mild indirect hyperbilirubinemia, known Gilbert's syndrome, and elevation in ALT >3 X ULN should be managed as per the recommendations outlined for isolated ALT elevations.

Blood pressure should be monitored and managed promptly using a combination of anti-hypertensive therapy and dose modification of pazopanib (interruption and re-initiation at a reduced dose based on clinical judgment).

Increased blood pressure should be treated promptly with standard anti-hypertensive therapy and dose reduction or interruption of pazopanib as clinically warranted. pazopanib should be discontinued if there is evidence of hypertensive crisis or if hypertension is severe and persistent

despite anti-hypertensive therapy and dose reduction. Approximately 1% of patients required permanent discontinuation of pazopanib because of hypertension [67].

Interrupt pazopanib and dose reduce for 24-hour urine protein  $\geq$ 3 grams; discontinue pazopanib for repeat episodes despite dose reductions.

Institute appropriate anti-infective therapy promptly and consider interruption or discontinuation of pazopanib for serious infections.

Interruption of therapy with pazopanib is recommended in patients undergoing surgical procedures [67]. TRC105 and pazopanib should be held for two weeks prior and for two weeks following surgical procedures. For **minor procedures** (e.g., port placement), TRC105 (and pazopanib) should be held for at least 1 week prior and for at least 1 week after (or until adequate healing).

#### 6.2.7. Pazopanib Drug Accountability

Patients will be asked to return any unused tablets from the previous cycle for proper drug accountability and destruction according to institution guidelines. A new prescription will be dispensed for the following cycle.

# **6.3.** Concomitant Medications

No other approved or investigational anticancer treatment will be permitted during the study period. No other investigational drug may be used during treatment on this protocol, and concurrent participation in another clinical trial is not allowed.

Patients who receive NSAIDs on study should also receive peptic ulcer disease (PUD) prophylaxis with an H2 or proton pump blocker.

Narcotic analgesics, nonsteroidal anti-inflammatory drugs, and triptans (e.g. sumatriptan) may be offered as needed for relief of pain or headaches. Antihistamines and decongestants may be offered for the treatment of sinus congestion.

Packed red blood cell, colony stimulating factors, and platelet transfusions should be administered as clinically indicated.

CYP3A4 Inhibitors: Avoid use of strong inhibitors (Table 14); co-administration of pazopanib with strong inhibitors of CYP3A4 increases pazopanib concentrations. Patients may not have received a strong CYP3A4 inhibitor within 7 days prior to cycle 1 day 1. If co-administration is warranted, reduce the dose of pazopanib to 400 mg.

CYP3A4 Inducers: Consider an alternate concomitant medication with no or minimal enzyme induction potential; CYP3A4 inducers may decrease plasma pazopanib concentrations. Pazopanib should not be used if chronic use of strong CYP3A4 inducers cannot be avoided. Patients may not have received a strong CYP3A4 inducer within 12 days prior to cycle 1 day 1.

CYP Substrates: Concomitant use of pazopanib with agents with narrow therapeutic windows that are metabolized by CYP3A4, CYP2D6, or CYP2C8 is not recommended.

Concomitant use of pazopanib and simvastatin increases the risk of ALT elevations and should be undertaken with caution and close monitoring.

Table 14: Strong CYP3A4 Inducers and Inhibitors<sup>a</sup>

| Inducers: | *aInhibitors: | |
|-----------------|---------------------|---------------|
| dexamethasone | Boceprevir | Conivaptan |
| phenytoin | Indinavir | Itraconazole |
| carbamazepine | Nelfinavir | Ketoconazole |
| rifampin | Lopinavir/ritonavir | Mibefradil |
| rifabutin | Saquinavir | Nefazodone |
| rifapentin | Telaprevir | Posaconazole |
| phenobarbital | Ritonavir | Voriconazole |
| St. John's Wort | Clarithromycin | Telithromycin |

<sup>&</sup>lt;sup>a</sup> Because the lists of these agents are constantly changing, it is important to regularly consult a comprehensive list such as the one located at http://medicine.iupui.edu/ clinpharm/ddis/.

# **6.4.** Treatment Compliance

# **6.4.1.** TRC105 Treatment Compliance

All TRC105 infusions will occur at the trial site under the direct supervision of the treating physician or his or her designee.

# **6.4.2.** Pazopanib Treatment Compliance

Patients will be asked to record the day and time of pazopanib home dosing on a TRACON supplied log to be reviewed by site personnel prior to initiation of each new cycle.

#### 6.5. Patient Enrollment

Patients will be manually enrolled by TRACON Pharmaceuticals and assigned an eight digit patient number. This eight digit number will be used to identify patients throughout their participation in the trial. A regulatory binder will be provided and will include detailed instructions for the manual enrollment process.

#### 7. ASSESSMENT OF EFFICACY

# 7.1. Radiological Tumor Assessment

The primary efficacy endpoint for phase 2 is PFS, defined as time from screening to either first disease progression or death from any cause per RECIST version 1.1 [68]. Patients alive at the time of analysis will be censored at the date of last disease assessment.

The primary efficacy assessment will be best overall response as defined in Section 7.1.2. The determination of antitumor efficacy will be based on objective tumor assessments made by the Investigator according to RECIST version 1.1 [68]. Investigators will make treatment decisions based on these assessments. All lesions will be classified as target or non-target lesions at the Screening visit. Each lesion designation will be maintained through the course of the study.

The same method and technique should be used to characterize each identified and reported lesion at Screening, during the study treatment period, and at the End of Study visit. Imaging-based evaluation over clinical examination is the required technique when both could be used to assess the antitumor effect of the treatment. Clinical Oncology review of all tumor measurements is desired.

Whenever possible, clinical evaluation of superficial lesions should not be used as the sole form of measurement. However, when necessary, color photograph with metric caliper is acceptable. Tumor evaluation by positron emission tomography (PET) scan or by ultrasound may not substitute for CT or MRI scans.

Radiological tumor assessments will be performed at screening, as outlined in the Schedule of Assessments (Table 4,Table 5, Table 6 and Table 7), and whenever disease progression is suspected. Another tumor assessment will be performed at the End of Study Visit if an assessment has not been performed within the prior 8 weeks. All patient files and radiological images must be available for CRF source verification.

#### 7.1.1. Measurability of Tumor Lesions

At Screening, individual tumor lesions will be categorized by the Investigator as either target or non-target according to RECIST 1.1 as described below.

- Measurable: Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with spiral CT scan. Lytic bone lesions, with an identifiable soft tissue component, evaluated by CT or MRI, can be considered measurable lesions if the soft tissue component otherwise meets the definition of measurability previously described. Blastic bone lesions are non-measurable. Lesions in previously irradiated areas (or areas treated with local therapy) should not be selected as target lesions, unless there has been demonstrated progression in the lesion. Clinical lesions will only be considered measurable when they are superficial (e.g. skin nodules, palpable lymph nodes) and ≥ 10 mm. Clinical lesions must be measured with calipers.
- Non-Measurable: All other lesions, including small lesions and bone lesions other than lytic bone lesions, leptomeningeal disease, ascites, pleural or pericardial effusions, lymphangitis of the skin or lung, abdominal masses that are not confirmed and followed by imaging techniques, previously irradiated lesions (unless there has been demonstrated

progression in the lesion), and disease documented by indirect evidence only (e.g. by laboratory tests such as alkaline phosphatase).

#### **7.1.1.1.** Recording Tumor Measurements

Measurable lesions up to a maximum of 5 lesions representative of all involved organs (with a maximum of 2 lesions per organ) should be identified as target lesions and measured and recorded at Screening and at the stipulated intervals during treatment. Target lesions should be selected on the basis of their size (lesion with the longest diameters) and their suitability for accurate repetitive measurements (either by imaging techniques or clinically). Target lesions may include lymph nodes with a short axis > 15 mm.

The longest diameter will be recorded for each target lesion (with the exception of lymph nodes, where the short axis will be used). The sum of the diameter for all target lesions at Screening will be calculated and recorded as the baseline sum diameter to be used as reference to further characterize the objective tumor response of the measurable dimension of the disease during treatment. All measurements should be performed using a caliper or ruler and should be recorded in metric notation in millimeters.

All other lesions (or sites of disease) should be identified as non-target lesions and should also be recorded at baseline. Measurements are not required and these lesions should be followed as "present", "stable", "absent", "increased" or "decreased".

#### 7.1.2. Definitions of Tumor Response

# 7.1.2.1. Target Lesions

- Complete response (CR) is defined as the disappearance of all target lesions.
- Partial response (PR) is defined as  $a \ge 30\%$  decrease in the sum of the dimensions of the target lesions taking as a reference the baseline sum dimensions.
- **Progressive disease (PD)** is defined as a ≥ 20% relative increase and ≥ 5 mm absolute increase in the sum of the dimensions of the target lesions taking as a reference the smallest sum of the dimensions recorded since the treatment started, or the appearance of one or more new lesions.
- Stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as a reference the smallest sum of the dimensions since the treatment started.

#### 7.1.2.2. Non-Target Lesions

- Complete response (CR) is defined as the disappearance of all non-target lesions.
- non-CR/non-PD is defined as a persistence of  $\geq 1$  non-target lesions.
- **Progressive disease (PD)** is defined as unequivocal progression of existing non-target lesions, or the appearance of  $\geq 1$  new lesions.

The cytological confirmation of the neoplastic origin of any effusion that appears or worsens during treatment when the measurable tumor has met criteria for response or stable disease is mandatory to differentiate between response or stable disease and progressive disease.

#### 7.1.2.3. Determination of Overall Response

#### **7.1.2.3.1.** By RECIST

When both target and non-target lesions are present, individual assessments will be recorded separately. The overall assessment of response will involve all parameters as depicted in Table 15. Per RECIST 1.1, in non-randomized trials with response as a primary endpoint, confirmation of PR or CR is required. Per RECIST 1.1, a modest increase in the size of one or more non-target lesions is usually not sufficient to qualify for unequivocal progression status.

**Table 15:** Response Evaluation Criteria in Solid Tumors

| Target Lesions <sup>a</sup> | Non-target Lesions <sup>b</sup> | New Lesions <sup>c</sup> | Overall Response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | Not Evaluable |
| PD | Any Response | Yes or No | PD |
| Any Response | PD | Yes or No | PD |
| Any Response | Any Response | Yes | PD |

<sup>&</sup>lt;sup>a</sup>Measurable lesions only.

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

NOTE: Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "Need for additional anti-cancer therapy/surgery". Every effort should be made to document the objective progression even after discontinuation of treatment.

In some circumstances, it may be difficult to distinguish residual disease from normal tissue. When the evaluation of complete response depends upon this determination, it is recommended that the residual lesion be investigated by fine needle aspirate or biopsy before confirming the complete response status.

<sup>&</sup>lt;sup>b</sup>May include measurable lesions not followed as target lesions or non-measurable lesions.

<sup>&</sup>lt;sup>c</sup>Measurable or nonmeasurable lesions.

#### 8. ASSESSMENT OF SAFETY

# 8.1. Safety Parameters

Safety will be characterized in terms of the incidence, timing, severity (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], Version 4.0), seriousness, and relatedness of adverse events and laboratory abnormalities. In addition, physical examination, vital signs, and ECOG performance status will be serially monitored. Laboratory safety analyses will be based on the local laboratory data, and will include hematology, serum chemistry (including liver and kidney function), urinalysis, serum or urine pregnancy testing, and coagulation profile. Serum will also be assessed for immunogenicity to TRC105 (including anti-product antibody titers). In addition, single tracing 12-lead ECGs will be performed at the time-points indicated in the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7). QT, PR and QRS intervals and heart rate will be captured. ECGs will also be collected as clinically indicated throughout the study.

#### 8.1.1. Laboratory Safety Assessments

Abnormal <u>and</u> clinically significant laboratory tests should be recorded as adverse events. To meet the definition of clinically significant, the test result generally requires a change in medical management (e.g. new medication, unplanned treatment, additional tests, etc.).

#### 8.1.1.1. Hematology, Serum Chemistry, Coagulation, Pregnancy Test

Assessments will be performed at the time points indicated in the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7) and analyzed at local laboratories. Investigators may have additional blood tests performed for the purpose of planning treatment administration, or for following adverse events as clinically indicated.

- Hematology: CBC with differential and platelet count. Iron studies (serum iron, ferritin and total iron binding capacity).
- Coagulation: International Normalized Ratio (INR) will be assessed
- Serum Chemistry: Total bilirubin, alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase, lipase, amylase, total protein, albumin, sodium, potassium, bicarbonate, chloride, calcium, phosphorus, blood urea nitrogen, creatinine, magnesium, thyroid stimulating hormone and glucose
- Pregnancy Test: Serum or urine pregnancy tests will be performed locally on all female patients of childbearing potential. Patients must be surgically sterile (i.e.: hysterectomy) or be postmenopausal, or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. The definition of effective contraception will be based on the judgment of the Principal Investigator or a designated associate.

#### **8.1.1.2.** Urinalysis

Urinalysis (without microscopic analysis, unless indicated) will be performed at time points indicated in the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7) and analyzed

by local laboratories. Microscopic analysis, urine protein-creatinine ratio (UPCR), and 24 urine collection for protein should be performed as clinically indicated.

#### 8.1.1.3. Physical Examination

A physical examination including, but not limited to, general appearance, head, eyes, ears, nose, throat, neck, heart, chest, abdomen, musculoskeletal, extremities, skin, lymph nodes, neurological genitourinary (as appropriate), and rectal (as appropriate) will be assessed at timepoints indicated within the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7). The physical examination will include examination of known and suspected sites of disease.

# **8.1.1.4.** Vital Signs

Heart rate, temperature, blood pressure, respiratory rate and weight will be assessed at time points indicated within the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7). Heart rate, temperature, blood pressure, and respiratory rate will also be assessed during TRC105 infusions as described in Section 4.1.2.2 and the footnotes of Table 4, Table 5, Table 6 and Table 7(Schedule of Assessments).

#### 8.1.1.5. Performance Status

The ECOG scale will be used to assess performance status at Screening.

#### 8.1.1.6. ECG

A single 12-lead (with a 10-second rhythm strip) tracing will be used for all ECGs. It is preferable that the machine used has a capacity to calculate standard intervals automatically. ECG will be performed at the time-points indicated in the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7) and as clinically indicated throughout the study.

#### 8.2. Adverse Events

All observed or volunteered adverse events regardless of suspected causal relationship to TRC105 study drug will be reported as described below.

# 8.2.1. Definition of Adverse Event

An adverse event is any untoward medical occurrence in a trial patient who is administered a drug or biologic (medicinal product); the event may or may not have a causal relationship with the medicinal product. Examples of adverse events include, but are not limited to the following:

- Clinically significant symptoms and signs including:
  - Worsening of signs and symptoms of the malignancy under trial (disease progression without worsening of signs and symptoms assessed by measurement of malignant lesions on radiographs or other methods should not be reported as adverse events).
  - O Signs and symptoms resulting from drug overdose, abuse, misuse, withdrawal, sensitivity, dependency, interaction or toxicity.

- All possibly related and unrelated illnesses, including the worsening of a preexisting illness.
- o Injury or accidents. Note that if a medical condition is known to have caused the injury or accident (hip fracture from a fall secondary to dizziness), the medical condition (dizziness) and the outcome of the accident (hip fracture from a fall) should be reported as 2 separate adverse events.
- O Symptoms or signs resulting from exposure *in utero*.
- Abnormalities in physiological testing or physical examination findings that require clinical intervention or further investigation (beyond ordering a repeat confirmatory test).
- Laboratory abnormalities that meet any of the following (Note: merely repeating an abnormal test, in the absence of any of the below conditions, does not constitute an adverse event. Any abnormal test result that is determined to be an error does not require reporting as an adverse event.):
  - o Test result that is associated with accompanying symptoms
  - Test result that requires additional diagnostic testing or medical/surgical intervention
  - Test result that leads to a change in TRC105 study drug dosing outside of protocol-stipulated dose adjustments or discontinuation from the trial, significant additional concomitant drug treatment, or other therapy
  - Test result that is considered to be an adverse event by the Investigator or TRACON

#### 8.2.2. Serious Adverse Events

An adverse event that meets one or more of the following criteria/outcomes is classified as serious:

- Results in death
- Is life-threatening (i.e., at immediate risk of death)
- Requires in patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Results in congenital anomaly/birth defect
- Other important medical events that may not result in death, be life-threatening, or
  require hospitalization may be considered serious when, based upon appropriate medical
  judgment, they may jeopardize the patient or may require medical or surgical intervention
  to prevent one of the outcomes listed above. Examples of such events are intensive
  treatment in an emergency room for allergic bronchospasm; blood dyscrasias or
  convulsions that do not result in hospitalization; or the development of drug dependence
  or drug abuse.

Serious also includes any other event that the Investigator or sponsor judges to be serious, or which is defined as serious by the HRA in the country in which the event occurred.

Progression of the malignancy under study (including signs and symptoms of progression) should not be reported as SAEs unless the outcome is fatal during the trial or within the safety reporting period. Hospitalizations due to signs and symptoms of disease progression should not be reported as SAEs. If the malignancy has a fatal outcome during the trial or within the safety reporting period, then the event leading to death must be recorded as an adverse event and as an SAE with CTC grade 5.

The onset date of an SAE is defined as the date on which the event initially met serious criteria (e.g., the date of admission to a hospital). The end date is the date on which the event no longer met serious criteria (e.g., the date the patient was discharged from a hospital).

# 8.2.2.1. Hospitalization

Adverse events associated with in-patient hospitalization, or prolongation of an existing hospitalization, are considered serious. Any initial admission, even if the duration is less than 24 hours is considered serious. In addition, any transfer within the hospital to an acute/intensive care unit is considered serious (e.g., transfer from the psychiatric wing to a medical floor or transfer from a medical floor to a coronary care unit). However, the following hospitalizations **should not** be considered serious:

- Rehabilitation facility admission
- Hospice facility admission
- Respite care
- Skilled nursing facility admission
- Nursing home admission
- Emergency room visit
- Outpatient same day surgery/procedure
- Hospitalization or prolongation of hospitalization in the absence of precipitating clinical adverse events as follows:
  - Admission for treatment of preexisting condition not associated with the development of a new adverse event or with a worsening of the preexisting condition
  - Social admission
  - o Administrative admission (e.g. for yearly physical exam)
  - o Protocol-specified admission during a clinical trial
  - Optional admission not associated with a precipitating clinical adverse event (e.g. for elective cosmetic surgery)
  - o Preplanned treatments or surgical procedures that are not related to an SAE

- Hospitalization for observation without an AE
- Diagnostic and therapeutic noninvasive and invasive procedures, such as surgery, should not be reported as adverse events. The medical condition for which the procedure was performed should be reported if it meets the definition of an adverse event (e.g. acute appendicitis that begins during the adverse event reporting period should be reported as an adverse event and the appendectomy should be recorded as a concomitant treatment).

# **8.3.** Reporting Adverse Events

#### **8.3.1.** Eliciting Adverse Event Information

The Investigator is to report all directly observed adverse events and all adverse events spontaneously reported by the trial patient using concise medical terminology. In addition, each trial patient will be questioned about adverse events at each clinic visit following initiation of treatment. The question asked will be, "Since your last clinic visit have you had any health problems?"

#### **8.3.2.** Adverse Event Reporting Period

Safety information for each patient will be collected from the date of informed consent. Adverse events occurring prior to the initiation of the study treatment with pazopanib or TRC105 study drug will be considered "baseline-signs and symptoms", will be recorded on corresponding case report forms and will not be retained for patients who fail screening. The adverse event reporting period for this trial begins when the patient has received even a portion of the first dose of pazopanib or TRC105 study drug and ends 28 days after the last dose of pazopanib or TRC105 study drug is administered.

All adverse events that occur in trial patients during the adverse event reporting period specified in the protocol must be reported to TRACON, whether or not the event is considered study treatment-related. In addition, any known untoward event that occurs beyond the adverse event reporting period that the Investigator assesses as possibly related to the investigational medication/product should also be reported as an adverse event.

#### **8.3.3.** Reporting Requirements

Each adverse event is to be classified by the Investigator as SERIOUS or NONSERIOUS. This classification of the gravity of the event determines the reporting procedures to be followed. If an SAE occurs, reporting will follow local and international regulations, as appropriate.

The Investigator must notify the Sponsor of any event that meets one of the criteria for an SAE immediately upon learning of the event. Any subsequent revisions that are made to information pertaining to serious suspected TRC105 adverse drug reactions (e.g.,: change in grade etc.), including a change in attribution to TRC105 study drug from "not related" to "suspected adverse drug reaction" should also be communicated to TRACON immediately. This notification should be made to:

#### PRIMARY MEDICAL MONITOR

Charles Theuer, MD PhD
TRACON Pharmaceuticals Inc.
8910 University Center Lane, Suite 700
San Diego, California 92122
Email: ctheuer@traconpharma.com

Cell Phone: 1.858.344.9400 Office Phone: 1.858.550.0780 x233

# **SECONDARY MEDICAL MONITOR**

Ron Shazer, MD MBA Email: <a href="mailto:rshazer@traconpharma.com">rshazer@traconpharma.com</a> Cell Phone: 1.310.922.8039

Following notification, the Investigator will report the SAE via the AE CRF via the data management system. The initial AE CRF is to be updated with more detailed adverse event information within **5 calendar days** of the event.

In the rare event that the Investigator is not immediately aware of an SAE (for example, if the study subject seeks urgent medical attention elsewhere), the Investigator is to notify the Sponsor immediately upon learning of it and document his/her first awareness.

Each SAE should be followed until resolution, or until such time as the Investigator determines its cause or determines that it has become stable. Information pertaining to follow-up of SAEs should also be sent to the TRACON Pharmaceuticals Inc.

Serious adverse events that are unexpected and associated with use of the study medication will be reported to the US Food and Drug Administration (FDA) and all participating clinical sites by TRACON via MedWatch forms. For events which are fatal or life-threatening, unexpected, and associated with use of the investigational product, a 7-Day Alert Report will be submitted to the FDA within 7 calendar days of receipt of the SAE information. For all other events that are serious, unexpected, and associated with use of the investigational product, a written report will be made no more than 15 calendar days from the date TRACON learns of the event. Participating clinical sites will be notified of these events in parallel.

All adverse events, including SAEs, are to be reported on the adverse event CRFs.

# 8.3.4. Recording Adverse Events in the Case Report Forms

The Investigator is to report all directly observed adverse events and all adverse events spontaneously reported by the trial patient. In addition, each trial patient will be questioned about adverse events. All adverse events that meet the criteria specified in Section 8.2.1 are to

be recorded on patient source documents and on the CRFs. Adverse events should be reported using concise medical terminology on the CRFs.

# 8.3.5. Grading of Adverse Event Severity

To report adverse events on the CRFs, the Investigator will use the severity grading as described in NCI CTCAE (Version 4.0).

Every effort should be made by the Investigator to assess the adverse event according to CTCAE criteria. If the Investigator is unable to assess severity because the term is not described in NCI (Version 4.0), severity of MILD, MODERATE, SEVERE, LIFE-THREATENING, or FATAL may be used to describe the maximum intensity of the adverse event. For purposes of consistency, these intensity grades are defined as follows:

**Table 16:** Adverse Event Grading

| Grade | Non-CTCAE Severity | Definition |
|---|---|---|
| 1 | Mild | Does not interfere with patient's usual function |
| 2 | Moderate | Interferes to some extent with patient's usual function |
| 3 | Severe | Interferes significantly with patient's usual function |
| 4 | Life-Threatening | Results in immediate risk of patient's death |
| 5 | Fatal | Results in patient's death |

Note the distinction between the severity and the seriousness of an adverse event. A severe event is not necessarily a serious event. For example, a headache may be severe (interferes significantly with patient's usual function) but would not be classified as serious unless it met one of the criteria for serious events.

# 8.3.6. Relationship to TRC105 Study Drug/Pazopanib

In this study, TRC105 study drug is given in combination with Pazopanib. The relationship of an adverse event to TRC105 study drug and/or Pazopanib should be classified by the Investigator using the following guidelines:

- Suspected Adverse Reaction: There is a reasonable possibility that TRC105 caused the adverse event (i.e.: there is evidence to suggest a causal relationship between TRC105 and adverse event).
- Not Related: There is no reasonable possibility that the adverse event is associated with TRC105 study drug.

AE's related to TRC105 study drug or Pazopanib are considered Adverse Drug Reactions (ADR).

#### 8.3.7. Expectedness

All TRC105 adverse events and adverse drug reactions are considered "unexpected" if it's not listed in the investigator brochure or not listed at the specificity or severity that has been observed. For example, under this definition, hepatic necrosis would be unexpected (by virtue of

greater severity) if the investigator brochure referred only to elevated hepatic enzymes or hepatitis. Similarly, cerebral thromboembolism and cerebral vasculitis would be unexpected (by virtue of greater specificity) if the investigator brochure listed only cerebral vascular accidents. "Unexpected," as used in this definition, also refers to adverse events or suspected adverse reactions that are mentioned in the investigator brochure as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the particular drug under investigation.

All Pazopanib adverse events and adverse drug reactions are considered "unexpected" if it's not listed in the package insert or not listed at the specificity or severity that has been observed. "Unexpected," as used in this definition, also refers to adverse events or suspected adverse reactions that are mentioned in the package insert as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with Pazopanib.

# 8.3.8. Exposure in Utero

If any trial patient (or partner of a trial patient) becomes or is found to be pregnant during the study or within 28 days of discontinuing the investigational medication/product, the Investigator must report the information to TRACON, or designee via the Pregnancy Notification Report Form. This must be done irrespective of whether an adverse event has occurred and within 24 hours of awareness of the pregnancy. The information submitted should include the anticipated date of delivery.

The Investigator will follow the patient (or partner of a trial patient) until completion of the pregnancy or until pregnancy termination (i.e., induced abortion) and then notify TRACON, or its designee, of the outcome within 5 days or as specified below. The Investigator will provide this information as a follow-up to the initial report. The reason(s) for an induced abortion must be specified.

The Investigator should follow procedures for reporting an SAE if pregnancy outcome meets criteria for an SAE (i.e., spontaneous abortion, stillbirth, neonatal death, or congenital anomaly [including that in an aborted fetus]).

In the case of a live birth, the "normality" of the newborn can be assessed at the time of birth and the Pregnancy Outcome Report Form should be completed (i.e., no minimum follow-up period of a presumably normal infant must pass before a Pregnancy Outcome Report Form can be completed). The "normality" of an aborted fetus can be assessed by gross visual inspection unless pre-abortion laboratory findings are suggestive of a congenital anomaly.

Additional information about pregnancy outcomes that are classified as SAEs follows:

- "Spontaneous abortion" includes miscarriage and missed abortion.
- All neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, any infant death after 1 month that the Investigator assesses as possibly related to the *in utero* exposure to the investigational medication should also be reported.

#### 8.3.9. Follow-up of Unresolved Adverse Events

All adverse events should be followed until they are resolved or the Investigator assesses them as chronic or stable. Any increase or decrease in adverse event grade should be recorded as a new adverse event.

All serious and those non-serious events assessed by the Investigator as possibly related to the investigational medication/product should continue to be followed even after the patient's participation in the trial is over. Such events should be followed until they resolve or until the Investigator assesses them as "chronic" or "stable." The event should also be documented on the adverse event CRF.

# 8.4. Safety Monitoring

The TRACON Clinical Team will monitor safety throughout the study via the following activities:

- Surveillance for SAEs according to regulatory guidelines
- Routine monitoring of non-serious adverse experiences as they are recorded in the case report forms and the source documents at study sites
- A formally chartered TRACON in-house Safety Review Team that includes, among other staff, two physicians
- A formally chartered external Safety Review Team that includes three physicians
- Periodic teleconferences with the Principal Investigators to share experiences and ensure communication
- Toxicity information that may affect the treatment of patients on this study will be promptly communicated in writing to all participating clinical sites and institutions participating in this clinical trial.

# 9. OTHER ASSESSMENTS

# 9.1. Other Laboratory Assessments

#### 9.1.1. Pharmacokinetics

Samples will be sent to Fisher BioServices (Franklin, MA 02038) for storage. See separate laboratory manual for specific collection, storage and shipping information.

# 9.1.1.1. TRC105 Peak and Trough Concentration (Phase 1b dose levels -1, 1, 2 and expanded cohort 1 and angiosarcoma cohort 2)

A 5 mL blood sample will be collected prior to dosing with TRC105 on the days indicated within the Schedule of Assessments (Table 4 and Table 7).

A 5 mL blood sample will be collected within 10 minutes following each TRC105 infusion on the days indicated within the Schedule of Assessments (Table 4 and Table 7).

Samples will be separated and stored at approximately -70 °C for shipment to third party laboratory. See separate laboratory guide for further collection and shipment information.

# 9.1.1.2. TRC105 and Pazopanib Trough Concentration (Phase 1b dose levels 3, expanded cohort 2 and Phase 2 including angiosarcoma cohort 1)

A 5 mL blood sample each for TRC105 and pazopanib pharmacokinetics to be collected at the time-points indicated in the Schedule of Assessments (Table 5, Table 6 and Table 7), prior to starting the TRC105 infusion and prior to pazopanib dosing. Samples will be stored at approximately -70°C. Samples will be batch shipped as indicated in the laboratory manual to a third-party laboratory. See separate laboratory guide for further collection and shipment information. Additional PK samples may also be collected at the time of unexpected clinical events.

#### 9.1.2. TRC105 Immunogenicity

Samples will be sent to Fisher BioServices (Franklin, MA 02038). See separate laboratory manual for specific collection, storage and shipping information.

Anti-product antibody concentrations will be measured using validated ELISA methods at the time oints specified in the Schedule of Assessments ((Table 4, Table 5, Table 6 and Table 7) in all patients. Anti-product antibody concentrations will be evaluated in the context of pharmacokinetic parameters and AE profiles. Samples will be separated and stored at approximately -70 °C for shipment to Fisher BioServices. See separate laboratory guide for further collection and shipment information.

#### 9.1.3. Protein Biomarkers

One 10mL purple top (K<sub>2</sub>EDTA) tube of blood will be collected on the days indicated within the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7). Samples will be stored at approximately -70 °C and shipped to Fisher BioServices Inc. (10 Forge Park, Franklin, MA 02038) for storage until the time of analysis. Duke University Medical Center will analyze plasma for several biomarkers including but not limited to VEGF, VEGF-R2, PIGF and sCD105

(Phase 1 Biomarker Laboratory, Duke University Medical Center, 309 MSRB, Research Dr., Durham, NC 27710). Please see the separate laboratory guide for further collection and shipment information.

# 9.1.4. Archival Tumor Specimens

Archival specimens (formalin-fixed, paraffin-embedded) of the primary cancer and/or metastatic cancer specimen for each study participant will be obtained. It is preferable that the entire paraffin block be submitted, but if this is not feasible, then at least 20 unstained slides are requested for immunohistochemical analysis (sections of  $\sim 5$  microns are preferred).

Samples will be stored at room temperature and shipped to Fisher BioServices Inc. (10 Forge Park, Franklin, MA 02038) for storage until the time of analysis. See separate laboratory guide for further collection and shipment information.

#### 10. STATISTICS

# 10.1. Statistical Design/Sample Size

#### 10.1.1. Phase 1b Statistical Design/Sample Size

The number of patients to be enrolled in this study will depend upon the observed safety profile, which will determine the number of patients per dose level and the number of dose escalations. It is anticipated that up to 30 patients will be enrolled in the phase 1b portion of the study.

The probability of escalation to the next higher dose for each underlying true DLT rate is shown in Table 17. For example, at a dose level with a true DLT rate of 5%, there is a greater than 95% probability of escalating. Conversely, for a dose level with a true DLT rate of 70%, the probability of escalating is < 5%.

Table 17: Probability of Escalation to the Next Dose for Each True Underlying DLT Rate at a Dose Level

| True Underlying DLT Rate | 5% | 10% | 20% | 30% | 40% | 50% | 60% | 70% | 80% | 90% |
|---|---|---|---|---|---|---|---|---|---|---|
| Probability of Escalating Dose | 0.97 | 0.91 | 0.71 | 0.49 | 0.31 | 0.17 | 0.08 | 0.03 | 0.01 | 0.001 |

The probability of failing to observe DLT in a sample size of 3 or 6 patients given various true underlying DLT rates in shown in Table 18. For example, with 6 patients, the probability of failing to observe DLT occurring at least 40% of the time is less than 5%.

Table 18: Probability of Failing to Observe True Underlying DLT Rate at a Dose Level

| True Underlying DLT<br>Rate | 5% | 10% | 20% | 30% | 40% | 50% | 60% | 70% | 80% | 90% |
|---|---|---|---|---|---|---|---|---|---|---|
| Probability of Failing to<br>Observe Toxicity if N = | 0.86 | 0.73 | 0.51 | 0.34 | 0.22 | 0.13 | .0064 | 0.027 | 0.008 | 0.001 |
| Probability of Failing to<br>Observe Toxicity if N = | 0.74 | 0.53 | 0.26 | 0.12 | 0.047 | 0.016 | 0.0041 | <0.001 | <0.001 | <0.001 |

The estimated MTD is the highest tested dose level with a DLT rate < 33% in at least 6 DLT evaluable patients.

# 10.1.1.1. Definition of Analyzed Study Populations

The following study populations will be considered when reporting study results:

- The study population for safety includes all patients receiving at least a portion of 1 dose of TRC105.
- The study population for PK includes also subjects with adequate data for PK modeling of TRC105.

• The study population for efficacy will include all safety population patients who have baseline and follow-up tumor measurements as required for assessment by RECIST 1.1.

Patients who experience DLT who receive less than the prescribed dose of TRC105 or pazopanib due to documented toxicity in cycle 2 will be considered evaluable for dose escalation purposes.

Only those patients who are deemed "ineligible" or who receive no therapy (i.e. no TRC105 or pazopanib) will be eliminated from the analysis. Ineligible patients who receive therapy will not be included in the assessment of efficacy endpoints, but their data will be included in the assessment of all adverse event reporting.

#### 10.1.2. Phase 2 Statistical Design/Sample Size

Sixty three patients will be treated in the phase 2 portion of the study.

The study population for safety and efficacy will include all patients receiving at least a portion of one dose of TRC105.

Assuming a true median PFS of 4.6 months, a 9-month accrual period, a 6-month follow-up period, and based on the use of a one-sided test at the alpha=0.05 level of significance, a sample size of 63 patients will provide 86% power to detect a 50% increase in the median PFS (i.e., a median of 6.9 months). These power estimates are based on the approach of Lawless [1].

Two additional phase 2 cohorts of up to 13 patients each with angiosarcoma will be enrolled into separate cohorts, angiosarcoma cohort 1 and 2. Angiosarcoma cohort 1: Assuming a 15% response rate by RECIST with pazopanib alone, 5 responders with TRC105 alone or in combination with pazopanib will provide >90% confidence the true response rate is >15% (two-sided exact 90% binomial with 5 of 13 responders is 16.57 and 64.52%). Angiosarcoma cohort 2: Assuming a 15% response rate by RECIST with pazopanib alone, 5 responders with TRC105 in combination with pazopanib will provide >90% confidence that the true response rate is >15%.

For each of the angiosarcoma cohorts, the two-sided exact 90% binomial with 5 of 13 responders is 16.57% and 64.52%.

# 10.1.2.1. Definition of Analyzed Study Populations

The following study populations will be considered when reporting study results for the phase 2 portion:

- The study population for safety includes all patients receiving at least a portion of 1 dose of TRC105.
- The study population for efficacy will include all safety population patients who have baseline and follow-up tumor measurements as required for assessment by RECIST 1.1.

Only those patients who are deemed "ineligible" or who receive no therapy (i.e., no TRC105 or pazopanib) will be eliminated from the analysis. Ineligible patients who receive therapy will not

be included in the assessment of efficacy endpoints, but their data will be included in the assessment of all adverse event reporting.

# 10.2. Data Analysis

Descriptive statistics (such as means, medians, standard deviations and ranges for continuous data and percentages for categorical data) will be used to summarize patient characteristics, treatment administration/compliance, immunogenicity (anti-product antibodies), efficacy, pharmacokinetic parameters, protein biomarkers, and archival tumor tissue. Data will also be displayed graphically, where appropriate.

# 10.2.1. Analysis of Primary Objective

# 10.2.1.1. Phase 1b Analysis of Primary Objective

For each cohort, DLTs will be summarized by category (hematologic and non-hematologic) and by MedDRA preferred term.

All AEs with an onset after initiation of treatment will be considered as treatment-emergent AEs. A preexisting condition that worsens during the treatment period will also be considered as a treatment emergent AE. All AEs will be coded by system organ class (SOC) and preferred term using NCI CTCAE (MedDRA) version 4.0.

The number and percentage of patients with the following types of treatment-emergent AEs will be summarized: common and serious AEs, AEs related to study medication, AEs resulting in study discontinuation, and clinically significant laboratory abnormalities. Non-treatment-emergent serious AEs will be described separately. Deaths will be reported with demographic information.

#### 10.2.1.2. Phase 2 Analysis of Primary Objective

The primary analysis will test the null hypothesis that the median PFS is equal to 4.6 months. The time-to-event distribution for PFS will be estimated using the Kaplan-Meier method and the analysis will be based on the two-sided 90% confidence interval for the median (equivalent to the use of a one-sided test at the alpha=0.05 level of significance).

Additional exploratory analyses of PFS will be conducted in subgroups defined based on number of prior therapies (one versus two or more), histology, and endoglin expression on sarcoma tissue.

For the angiosarcoma cohorts, the overall response rate and median duration of response by RECIST 1.1 will be calculated and the response rate will include the two-sided 90% confidence interval.

# 10.2.2. Analysis of Pharmacokinetics

Peak and trough serum TRC105 concentrations will be measured using validated ELISA methods. The TRC105 pharmacokinetic data will be assessed for potential correlations with response, PFS, survival, adverse events, and baseline characteristics using descriptive statistics and models as appropriate.

#### 10.2.3. Objective Response

The best response (CR, PR, SD or PD according to RECIST 1.1) for each patient with measurable disease who received at least one dose of TRC105 study drug will be listed by cohort. Stable disease will be defined as lack of tumor progression lasting for 2 cycles or longer.

# 10.2.4. Analysis of Protein Biomarkers

Angiogenic protein biomarker data for each patient who received at least one dose of TRC105 study drug will be listed.

# 10.2.5. Analysis of Immunogenicity

Anti-product antibody concentrations will be measured using validated ELISA methods at the timepoints specified in the Schedule of Assessments (Table 4, Table 5, Table 6 and Table 7). Anti-product antibody concentrations will be evaluated in the context of pharmacokinetic parameters and AE profiles.

#### 10.2.6. Analysis of Archival Tumor Tissue

Endoglin expression within the tumor vasculature and on sarcoma tissue will be quantified for each patient who received at least one dose of TRC105 study drug and will be listed by histologic type of soft tissue sarcoma. Expression will be determined by immunohistochemistry (IHC). Other markers that may relate to efficacy or toxicity of TRC105 may also be explored.

# 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

All data entered on CRFs/eCRFs must be verifiable within the patients' source documents (written or electronic record). The Investigator /institution guarantees TRACON representatives and appropriate regulatory authorities direct access to the original source records for the duration of the agreed study record retention period. Printouts of source records that are electronically obtained and stored will not be acceptable for audit/inspection unless provided as certified exact copies and the data remains as meaningful and useful as in its original electronic state.

Legally protected subject identification and other personal health information must be securely stored with limited access by the participating institutions. Unless secure provisions are established by the institution to allow TRACON (or designee) to perform remote monitoring of electronic source records, TRACON (or designee) will review source records/data on site and will not remove any such protected health information.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

Monitoring visits to clinical investigator sites will be made by TRACON or its representatives periodically during the trial to ensure that GCPs and all aspects of the protocol are being followed.

The trial site will also be subject to possible inspection by the institutional review board (IRB) or independent ethics committee (IEC) or other appropriate regulatory authority. The trial site is also subject to quality assurance audits performed by TRACON or its representatives.

It is important that the Investigator(s) and their relevant personnel are available during the monitoring visits, audits, and inspections and that sufficient attention, time, and support is devoted to the process.

TRACON and its representatives will be governed by applicable regulations, good clinical practice standards, and internal SOPs for the conduct of monitoring visits and QA audits.

#### 13. ETHICS

# 13.1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

It is the responsibility of the Investigator to have approval of the trial protocol, protocol amendments, informed consent forms, and advertisements from the IRB/IEC before potential patients are consented for participation on the trial. All correspondence and other evidence of appropriate and timely communications with the IRB/IEC should be retained in the Investigator/site files. Copies of all IRB/IEC approvals should also be forwarded to TRACON.

The only circumstance in which an amendment may be initiated prior to IRB/IEC approval is where the change is necessary to eliminate apparent immediate hazards to the patients. In that event, the Investigator must notify the IRB/IEC and TRACON in writing within 5 business days after the implementation.

# 13.2. Ethical Conduct of the Study

The trial will be performed in accordance with the protocol, applicable local regulatory requirements and laws, and the International Conference on Harmonization Guideline on Good Clinical Practice, which supports the application of ethical principles that have their origin in the Declaration of Helsinki (see ICH E6, § 2.1).

# 13.3. Written Informed Consent

The informed consent form language must be agreed upon by TRACON and the IRB/IEC and must be in compliance with ICH GCP, local regulatory requirements, and legal requirements. The informed consent information must not be changed without prior approval by TRACON and the IRB/IEC. The informed consent form used in this trial, and any changes made during the course of the trial, must be approved by both the IRB/IEC and TRACON, or designee, before use.

It is the responsibility of the Investigator to give each patient full and adequate verbal and written information regarding the objective and procedures of the trial and the possible risks involved. This information must be provided to the patient prior to undertaking any trial-related procedure. Patients must be informed about their right to withdraw from the trial at any time. Furthermore, it is the responsibility of the Investigator to ensure all patients are appropriately informed before obtaining their signed and dated consent. Signatures from the investigator conducting the informed consent discussion should also be obtained, prior to undertaking any trial-related procedure. Consent by a legally authorized representative is not permitted. Should an impartial witness be needed, ICH E6 requirements for impartial witnesses will apply.

The Investigator will retain the original of each patient's signed consent form in the Investigator/site files.

# **13.4.** Patient Compensation

Patients will not be compensated for participation in this trial; this will be outlined in the patient informed consent form.

# 14. DATA HANDLING AND RECORDKEEPING

# 14.1. Inspection of Records

CRF's are required and should be completed for each patient who receives treatment with pazopanib or TRC105. Screen failure CRF's will not be collected. Nevertheless, records of potential patients identified and screened shall be retained on site screening logs. The completed original CRFs are the sole property of TRACON and should not be made available in any form to third parties without written permission from TRACON (except for authorized representatives of the HRA and in accordance with HIPAA regulations).

It is the Investigator's responsibility to ensure completion and to review and approve all CRF data. The investigator will sign off on his/her data per patient. These signatures serve to attest that the investigator has reviewed and approved the information contained on the case report forms and that the information is complete, accurate, and true. At all times, the Investigator has final personal responsibility for the accuracy and authenticity of all clinical and laboratory data entered on the CRFs.

The use of electronic CRFs (eCRFs) to capture study data using automated computerized data capture systems does not change the principles and requirements for collecting study data. The investigator still retains final personal responsibility for eCRF data and any associated data pertaining to it (e.g. metadata including any record of change to the originally recorded data). The investigator's signed approval of the eCRF data serves to attest that the electronic data and all of its associated metadata (including changes) has been reviewed and accepted as complete, accurate, and true for each patient in the study.

#### 14.2. Retention of Records

To allow for appropriate evaluations and/or audits by regulatory authorities or TRACON, the Investigator agrees to keep records, including the identity of all participating patients (sufficient information to link records, CRFs and hospital records), all original signed informed consent forms, copies of all CRFs, source documents, and detailed records of treatment disposition. The Investigator should retain these records according to local regulations or as specified in the Clinical Trial Agreement, whichever is longer.

If the Investigator relocates, retires, or for any reason withdraws from the study, then TRACON should be prospectively notified. The study records must be transferred to an acceptable designee, such as another Investigator or another institution. The Investigator must inform TRACON of any such transfer of responsibilities and properly identify the person or institution assuming the responsibility. The responsible investigator/institution must obtain TRACON's written permission before disposing of any records.

#### 15. DEFINITION OF END OF TRIAL

# 15.1. End of Trial in all Participating Countries

End of trial in all participating countries is defined as the time at which all patients enrolled in the study have completed treatment on study.

#### 15.2. End of Trial in a Member State

End of trial in a Member State of the European Union is defined as the time at which it is deemed that sufficient patients have been recruited and completed the trial as stated in the regulatory application (e.g. the Clinical Trials Agreement (CTA)) and ethics application in the Member State. Poor recruitment is not a reason for premature termination but is considered a normal conclusion to the trial in that Member State.

#### 15.3. TRACON Discontinuation Criteria

Premature termination of this trial may occur because of a regulatory authority decision, change in opinion of the IRB/IEC, drug safety problems, or at the discretion of TRACON. In addition, TRACON retains the right to discontinue development of TRC105 at any time.

TRACON reserves the right to discontinue the trial prior to inclusion of the intended number of patients, but intends only to exercise this right for valid scientific or administrative reasons. If a trial is prematurely terminated or discontinued, TRACON will promptly notify the Investigator. After notification, the Investigator must contact all participating patients within a 28 day time period. As directed by TRACON, all trial materials must be collected and all CRF data must be completed to the greatest extent possible.

# 16. PUBLICATION OF TRIAL RESULTS

Publication of trial results is discussed in the Clinical Trial Agreement.

# 17. FINANCING AND INSURANCE

Financing and Insurance are discussed in the Clinical Trial Agreement.

# 18. INVESTIGATOR PROTOCOL AGREEMENT: 105SAR101

I understand that all information concerning this study supplied to me by TRACON Pharmaceuticals, Inc. is confidential information. I have read this protocol and agree to conduct the study according to all applicable regulations, Good Clinical Practice Guidelines, and in accordance with the Clinical Trial Agreement.

I understand that this protocol and all amendments must be submitted to the appropriate IRB/IEC.

| Investigator Name (PLEASE PRINT): | |
|-----------------------------------|-------|
| Signature: | Date: |

# Please sign and return this agreement to:

TRACON Pharmaceuticals, Inc. Attn: Clinical Operations 8910 University Center Lane, Suite 700 San Diego, CA 92122

Please keep a copy for your records.

# 19. REFERENCES

- 1. J., L., Statistical Models and Methods for Lifetime Data1982, New York John Wiley and Sons.
- 2. Carmeliet, P., Angiogenesis in health and disease. Nat Med, 2003. 9(6): p. 653-60.
- 3. Folkman, J. and Y. Shing, *Angiogenesis*. J Biol Chem, 1992. **267**(16): p. 10931-4.
- 4. Hurwitz, H., et al., *Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer.* N Engl J Med, 2004. **350**(23): p. 2335-42.
- 5. Sandler, A., et al., *Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer.* N Engl J Med, 2006. **355**(24): p. 2542-50.
- 6. Miller, K.D., et al., Randomized phase III trial of capecitabine compared with bevacizumab plus capecitabine in patients with previously treated metastatic breast cancer. J Clin Oncol, 2005. **23**(4): p. 792-9.
- 7. Friedman, H.S., et al., *Bevacizumab alone and in combination with irinotecan in recurrent glioblastoma*. J Clin Oncol, 2009. **27**(28): p. 4733-40.
- 8. Escudier, B., et al., *Phase III trial of bevacizumab plus interferon alfa-2a in patients with metastatic renal cell carcinoma (AVOREN): final analysis of overall survival.* J Clin Oncol, 2010. **28**(13): p. 2144-50.
- 9. Escudier, B., et al., *Sorafenib in advanced clear-cell renal-cell carcinoma*. N Engl J Med, 2007. **356**(2): p. 125-34.
- 10. Llovet, J.M., et al., *Sorafenib in advanced hepatocellular carcinoma*. N Engl J Med, 2008. **359**(4): p. 378-90.
- 11. Motzer, R.J., et al., *Sunitinib versus interferon alfa in metastatic renal-cell carcinoma*. N Engl J Med, 2007. **356**(2): p. 115-24.
- 12. Rini, B.I., *Vascular endothelial growth factor-targeted therapy in metastatic renal cell carcinoma*. Cancer, 2009. **115**(10 Suppl): p. 2306-12.
- 13. Jemal, A., et al., *Cancer statistics*, 2010. CA Cancer J Clin, 2010. **60**(5): p. 277-300.
- 14. Hogendoorn, P.C., et al., *Changing concepts in the pathological basis of soft tissue and bone sarcoma treatment.* Eur J Cancer, 2004. **40**(11): p. 1644-54.
- 15. Kawaguchi, S., et al., *A quest for therapeutic antigens in bone and soft tissue sarcoma*. J Transl Med, 2005. **3**: p. 31.
- 16. Dominici, M., et al., Minimal criteria for defining multipotent mesenchymal stromal cells. The International Society for Cellular Therapy position statement. Cytotherapy, 2006. **8**(4): p. 315-7.
- 17. Tolar, J., et al., *Sarcoma derived from cultured mesenchymal stem cells*. Stem Cells, 2007. **25**(2): p. 371-9.
- 18. Postiglione, L., et al., *Differential expression and cytoplasm/membrane distribution of endoglin (CD105) in human tumour cell lines: Implications in the modulation of cell proliferation.* Int J Oncol, 2005. **26**(5): p. 1193-201.

# **5.3.5.2 Clinical Protocol**

- 19. Gromova, P., et al., *ENDOGLIN/CD105* is expressed in KIT positive cells in the gut and in gastrointestinal stromal tumours. J Cell Mol Med, 2012. **16**(2): p. 306-17.
- 20. Pardali, E., et al., *Critical role of endoglin in tumor cell plasticity of Ewing sarcoma and melanoma*. Oncogene, 2011. **30**(3): p. 334-45.
- 21. Ciernik, I.F., et al., Expression of transforming growth factor beta and transforming growth factor beta receptors on AIDS-associated Kaposi's sarcoma. Clin Cancer Res, 1995. **1**(10): p. 1119-24.
- 22. Gibbs, C.P., et al., *Stem-like cells in bone sarcomas: implications for tumorigenesis*. Neoplasia, 2005. **7**(11): p. 967-76.
- 23. Morozov, A., et al., *Benign mesenchymal stromal cells in human sarcomas*. Clin Cancer Res, 2010. **16**(23): p. 5630-40.
- 24. Ohta, M., et al., *A case of angiosarcoma of the breast*. Jpn J Clin Oncol, 1997. **27**(2): p. 91-4.
- 25. Royer-Pokora, B., et al., Wilms tumor cells with WT1 mutations have characteristic features of mesenchymal stem cells and express molecular markers of paraxial mesoderm. Hum Mol Genet, 2010. **19**(9): p. 1651-68.
- 26. Haruta, Y. and B.K. Seon, *Distinct human leukemia-associated cell surface glycoprotein GP160 defined by monoclonal antibody SN6*. Proc Natl Acad Sci U S A, 1986. **83**(20): p. 7898-902.
- 27. Gougos, A. and M. Letarte, *Identification of a human endothelial cell antigen with monoclonal antibody 44G4 produced against a pre-B leukemic cell line*. J Immunol, 1988. **141**(6): p. 1925-33.
- 28. Seon, B.K., et al., Long-lasting complete inhibition of human solid tumors in SCID mice by targeting endothelial cells of tumor vasculature with antihuman endoglin immunotoxin. Clin Cancer Res, 1997. **3**(7): p. 1031-44.
- 29. Cheifetz, S., et al., *Endoglin is a component of the transforming growth factor-beta receptor system in human endothelial cells.* J Biol Chem, 1992. **267**(27): p. 19027-30.
- 30. Li, D.Y., et al., *Defective angiogenesis in mice lacking endoglin*. Science, 1999. **284**(5419): p. 1534-7.
- 31. Burrows, F.J., et al., *Up-regulation of endoglin on vascular endothelial cells in human solid tumors: implications for diagnosis and therapy*. Clin Cancer Res, 1995. **1**(12): p. 1623-34.
- 32. Seon, B.K., *Expression of endoglin (CD105) in tumor blood vessels*. Int J Cancer, 2002. **99**(2): p. 310-1; author reply 312.
- 33. Horsman, M.R. and D.W. Siemann, *Pathophysiologic effects of vascular-targeting agents and the implications for combination with conventional therapies*. Cancer Res, 2006. **66**(24): p. 11520-39.
- 34. Matsuno, F., et al., *Induction of lasting complete regression of preformed distinct solid tumors by targeting the tumor vasculature using two new anti-endoglin monoclonal antibodies.* Clin Cancer Res, 1999. **5**(2): p. 371-82.

- 35. Takahashi, N., et al., Antiangiogenic therapy of established tumors in human skin/severe combined immunodeficiency mouse chimeras by anti-endoglin (CD105) monoclonal antibodies, and synergy between anti-endoglin antibody and cyclophosphamide. Cancer Res, 2001. **61**(21): p. 7846-54.
- 36. Tsujie, M., et al., *Anti-tumor activity of an anti-endoglin monoclonal antibody is enhanced in immunocompetent mice.* Int J Cancer, 2008. **122**(10): p. 2266-73.
- 37. Uneda, S., H. Toi, and B.K. Seon, *Anti-endoglin monoclonal antibodies are effective for suppressing metastasis and the primary tumors by targeting tumor vasculature*. Int J Cancer, 2009. **125**: p. 1446.
- 38. Barbara, N.P., J.L. Wrana, and M. Letarte, *Endoglin is an accessory protein that interacts with the signaling receptor complex of multiple members of the transforming growth factor-beta superfamily.* J Biol Chem, 1999. **274**(2): p. 584-94.
- 39. She, X., et al., Synergy between anti-endoglin (CD105) monoclonal antibodies and TGF-beta in suppression of growth of human endothelial cells. Int J Cancer, 2004. **108**(2): p. 251-7.
- 40. Olivier Nolan-Stevaux, W.Z., Stacey Culp, Kathy Shaffer, Joseph Hoover, Dineli Wickramasinghe, Astrid Ruefli-Brasse, *Endoglin Requirement for BMP9 Signaling in Endothelial Cells Reveals New Mechanism of Action for Selective Anti-Endoglin Antibodies*. PLOS ONE, 2012. 7(12): p. e50920.
- 41. Guo, B., et al., *CD105 inhibits transforming growth factor-beta-Smad3 signalling*. Anticancer Res, 2004. **24**(3a): p. 1337-45.
- 42. Warrington, K., et al., Functional role of CD105 in TGF-beta1 signalling in murine and human endothelial cells. Anticancer Res, 2005. **25**(3B): p. 1851-64.
- 43. Sanchez-Elsner, T., et al., *Endoglin expression is regulated by transcriptional cooperation between the hypoxia and transforming growth factor-beta pathways*. J Biol Chem, 2002. **277**(46): p. 43799-808.
- 44. van Laake, L.W., et al., *Endoglin has a crucial role in blood cell-mediated vascular repair*. Circulation, 2006. **114**(21): p. 2288-97.
- 45. Lenato, G.M. and G. Guanti, *Hereditary Haemorrhagic Telangiectasia (HHT): genetic and molecular aspects*. Curr Pharm Des, 2006. **12**(10): p. 1173-93.
- 46. Sabba, C., et al., *Life expectancy in patients with hereditary haemorrhagic telangiectasia*. Qjm, 2006. **99**(5): p. 327-34.
- 47. Rokhlin, O.W., et al., *Differential expression of endoglin on fetal and adult hematopoietic cells in human bone marrow.* J Immunol, 1995. **154**(9): p. 4456-65.
- 48. Kumar, S., et al., *Breast carcinoma: vascular density determined using CD105 antibody correlates with tumor prognosis.* Cancer Res, 1999. **59**(4): p. 856-61.
- 49. Vo, M.N., et al., Elevated plasma endoglin (CD105) predicts decreased response and survival in a metastatic breast cancer trial of hormone therapy. Breast Cancer Res Treat, 2008.

# **5.3.5.2 Clinical Protocol**

- 50. Tanaka, F., et al., Evaluation of angiogenesis in non-small cell lung cancer: comparison between anti-CD34 antibody and anti-CD105 antibody. Clin Cancer Res. 2001. 7(11): p. 3410-5.
- 51. El-Gohary, Y.M., et al., Endoglin (CD105) and vascular endothelial growth factor as prognostic markers in prostatic adenocarcinoma. Am J Clin Pathol, 2007. 127(4): p. 572-9.
- 52. Svatek, R.S., et al., Preoperative plasma endoglin levels predict biochemical progression after radical prostatectomy. Clin Cancer Res. 2008. 14(11): p. 3362-6.
- 53. Li, C., et al., Both high intratumoral microvessel density determined using CD105 antibody and elevated plasma levels of CD105 in colorectal cancer patients correlate with poor prognosis. Br J Cancer, 2003. 88(9): p. 1424-31.
- 54. Romani, A.A., et al., The risk of developing metastatic disease in colorectal cancer is related to CD105-positive vessel count. J Surg Oncol, 2006. 93(6): p. 446-55.
- 55. Rubatt, J.M., et al., Independent prognostic relevance of microvessel density in advanced epithelial ovarian cancer and associations between CD31, CD105, p53 status, and angiogenic marker expression: A Gynecologic Oncology Group study. Gynecol Oncol, 2009. **112**(3): p. 469-74.
- 56. Taskiran, C., et al., The prognostic value of endoglin (CD105) expression in ovarian carcinoma. Int J Gynecol Cancer, 2006. 16(5): p. 1789-93.
- Ding, S., et al., Comparative evaluation of microvessel density determined by CD34 or 57. CD105 in benign and malignant gastric lesions. Hum Pathol, 2006. 37(7): p. 861-6.
- 58. Erdem, O., et al., CD105 expression is an independent predictor of survival in patients with endometrial cancer. Gynecol Oncol, 2006. 103(3): p. 1007-11.
- 59. Yao, Y., et al., Prognostic significance of microvessel density determined by an anti-CD105/endoglin monoclonal antibody in astrocytic tumors: comparison with an anti-CD31 monoclonal antibody. Neuropathology, 2005. 25(3): p. 201-6.
- 60. Yang, L.Y., et al., Correlation between CD105 expression and postoperative recurrence and metastasis of hepatocellular carcinoma. BMC Cancer, 2006. 6: p. 110.
- 61. Saad, R.S., et al., Endoglin (CD105) and vascular endothelial growth factor as prognostic markers in esophageal adenocarcinoma. Hum Pathol, 2005. **36**(9): p. 955-61.
- 62. Kyzas, P.A., N.J. Agnantis, and D. Stefanou, Endoglin (CD105) as a prognostic factor in head and neck squamous cell carcinoma. Virchows Arch, 2006. 448(6): p. 768-75.
- 63. Marioni, G., et al., Endoglin expression is associated with poor oncologic outcome in oral and oropharyngeal carcinoma. Acta Otolaryngol, 2006. 126(6): p. 633-9.
- 64. Bockhorn, M., et al., Differential vascular and transcriptional responses to anti-vascular endothelial growth factor antibody in orthotopic human pancreatic cancer xenografts. Clin Cancer Res, 2003. 9(11): p. 4221-6.
- Davis, D.W., et al., Regional effects of an antivascular endothelial growth factor receptor 65. monoclonal antibody on receptor phosphorylation and apoptosis in human 253J B-V bladder cancer xenografts. Cancer Res, 2004. 64(13): p. 4601-10.

- 66. Shiozaki, K., et al., *Antiangiogenic chimeric anti-endoglin (CD105) antibody:* pharmacokinetics and immunogenicity in nonhuman primates and effects of doxorubicin. Cancer Immunol Immunother, 2006. **55**(2): p. 140-50.
- 67. GlaxoSmithKline, *VOTRIENT (pazopanib) tablets*. <a href="http://www.accessdata.fda.gov/drugsatfda\_docs/label/2012/022465s-010S-012lbl.pdf">http://www.accessdata.fda.gov/drugsatfda\_docs/label/2012/022465s-010S-012lbl.pdf</a>, 2009.
- 68. Eisenhauer, E.A., et al., *New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1).* Eur J Cancer, 2009. **45**(2): p. 228-47.

# 20. APPENDICES

# **20.1.** Appendix 1: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)

The NCI CTCAE (Version 4.0) should be used to assess Adverse Events and may be reviewed on-line at the following NCI website:

http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/ctcaev4.pdf

# 20.2. Appendix 2: ECOG Performance Status

| Grade | Performance |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction. |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours. |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. |
| 5 | Dead. |